

# PM1183-A-003-10 (NCT01970540)

Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM01183 in Combination with Doxorubicin in Non-heavily Pretreated Patients with Selected Advanced Solid Tumors

## STATISTICAL ANALYSIS PLAN

Version Date V4.0 12Feb2018

# **Table of Contents**

| Li | st of A | bbreviationsbbreviations | 5 |
|---|---|---|---|
| 1. | Intr | roduction | 7 |
| 2. | Stu | dy Objectives | <i>7</i> |
| | 2.1. | Primary Objective | |
| | 2.2. | Secondary Objectives. | |
| <i>3</i> . | | dy Design. | |
| | | • | |
| <i>4</i> . | San | nple Size and Dose Escalation | |
| | 4.1. | Sample Size | |
| | 4.2. | Dose Escalation Schedule. | 10 |
| <b>5.</b> | Pop | pulation and Endpoints | 10 |
| | 5.1. | Patient Evaluability Criteria | 11 |
| | 5.2. | Endpoints | 11 |
| | 5.2.1 | | |
| | 5 | .2.1.1. Determination of MTD and RD. | 12 |
| | 5. | .2.1.2. DLT Criteria | 13 |
| | 5.2.2 | | |
| | | .2.2.1. Safety | |
| | | .2.2.2. Efficacy. | |
| | | .2.2.3. Pharmacokinetics. | |
| | | .2.2.4. Pharmacogenomics. | |
| <b>6.</b> | Gen | neral analysis methods | 15 |
| | 6.1. | Statistical Software. | 15 |
| | 6.2. | Data Analysis Conventions. | 15 |
| <i>7</i> . | Stat | tistical analysis | 15 |
| | 7.1. | Patient Disposition and Protocol Deviations | 15 |
| | 7.2. | Baseline Characteristics. | |
| | 7.2.1 | | |
| | 7.3. | Statistical Analysis for Safety. | 17 |
| | 7.3.1 | | |
| | 7.3.2 | <u>.</u> | |
| | 7.3.3 | · | |
| | 7.3.4 | 4. Adverse Events | 18 |
| | 7.3.5 | | |
| | 7.3.6 | | |
| | | 3.6.1. Hematology | |
| | | .3.6.2. Serum Biochemistry and Coagulation Tests. | |
| | 7.3.7 | • | |
| | 7.3.8 | | |
| | 7.3.9 | Č | |
| | 7.3.1 | | |
| | 7.4. | Statistical analysis for efficacy | 21 |

| 7.4.1.<br>7.4.2. | Exploratory Analysis of Antitumor Activity. Level of Significance. | |
|---|---|---|
| | statistical analysis | |
| | Stratification and Covariate Analysis | |
| | Multivariate Analysis | |
| | Subgroup Analysis | |
| | nterim Analysis. | |
| | Missing Values Management. | |
| | Decimals Places. | |
| | s, Listings and Figures | |
| | vendix I. Patients Disposition | |
| | General Characteristics | |
| 10.1. | | |
| 10.1.1. | , | |
| 10.1.2. | | |
| 10.2. F | Patient Characteristics | 36 |
| 10.2.1. | | |
| 10.2.2. | Cancer History. | 40 |
| 10.2.3. | | |
| 10.2.4. | <b>J</b> | |
| 10.2.5.<br>10.2.6. | | |
| 10.2.6. | 1. | |
| 10.2.7. | | |
| 10.2.9. | $\epsilon$ | |
| 10.2.10 | | |
| 10.2.11 | | |
| 10.2.12 | $\mathcal{E}$ | |
| 10.2.13 | | |
| 11. App | pendix II. Safety Evaluation | 52 |
| | Extent of Exposure | |
| 11.1.1. | | |
| 11.1.2.<br>11.1.3. | - <b>,</b> - , - | |
| 11.1.3. | | |
| 11.2. I | Oose-Limiting Toxicities | 58 |
| 11.2.1. | e e | |
| | Adverse Events (AEs) | |
| 11.3.1. | Display of Adverse Events | |
| | Deaths and Other Serious Adverse Events | |
| 11.4.1.<br>11.4.2. | Deaths. Serious Adverse Events. | |
| | Clinical Laboratory Evaluation | |
| 11.5.1.<br>11.5.2. | Hematological Abnormalities. Biochemical Abnormalities. | |
| 11.5.2. | | |
| 11.5.4. | | |

| 11.6. | Vital Signs, Physical Findings, ECG, LVEF and Pregnancy tests | 74 |
|--------|---------------------------------------------------------------|-----|
| | 1. Vital Signs and Physical Findings. | |
| | 2. Electrocardiogram | |
| | 3. LVEF | |
| 11.7. | Concomitant and Prophylactic Medication | 78 |
| 11.7. | | 78 |
| 12. A | ppendix III. Efficacy Evaluation | 81 |
| 12.1. | Efficacy Analysis. | 81 |
| | 1. Response. | |
| 13. F | igures | 84 |
| 14. D | atabase Listings | 93 |
| 15. S. | AP Version History | 95 |
| 15.1. | SAP Version History v1 | 95 |
| 15.2. | SAP Version History v2 | 102 |
| 15.3. | SAP Version History v3 | 104 |

### **List of Abbreviations**

AE(s) Adverse Event(s) AFP Alpha-fetoprotein

ALT Alanine Aminotransferase
ANC Absolute Neutrophil Count
AP Alkaline phosphatase

**ASCO** American Society of Clinical Oncology

**AST** Aspartate Aminotransferase

BSA Body Surface Area
BPD Blood Diastolic Pressure
BPS Blood Systolic Pressure
CA-125 Carbohydrate Antigen-125
CA15-3 Carbohydrate Antigen 15-3
CA19-9 Carbohydrate Antigen 19-9
CEA Carcinoembryonic Antigen

**CI** Confidence Interval

**CL** Clearance

**Cmax** Maximum Plasma Concentration

**CPK** Creatine Phosphokinase

**CPK-MB** Creatine Phosphokinase Muscle-Brain (serum CPK isoenzymes found in

cardiac muscle)

**CR** Complete Response/Complete Regression

CrCl Creatinine Clearance CRF Case Report Form

CTFI Chemotheraphy Free-Interval
CT-scan Computed Tomography Scan
DAC Data Analysis Conventions

d/D Day(s)

DI Dose Intensity
DL Dose Level

DLT Dose-Limiting ToxicityECG ElectrocardiogramECHO Echocardiography

**ECOG-PS** Performance Status according to Eastern Cooperative Oncology Group

FD Flat Dose FUP Follow-up

**G-CSF** Granulocyte Colony-stimulating Factor

CSF Colony-stimulating Factor
GCIG Gynecologic Cancer Intergroup

GCP Good Clinical Practice
GGT Gama-glutamyltransferasa

**HR** Heart Rate

i.v. Intravenous (intravenously)IB Investigator's Brochure

**ICF** Informed Consent Form

**ICH** International Conference on Harmonization

IEC Independent Ethics Committees
INR International Normalized Ratio

**LDH** Lactate Dehydrogenase

**LVEF** Left Ventricular Ejection Fraction

minMinutesmlMilliliter

MRIMagnetic Resonance ImagingMTDMaximum Tolerated DoseMUGAMultiple-gated Acquisition Scan

NCI National Cancer Institute

NCI-CTCAE National Cancer Institute - Common Terminology Criteria for Adverse

Events (version 4 will be used for this trial)

**NSCLC** Non-small Cell Lung Cancer

OS Overall Survival

PFS Progression Free Survival
PD Progressive Disease
PGx Pharmacogenomic(s)
PK Pharmacokinetic(s)
PR Partial Response
PS Performance Status
PT Prothrombin Time

**PTT** Partial Thromboplastin Time

**q3wk** Every 3 Weeks **RD** Recommended Dose

QT Interval (measure of the time between the start of the Q wave and the

end of the T wave in the heart's electrical cycle)

QTcF Louis Sigurd Fridericia's formula for the correction of the QT interval RECIST Response Evaluation Criteria In Solid Tumors (version 1.1 will be used for

this trial)

**RT** Radiotherapy

SAE(s) Serious Adverse Event(s) SAP Statistical Analysis Plan

SecSecondsSDStable DiseaseTATumor AssessmentSTDStandard Deviation

**TFI** Systemic Chemotheraphy Free Interval

TTP Time to Progression
ULN Upper Limit of Normal
WBC White Blood Cells

WHO World Health Organization

#### 1. Introduction.

This document [Statistical Analysis Plan (SAP)] explains in detail the statistical analyses that will be carried out for the PharmaMar PM1183-A-003-10 study.

The analyses described in this SAP are based upon and supplement those described in the study protocol version 1.0, version 2.0 and version 3.0 and the protocol amendments No.1, dated 21 November 2011, No.2, dated 10 July 2013, No.3, dated 17 October 2014 and No.1 Non substantial amendment, dated 30 January 2015.

# 2. Study Objectives.

The clinical trial protocol states the following:

## 2.1. Primary Objective.

• To determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 in combination with doxorubicin in patients with selected advanced solid tumors.

## 2.2. Secondary Objectives.

- To determine the MTD and the RD of PM01183 in combination with doxorubicin with primary prophylaxis with granulocyte-colony stimulating factor (G-CSF) in patients with selected advanced solid tumors [if dose-limiting toxicities (DLTs) of the combination without G-CSF prophylaxis are exclusively related to neutropenia].
- To characterize the safety profile and feasibility of this combination in patients with selected advanced solid tumors.
- To characterize the pharmacokinetics (PK) of this combination and to detect major drug-drug PK interactions.
- To obtain preliminary information on the clinical antitumor activity of this combination in non-heavily pretreated selected solid tumor patients.
- Based on promising findings, to explore the feasibility, safety and efficacy of a potential improvable dose of this combination in selected tumor types [i.e. small cell lung cancer (SCLC) and endometrial cancer).
- To evaluate the pharmacogenomics (PGx) in tumor samples of patients exposed to PM01183 and doxorubicin at the RD in order to assess potential markers of response and/or resistance.

## 3. Study Design.

Prospective, open-label, dose-ranging, uncontrolled phase I study with escalating doses of PM01183 in combination with fixed doses of doxorubicin (see escalation dose scheme in section 4.2).

Patients will start receiving intravenous (i.v). doxorubicin 50 mg/m<sup>2</sup> (fixed dose) as bolus followed by PM01183 3.5 mg flat dose (FD) i.v. over one hour on Day 1 q3wk. A cycle is defined as an interval of three weeks.

Cohorts of three to six patients will be included at each dose level (DL). If no DLT occurs in more than one patient within each cohort, escalation will proceed to the following dose level. If one of the first three evaluable patients experiences a DLT, the dose level should be expanded up to six patients.

The MTD will be the lowest dose level explored during the dose escalation at which more than one evaluable patient experience a DLT in Cycle 1. All evaluable patients within a dose level will be followed for at least one cycle (i.e., three weeks) before dose escalation may proceed. Dose escalation will be terminated once the MTD or the last dose level (DL4) is reached, whichever occurs first, except if all DLTs occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than seven days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis. An expansion cohort to complete a minimum of nine evaluable patients will be recruited at the immediate lower dose level, or at the last dose level (DL4) if the MTD is not defined yet. This level will be confirmed as the RD if less than one third of the first nine evaluable patients experience DLT during Cycle 1.

Further to the finding of encouraging antitumor activity in the first 43 evaluable patients (13 responses, including four complete responses, with five partial responses in eight patients with small cell lung cancer, and one complete and one partial response in three patients with endometrial cancer), expansion of the cohort treated at the RD has been increased to include approximately 30 additional patients, for a total of around 39 patients.

In addition, a new cohort B of 20 evaluable patients with small cell lung cancer (SCLC) who failed treatment after first-line standard cytotoxic-containing therapy and at least nine evaluable patients with endometrial cancer will be included to further define the efficacy, safety and feasibility of a doxorubicin dose adaptation (doxorubicin 40 mg/m² and PM01183 2.0 mg/m²). The administered doses of both PM01183 and doxorubicin will be capped at 2.0 m² of body surface area (BSA) for any patients exceeding this BSA value. Patients in this cohort who have received ten cycles of the doxorubicin/PM01183 combination or have to discontinue doxorubicin due to a cardiac AE may continue receiving treatment with single-agent PM01183 at 4.0 mg/m² q3wk if patient benefit is perceived according to the Investigator. These patients will be followed every three months until death or the date of study termination, whichever occurs first.

Patients will be divided into two cohorts. Cohort A will consist of all patients included before the implementation of protocol amendment #3, and Cohort B will consist of all patients included after the implementation of protocol amendment #3.

In the event of DLTs occurring in the first patient at the first level, the second and third patients will be included at least two weeks apart. Otherwise and/or at subsequent dose levels, all patients within a dose level may be treated simultaneously.

Patients treated at the expansion cohort must be evaluable by RECIST v.1.1 and/or by serum markers (carbohydrate antigen-125, CA-125) in the case of ovarian cancer, as appropriate [according to the Gynecologic Cancer Intergroup (GCIG) specific criteria] (see study protocol, section 9.7), and must have documented disease progression according to any of these criteria. The tumor type(s) that will be eligible to be included in the expansion cohort at the RD will be chosen according to the preliminary efficacy observed among those previously treated during the escalation phase, and will be discussed and agreed between the investigators and the Sponsor.

Intermediate dose levels could be tested on agreement between the Investigator and the Sponsor, if deemed appropriate.

Patients will receive PM01183 and doxorubicin until progression, unacceptable toxicity, consent withdrawal or while it is considered to be in their best interest. More specifically, doxorubicin will be administered in the absence of disease progression or unacceptable toxicity before a maximal total cumulative dose of 450 mg/m² is reached. Thus, a maximum of ten cycles of the combination will be administered to patients with SCLC and endometrial cancer included in the new cohort B. Once this dose has been reached, the patients may continue treatment with PM01183 alone at the established single-agent RD, 7.0 mg FD q3wk and for patients included in the new cohort B they may continue treatment with PM01183 alone at 4.0 mg/m² q3wk.

Tumor assessments will be done every six weeks while on treatment. After treatment discontinuation, patients will be followed every four weeks until resolution or stabilization of all toxicities, if any. Patients discontinuing treatment without progression will be followed every two months until disease progression, other antitumor therapy, death or the date of study termination, whichever occurs first (see study protocol, section 5.9).

In the new cohort B, patients with SCLC and endometrial cancer will be followed every three months until death or the date of study termination, whichever occurs first. Antitumor response will be assessed using the RECIST v.1.1 and/or serum tumor markers as appropriate (e.g., ovarian cancer markers).

No serum markers will be evaluated in patients with SCLC and endometrial cancer included in the new cohort B. Patients will be evaluated at scheduled visits on three study periods: Pretreatment, Treatment and Follow-up (see study protocol, section 5.2).

## 4. Sample Size and Dose Escalation.

## 4.1. Sample Size.

The number of patients may vary depending both on the tolerability to PM01183 combined with doxorubicin and the number of dose levels required to identify the MTD. Approximately, 100 evaluable patients will participate in this study.

#### 4.2. Dose Escalation Schedule.

Doxorubicin will be given at 50 mg/m<sup>2</sup> as an i.v. bolus on Day 1 q3wk, which corresponds to 100% of its actual RD when combined with other myelosuppressive agents. It will not be escalated in this study.

The starting dose (DL1) for PM01183 will be 3.5 mg given as FD on Day 1 q3wk, which corresponds to 50% of the RD for this schedule when given as single agent.

The dose escalation schedule is summarized in the following table:

| Dosc escaration senedate recitor 111 | Dose of | escalation | schedu | le (co | hort A` | ١. |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

| DL | No. of patients | Relative DI (%) of<br>doxorubicin /<br>PM01183 | Dose of doxorubicin<br>(mg/m²) / PM01183 (mg FD)<br>on Day 1 q3wk |
|---|---|---|---|
| DL-1 | 0-6 | 100 / 42.85 | 50 / 3.0 |
| DL1 | 3-6 | 100 / 50 | 50 / 3.5 |
| DL2 | 3-6 | 100 / 71.4 | 50 / 5.0 |
| DL3 | 3-6 | 100 / 85.7 | 50 / 6.0 |
| DL4 | 3-6 | 100 / 100 | 50 / 7.0 |

The DL-1 level is to be explored only if DL1 is defined as the MTD.

DI, dose intensity; DL, dose level; FD, flat dose.

According to the toxicity observed, intermediate dose levels may be explored if considered appropriate by the investigators and the Sponsor.

Intra-patient dose escalation will not be allowed under any circumstances.

## New cohort (cohort B) after implementation of protocol amendment #3 (Cohort B):

Patients with SCLC and endometrial cancer will consecutively receive the following on Day 1 q3wk (three weeks = one treatment cycle):

- Doxorubicin: i.v. bolus/short infusion at a dose of 40 mg/m<sup>2</sup>, administered as described above, immediately followed by:
- PM01183: i.v. infusion over one hour at a dose of 2.0 mg/m<sup>2</sup>, administered as described above.

Both doxorubicin and PM01183 doses will be capped at 2.0 m<sup>2</sup> of BSA for individuals exceeding this BSA value. Doses will have to be recalculated for patients showing a  $\geq$  10% change in total body weight value compared to previous cycle.

PM01183 doses will be rounded to the first decimal, if necessary. Doxorubicin doses will be rounded according to institutional guidelines/standard practices.

## 5. Population and Endpoints.

Patients must fulfill all the inclusion/exclusion criteria to be eligible for admission to the study. See clinical trial protocol, sections 4.1 Inclusion Criteria and 4.2 Exclusion Criteria.

## 5.1. Patient Evaluability Criteria.

The analysis sets are defined as follows:

The "All Included Patients" analysis set is defined as all patients who are included in the study, regardless of whether they have received any study drug or not.

The "All Treated Patients" analysis set is defined as all included patients who have received at least part of one infusion of PM01183.

The "All Evaluable Patients for the Assessment of the Primary Endpoint" analysis set is defined as all included patients who have received at least one complete cycle (including observation period), except if early discontinuations or missed doses or delays and/or assessments were the consequence of drug-related toxicity (excluding hypersensitivity reactions and/or extravasations).

The "All Evaluable for Efficacy Patients" analysis set is defined as all evaluable patients measured according to the RECIST v.1.1 at least six weeks after treatment initiation in all patients with measurable disease, and/or by CA-125 levels if applicable, i.e. ovarian cancer with at least 2 x upper limit of normal (ULN) at baseline [according to the Gynecologic Cancer Intergroup (GCIG/Rustin) specific criteria]. No serum markers will be evaluated in patients with SCLC and endometrial cancer included in the new cohort B.

If early progression occurs (i.e., before six weeks since treatment) or if treatment should be discontinued due to any treatment-related toxicity before appropriate tumor assessments have been performed, the patient's objective response will be considered as a treatment failure or progressive disease (PD); therefore, their data will be included in the analysis of objective response as per RECIST v.1.1.

In the new cohort B of patients with SCLC and endometrial cancer, a patient evaluable for efficacy should have received at least one complete cycle (including observation period) and be evaluable as per RECIST, except if non-evaluability is due to treatment failure such as drug-related toxicity, death or early unequivocal PD outside the central nervous system.

All analyses will be performed as per protocol rather than on an intention-to-treat-basis. Any departure from the planned treatment according to the study schedule will be listed and documented in the clinical study report.

## 5.2. Endpoints.

#### 5.2.1. Primary Endpoint.

- The MTD will be the lowest dose level explored during the dose escalation at which more than one evaluable patient experience a DLT in Cycle 1.
- The RD will be the highest dose level explored in which less than one third of evaluable patients experience a DLT during Cycle 1.

If the DLTs of the doxorubicin and PM01183 combination without G-CSF prophylaxis are exclusively related to neutropenia, the MTD and RD will also be determined with primary G-CSF prophylaxis.

#### 5.2.1.1. Determination of MTD and RD.

A minimum of three patients will be included at each dose level. If no patients experience a DLT during the first cycle, the dose will be escalated. If one of three patients experiences a DLT, three additional patients will be included at that level. If >1 evaluable patient during dose escalation at a given dose level experience a DLT during the first cycle, that level will be considered the MTD and dose escalation will be terminated except if all DLTs occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than 7 days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis The DL immediately below the MTD, or DL4 if the MTD is not reached during dose escalation and the last dose level (DL4) is reached, was to be initially expanded up to a minimum of nine evaluable patients. If less than three among the first nine evaluable patients treated within the expansion cohort experience a DLT during Cycle 1 this DL will be the RD.

Further to the finding of encouraging antitumor activity in the first 43 evaluable patients (13 responses, including four complete responses, with five partial responses in eight patients with SCLC, and one complete and one partial response in three patients with endometrial cancer), expansion of the cohort treated at the RD has been increased to include approximately 30 additional patients, for a total of around 39 patients.

Determination of the maximum tolerated dose.

| No. of patients<br>evaluable*<br>for DLT | No. of patients<br>with DLTs<br>in Cycle 1 | Action |
|---|---|---|
| | 0 | Escalate DL until DL4 is reached |
| 3 | 1 | Add 3 patients |
| | >1 | MTD |
| 6 | 1 | Escalate DL until DL4 is reached |
| U | >1 | MTD |

DL, dose level; DLT, dose-limiting toxicities; MTD, maximum tolerated dose.

Decisions on delayed-onset DLTs (i.e., those DLTs occurring after Cycle 1) will be individually discussed between the Investigators and Sponsor, and might end affecting the definition of the proposed RD for phase II clinical trials.

In the new cohort B of patients with SCLC and endometrial cancer, a patient evaluable for efficacy should have received at least one complete cycle (including observation period) and be evaluable as per RECIST, except if non-evaluability is due to treatment failure such as drug-related toxicity, death or early unequivocal PD outside the central nervous system.

<sup>\*</sup> Patients not evaluable for DLT during dose optimization must be replaced.

<sup>\*\*</sup> For replacement of patients and replacement of patients after implementation of Amendment #3 (see Protocol section 5.3).

#### 5.2.1.2. DLT Criteria.

DLTs are defined as adverse events (AEs) and laboratory abnormalities related to the study treatment during the first cycle of treatment and fulfilling at least one of the criteria outlined below.

- Grade 4 neutropenia [absolute neutrophil count (ANC)  $< 0.5 \times 10^9 / l$ ] lasting > 7 days.
- Grade  $\geq$  3 febrile neutropenia of any duration or neutropenic sepsis.
- Grade 4 thrombocytopenia (platelet count  $< 25 \times 10^9/l$ ) or grade 3 with any major bleeding episode requiring a platelet transfusion.
- Grade 4 alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) increase, or grade 3 lasting > 14 days.
- Treatment-related grade  $\geq 2$  ALT or AST increase concomitantly with  $\geq 2$  xULN total bilirubin increase and normal alkaline phosphatase (AP).
- Grade  $\geq$  3 creatine phosphokinase (CPK) increase.
- Any other grade 3/4 non-hematological AE that is suspected to be related to study drug(s), except nausea/vomiting (unless the patient is receiving an optimal anti-emetic regimen), hypersensitivity reactions, extravasations, grade 3 asthenia lasting less than one week, and non-clinically relevant isolated biochemical abnormalities [e.g., isolated increase in gamma-glutamyltransferase (GGT)]. In any case, the clinical relevance should be discussed between the Investigators and Sponsor's representatives.
- Delay in the administration of Cycle 2 of the combination exceeding 15 days of the theoretical date (i.e., Day 22), due to any AEs related to study drug(s).
- The following circumstances will be discussed between the Principal Investigator and the Sponsor, and the final consensus will be documented:
  - o DLTs with delayed onset (i.e., that occur after Cycle 1).

#### 5.2.2. Secondary Endpoints.

#### 5.2.2.1. Safety.

Safety parameters include:

- Adverse events.
- Hematology.
- Clinical chemistry.
- Coagulation tests.
- Vital signs.
- Electrocardiogram (ECG) and Left Ventricular Ejection Fraction (LVEF).
- Physical examinations.
- Delays and reductions.
- Withdrawals.

AEs will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4 and coded using the Medical Dictionary for Regulatory Activities (MedDRA).

#### **5.2.2.2.** Efficacy.

Although it is not the main objective of this study, antitumor activity will be measured according to the RECIST v.1.1 at least six weeks after treatment initiation in all patients with measurable disease, or by evaluation of tumor markers if applicable (e.g., ovarian cancer). Patients included at the RD in the expansion cohort must be evaluable per RECIST v.1.1 or by evaluation of tumor markers (see Section 7.4 for efficacy evaluation).

No serum markers will be evaluated in patients with SCLC and endometrial cancer included in the new cohort B.

If any particular tumor type is adequately represented, time-related parameters [i.e., progression-free survival (PFS), overall survival (OS)] will be analyzed according to the Kaplan-Meier method, if appropriate.

In the new cohort B, exploratory assessment for progression-free survival (PFS) and overall survival (OS) will be performed.

The best overall response is defined as the best response achieved during the study according to RECIST v.1.1 and/or GCIG, whenever is applicable, before disease progression, administration of subsequent anticancer treatment or study discontinuation.

The response rate is defined as the ratio of patients with any response [complete response (CR) or partial response (PR)] by the total number of patients included in the efficacy population. The number of patients with stable disease  $SD \ge 3$  and/or 4 months will also be shown.

Duration of response (DR), defined as the time between the date when the response criteria (PR or CR, the first that is reached) are fulfilled and the first date when disease progression, recurrence or death is objectively documented (taking the smallest measurements documented since the treatment started as reference for progressive disease).

Progression-free survival (PFS), defined as the time from the first day of study treatment to the day of negative assessment (progression or death) or last tumor evaluation.

In addition, patients with SCLC and endometrial cancer included in the cohort B will be followed for survival for up to 18 months after the first study dose.

#### 5.2.2.3. Pharmacokinetics.

Pharmacokinetic (PK) analyses will be described and reported in a different document out of the scope of this SAP.

### 5.2.2.4. Pharmacogenomics.

Pharmacogenomic (PGx) analyses will be described and reported in a different document out of the scope of this SAP.

## 6. General analysis methods.

#### 6.1. Statistical Software.

Oracle Clinical will be used for double data entry and clinical data management.

SAS® Software v.9.2 or higher will be used for all statistical analyses.

## 6.2. Data Analysis Conventions.

All data analysis conventions, derived data calculations and grouping needed to perform the statistical analysis will come in separate document not included in this SAP.

## 7. Statistical analysis.

## 7.1. Patient Disposition and Protocol Deviations.

Patients and dose levels will be summarized and listed by the populations used in the study:

- All Included Patients.
- All Treated Patients.
- All Evaluable Patients for the Assessment of the Primary Endpoint.
- All Evaluable for Efficacy Patients.

Reasons for not belonging to any population will be detailed.

The accrual and study discontinuation details will be presented descriptively.

Reasons for treatment discontinuation by number of cycles received will be described by counts and percentages. Reasons of treatment discontinuation other than disease progression will be detailed.

A protocol deviation is defined as any departure from what is described in the protocol of a clinical trial approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and Competent Authorities. Therefore, it applies to deviations related to patient inclusion and clinical procedures (e.g., assessments to be conducted or parameters to be

determined), and also to other procedures described in the protocol that concern the Good Clinical Practice (GCP) guidelines or ethical issues (e.g., issues related to obtaining the patients' Informed Consent, data reporting, the responsibilities of the Investigator, etc.).

Protocol deviations will be categorized by the PharmaMar's responsible physician and summarized for all patients. A summary table with the number of patients with inclusion/exclusion deviations will be presented per criterion. These patients will be listed with the unmet criteria. Deviations with no effects on the risk/benefit ratio of the clinical trial (such as minimal delays in assessments or visits) will be distinguished from those that might have an effect on this risk/benefit ratio.

A summary including but not necessarily restricted to the following categories will be presented:

- Ineligible patients as per protocol.
- Patient not withdrawn as per protocol.
- Excluded concomitant medication.
- Incorrect dose or schedule, including patients not meeting re-treatment criteria on Day 1 of subsequent cycles.

#### 7.2. Baseline Characteristics.

#### 7.2.1. Demographics.

Demographics and baseline characteristics will be summarized for all treated patients. All patient characteristics will be described by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable).

Continuous variables will be summarized and presented with summary statistics, i.e., mean, median, range and standard deviation.

Categorical variables will be summarized in frequency tables. Percentages in the summary tables will be rounded and may therefore not always add up to exactly 100%.

In case of pre-treatment characteristics with multiple measurements per patient before the start of treatment (laboratory assessments, vital signs), the baseline measurement will be considered the last value prior to or on the first day of treatment.

Baseline Eastern Cooperative Oncology Group (ECOG) performance status will be summarized with frequency counts.

For the cancer history, histologic diagnosis, time from diagnosis, number of baseline lesions, and involvement in the different sites will be summarized. Time from initial diagnosis to the start of study treatment and time from the latest disease progression to the start of study treatment will be calculated in months and summarized descriptively. If incomplete dates are recorded, the rules described in section 8.5 will be used for imputation.

The primary tumor sites and baseline lesions will be recoded by PharmaMar's physicians in order to categorize them accurately in the analysis.

The previous relevant medical history (other than cancer) will be listed by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable) and patient.

A frequency tabulation of the different types of previous oncologic surgery (excluding only diagnostic or palliative procedures), radiotherapy, or anticancer systemic therapy (number of lines for advanced and number of agents) will be given. Chemotherapy agents and lines will be recoded by PharmaMar's physicians in order to categorize them accurately in the analysis.

The signs and symptoms, hematology and serum biochemistry abnormalities at baseline will be displayed by tabulation of frequencies according to NCI-CTCAE v.4.0 toxicity grades. The signs and symptoms and laboratory abnormalities of grade ≥2 at baseline will be listed by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable) and patient.

## 7.3. Statistical Analysis for Safety.

All analysis of safety variables will be descriptive. Data retrieved at both scheduled and unscheduled visits will be tabulated and listed.

The safety population is composed by all patients that receive at least part of a PM01183 infusion. The safety patient population will be used for the general safety presentations.

The "All Evaluable Patients for the Assessment of the Primary Endpoint" population will be used for primary analysis.

For the evaluation of the main endpoint, the total number of patients included, the number of patients evaluable for determination of DLTs, and the number of patients with any DLT (and their categorization) will be summarized by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable). The toxicities meeting the DLT criteria in Cycle 1 and toxicities in subsequent cycles, if any, will be listed separately, and the description of laboratory abnormalities (hematology/ biochemistry) will be supported by graphs depicting the evolution in time of laboratory values (including nadir calculation and median time to recovery from baseline values).

#### 7.3.1. Treatment Administration and Exposure.

Exposure to each treatment will be described by dose level (or most adequate dose grouping/cohort/tumor type or other clinical relevant variable) for all patients who have received at least one of the study treatments.

<u>Total cumulative dose</u>, expressed in mg for PM01183 and in mg for doxorubicin and defined as the sum of all the product doses from the 1<sup>st</sup> dose received until the last dose received.

<u>Intended dose intensity</u> is the planned dose of the cycle divided by planned duration of a cycle in weeks.

<u>Absolute dose intensity</u>: is the total cumulative dose divided by the duration of the treatment. As a convention, the duration of the last cycle is considered to be 21 days (planed cycle duration).

<u>Relative dose intensity (%)</u>: is the ratio of absolute dose intensity divided by the intended dose intensity.

<u>Time on treatment:</u> is the interval expressed in weeks, between the first infusion date and the last infusion date plus 30 days or start of new treatment or date of death (whichever occurs first).

The number of cases, median, standard deviations, 95% confidence interval (CI), minimum and maximum values for the parameters defined above will be tabulated by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable) and drug (PM01183 and doxorubicin).

#### 7.3.2. Cycle Delays and Omissions.

The item "Infusion delayed: No/Yes" in the case report from (CRF) will be used to calculate the delay. For doses considered as delayed by the investigator, the delay will be calculated as:

Delay (in days) will be equal to the date of start of current cycle minus the date of start of previous cycle minus 21 days (planed cycle duration, in days).

Dose delay is defined by a delay in the administration of the first infusion of one cycle (Day 1 infusion).

Cycle 1 will be excluded from all calculations of cycle delay (and the denominator used for calculations will be equal to the number of cycles susceptible to be delayed).

The distribution of delays according to the infusion administered will be studied by means of counts and percentages. The reasons for infusion delay will be detailed, specifying how many were due to treatment-related toxicity and how many were not (administrative reasons will be analyzed separately and additional tables will be prepared after exclusion of these delays). Within delays attributable to treatment, hematological and/or non-hematological reasons will be outlined, and the specific reasons will be detailed, if possible.

Skipped dose or dose omission is defined as every doxorubicin infusion not administrated on Day 1 of the cycle. The distribution of skipped doses will be studied by means of counts and percentages (the denominator used for calculations will be equal to the number of patients/cycles susceptible to have an omission) and a detailed listing of patients with skipped dose and reason will be showed. Also reasons for dose omission will be detailed, specifying how many were due to treatment, how many were not and how many reached a maximal total cumulative dose of 450 mg/m<sup>2</sup>.

All cycles in which a maximal total cumulative dose of 450 mg/m<sup>2</sup> is not reached are susceptible of doxorubicin omission (the denominator used for calculations will be equal to the number of cycles susceptible to be omitted).

#### 7.3.3. Dose Reductions.

All dose reductions will be considered and described (per cycle and patient), specifying the magnitude and the reason(s) for reduction treatment-related (hematological toxicity, non-hematological toxicity or both), or if any, other causes unrelated to treatment.

#### 7.3.4. Adverse Events.

All adverse events will be coded using the MedDRA coding dictionary.

The toxicity evaluation will be made according to the National Cancer Institute- Common Toxicity Criteria (NCI-CTCAE) v.4 and the events will be coded and classified using the MedDRA dictionary.

As far as all the toxicities are concerned, the NCI-CTCAE grade will be used wherever an NCI-CTCAE grading exists. Otherwise, the severity will be noted. As a convention, the term "Grade" will always be used. Toxicities will be described according to the worst NCI-CTCAE grade or, for toxicities which do not form the subject of NCI-CTCAE classification, according to the worst severity.

Descriptive statistics will be used for the evaluation of safety. The incidence and grade of adverse events and laboratory abnormalities will be calculated considering the most severe grade per patient and cycle and will be displayed in frequency tables using counts and percentages.

The shift of severity grades from baseline to the worst occurrence during treatment will be tabulated.

Deaths, serious adverse events and events resulting in study discontinuation will be tabulated.

Additional safety analyses may be determined at any time, in order to most clearly enumerate rates of toxicities and to further define the safety profile of PM01183 in combination with doxorubicin. In order to categorize accurately the safety information, additional classifications other than system organ class (SOC)/preferred term (PT) could be populated in order to understand better the safety drug profile.

## 7.3.5. Serious Adverse Events (SAEs).

Database listings of deaths and serious adverse events will be provided, including at least date of onset and resolution (if applicable), severity, relationship to study drug, most important significant consequence and main action taken.

#### 7.3.6. Laboratory Evaluations.

#### **7.3.6.1.** Hematology.

Hematological toxicities classified according to the NCI-CTCAE v.4 will be calculated in all cycles by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable). Separate analyses will be carried out for the first cycle of treatment. The worst grade reached by each patient during treatment and Cycle 1 will also be determinated.

If serious toxicities occur, a special follow-up will be done to determine the pattern of thrombocytopenia and neutropenia within and between the different cycles. This follow-up will include the calculation of median and the range of nadir values and of the median time to recovery to baseline values and also descriptive tables.

If appropriate, these tables might be complemented with graphic representations of the nadir of neutrophil and platelets count by cycle during treatment by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable). Furthermore, graphs of the inter-cycle time course of neutropenia, thrombocytopenia or any other considered

parameter will be provided. If applicable, graphs comparing the time course of these parameters during the first and second cycles will be created.

### 7.3.6.2. Serum Biochemistry and Coagulation Tests.

The non-hematological laboratory abnormalities (i.e., NCI-CTCAE grades) of transaminases, creatinine, CPK, bilirubin, AP, etc. will be calculated by patient and cycle as explained for hematological toxicities. Separate analyses will be carried out for the first cycle of treatment. The worst grade reached by each patient during treatment and Cycle 1 will also be calculated.

If serious toxicities occur, a special follow-up that will include calculation of median and range of peak values and of median time to recovery to baseline values and, together with descriptive tables will be done to determine the pattern of these toxicities within and between cycles.

If appropriate, these tables might be complemented with boxplots for the peaks of transaminases, creatinine, CPK, bilirubin, AP, etc. by cycle along the treatment by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable). Furthermore, graphs of the inter-cycle time course of any considered parameter will be provided. If applicable, graphs comparing the time course during the first and second cycles will be created.

### 7.3.7. Physical Examination.

The evaluation of physical examination (i.e., normal/abnormal) will be summarized with frequency counts. All data will be listed by dose level (or most adequate dose grouping/cohort/Tumor type or other clinical relevant variable).

#### 7.3.8. ECG/LVEF.

Baseline ECG evaluation (normal/abnormal) will be summarized with frequency counts.

Continuous variables (PR Interval, QT Interval, QRS Complex, Ventricular Rate, LVEF and LVEF Normal Range) will be summarized and summary statistics will be provided (i.e., mean, standard deviation, median and range). Baseline values and their evolution during treatment will be tabulated with summary statistics.

$$QTcF = \frac{QT}{\sqrt[3]{RR}}$$

QTcF (Fridericia's formula) will be graded using the NCI-CTCAE v.4

#### 7.3.9. Vital Signs.

PS and weight gain / loss during the study will be summarized by frequency tabulation.

#### 7.3.10. Concomitant Medication.

Concomitant therapies will be coded using the World Health Organization Anatomical Therapeutic Chemical (WHO-ATC) classification system dictionary and categorized according to the ATC (levels 1, 2 and 4) class. The number of patients receiving each type of therapy will be tabulated in two separated frequency tables: one for therapies that started prestudy, and for those administrated during the study. The accompanying listing will include all concomitant therapies.

Additional listings for patients taking prohibited medications / therapies according to protocol will be provided.

## 7.4. Statistical analysis for efficacy.

#### 7.4.1. Exploratory Analysis of Antitumor Activity.

The "All Evaluable for Efficacy Patients" population will be used for the analysis of the efficacy and also "All Treated Patients" population will be used for the overall response analysis.

Response rates will be characterized using descriptive statistics (95% confidence interval). If applicable, overall response rate (percentage of patients with PR or CR), percentages for PR or CR separately and percentage of patients with  $SD \ge 4$  months will be analyzed.

Time-related parameters (DR and PFS) will be analyzed according to the Kaplan-Meier methodology, if applicable.

The characteristics of the patients achieving an objective response or  $SD \ge 4$  months by RECIST v.1.1, or a clinically significant improvement measured by tumor markers, will be displayed.

In addition, patients with SCLC and endometrial cancer included in the new cohort B will be followed for survival for up to 18 months after the first study dose.

### 7.4.2. Level of Significance.

Confidence intervals will be constructed using the 95% level. No formal statistical tests are defined, but if needed, all will be done at a significance level of 5% and will be considered exploratory.

## 8. Other statistical analysis.

## 8.1. Stratification and Covariate Analysis.

No stratification by prognostic factors or tumor types is planned. If a disease is adequately represented, response rates might be analyzed descriptively, and time-related parameters might be analyzed according to the Kaplan-Meier method. Efficacy parameters could also be subjected to further analysis (if appropriate), considering correlation with factors of known prognostic value such as patient ECOG performance status at entry, disease burden, prior therapies, other disease-specific known prognostic factor, or population characteristics, etc. using the appropriate test (Fisher's exact test, Spearman test, etc.).

## 8.2. Multivariate Analysis.

Exploratory *Cox* regression for multivariate analysis will be used for time-dependent efficacy parameters, and logistic regression for the evaluation of covariates associated with best overall response, if appropriate.

## 8.3. Subgroup Analysis.

If any cancer subtype or any other baseline characteristics of patients are adequately represented, a separate analysis by tumor type and efficacy as per RECIST v.1.1, will be performed.

If there is a representative number of patients who receive a maximal total cumulative dose of 450 mg/m<sup>2</sup> of doxorubicin and continue treatment with PM01183 alone, a separate analysis will be performed and tables, listings and graphic representations for this population will be provided when applicable.

## 8.4. Interim Analysis.

Non-scheduled interim analyses might be performed exclusively for enhancing patient's safety.

## **8.5.Missing Values Management.**

Missing laboratory values will be subtracted from the denominator of the tables.

#### Imputation of incomplete dates

#### Dates before randomization

If the day of a date is unknown, the imputed day will be 15. If the month is also unknown, the imputed date will 01/July/year. This assumption will be valid if the imputed date is earlier than the informed consent's date; otherwise the imputed date will be the first day of the informed consent's month date (i.e., 01/ informed consent's month date/year).

## Dates after end of treatment

To ensure the most conservative approach for the efficacy time-to-event variables (i.e., PFS) that can be affected by missing values the following rules will be implemented: if the day of a date is unknown, then the imputed day will be 01; if the month is also unknown, then the imputed date will be 01/July/year. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise, the imputed date will be the last drug administration date plus the planed cycle duration (21 days) or the last day of the reported month, whichever occurs first.

#### 8.6. Decimals Places.

By default, all numeric results will be rounded to one decimal, except in the case where variables are integer; in that case, they will be reported without decimals, for example, age in years, number of sites, etc.

## 9. Tables, Listings and Figures.

After the implementation of protocol amendment #3, a new cohort B of patients with SCLC and endometrial cancer has been included. All statistical outputs will be displayed according to dose level (grouped)/cohort/tumor type or primary site/ CSF use or not/other relevant clinical variable, whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

If the number of categories or items would not yield appropriate tabular or graphic representations, detailed listings will be shown instead.

The abbreviation DL shown in the mock tables might refer to dose level (grouped <RD, RD, etc...)/cohort (i.e. Cohort A and B)/tumor type or primary site (i.e. Ovarian, SCLC (2nd line), etc...)/CSF use or not/other clinical relevant variable). The following is a list of tables, listings and figures that will be produced:

| Table 10.1.1.1 Patient Accrual by Institution and Dose Level | 34 |
|---|---|
| Table 10.1.1.2 Disposition of Patients | 34 |
| Table 10.1.1.3 Time on Treatment by Dose Level | 34 |
| Table 10.1.1.4 Number of Patients Evaluable for Analysis | 34 |
| Table 10.1.1.5 Listing of Not Evaluable Patients | 34 |
| Table 10.1.2.1 Treatment Discontinuation by Dose Level* | 35 |
| Table 10.1.2.2 Treatment Discontinuation Details | 35 |
| Table 10.1.2.3 Reasons for Treatment Discontinuations by Cycle and Dose Level | 35 |
| Table 10.1.2.4 Listing of patients with Discontinuation with PM01183 alone | 35 |

| Table 10.1.2.6 Reasons for Treatment Discontinuation Other than Progressive Disease. 36 Table 10.1.2.7 Reasons for Study Discontinuation by Dose Level. 36 Table 10.1.3.1 Supportive Listing Relevant Protocol Deviations. 36 Table 10.2.1.1 Age at Entry by Dose Level. 36 Table 10.2.1.2 Age Median and Range by Dose Level. 37 Table 10.2.1.3 Gender by Dose Level. 37 Table 10.2.1.4 Race by Dose Level. 37 Table 10.2.1.5 Pregnancy Tests by Dose Level. 37 Table 10.2.1.6 Physical Examination Result by Dose Level. 37 Table 10.2.1.7 Physical Examination Parameters by Dose Level. 38 Table 10.2.1.8 ECOG Performance Status by Dose Level at Baseline. 38 Table 10.2.1.9 Vital Signs Parameters by Dose Level. 38 Table 10.2.1.10 ECG Result by Dose Level. 38 Table 10.2.1.11 ECG Parameters by Dose Level. 39 Table 10.2.1.12 Median LVEF for Patients with Previous Treatment with Anthracyclines by Dose Level. 40 Table 10.2.2.1 Time from Diagnosis to First Infusion. 46 Table 10.2.2.2 Time from last PD to First Infusion. 46 Table 10.2.2.3 TrP of Last Prior Therapy. 46 Table 10.2.2.4 Tumor type by Dose Level. 41 Table 10.2.3.5 Summary of Cancer History per Patient and Tumor type. 41 Table 10.2.3.5 Summary Statistics. No of Sites Involved by Tumor type Dose Level. 41 Table 10.2.3.5 Bulky disease by Tumor type and Dose Level. 41 Table 10.2.3.5 Bulky disease by Tumor type and Dose Level. 42 Table 10.2.3.6 Median sum of diameter of target lesions (mm). 42 Table 10.2.3.7 Previous Treatment Summary by Dose Level. 42 Table 10.2.3.8 Previous Systemic Therapy by Dose Level. 42 Table 10.2.4.1 Previous Radiotherapy by Dose Level (Curative/Palliative). 42 Table 10.2.5.1 Previous Radiotherapy by Dose Level (Curative/Palliative). 43 Table 10.2.6.1 Previous Radiotherapy by Dose Level (Curative/Palliative). 43 Table 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1 & 4) by Dose Level/Tumor type. 41 | Table 10.1.2.5 Treatment Discontinuation Due to Adverse Events | 36 |
|---|---|---|
| Table 10.1.3.1 Supportive Listing Relevant Protocol Deviations | Table 10.1.2.6 Reasons for Treatment Discontinuation Other than Progressive Disease. | 36 |
| Table 10.2.1.1 Age at Entry by Dose Level. 36 Table 10.2.1.2 Age Median and Range by Dose Level. 37 Table 10.2.1.3 Gender by Dose Level. 37 Table 10.2.1.4 Race by Dose Level. 37 Table 10.2.1.5 Pregnancy Tests by Dose Level. 37 Table 10.2.1.6 Physical Examination Result by Dose Level. 38 Table 10.2.1.7 Physical Examination Parameters by Dose Level. 38 Table 10.2.1.8 ECOG Performance Status by Dose Level at Baseline. 38 Table 10.2.1.9 Vital Signs Parameters by Dose Level. 38 Table 10.2.1.10 ECG Result by Dose Level. 35 Table 10.2.1.11 ECG Parameters by Dose Level. 35 Table 10.2.1.12 Median LVEF for Patients with Previous Treatment with Anthracyclines by Dose Level. 40 Table 10.2.2.1 Time from Diagnosis to First Infusion. 40 Table 10.2.2.2 Time from last PD to First Infusion. 40 Table 10.2.2.3 TTP of Last Prior Therapy. 40 Table 10.2.2.3 Two of Sites Involved by Tumor type and Dose Level. 41 Table 10.2.3.1 No of Sites Involved by Tumor type and Dose Level. 41 Table 10.2.3.2 Summary Statistics. No of Sites Involved by Tumor type Dose Level. 42 Table 10.2.3.3 Frequency of Patients Classified by Sites Involved by Tumor ty | Table 10.1.2.7 Reasons for Study Discontinuation by Dose Level | 36 |
| Table 10.2.1.1 Age at Entry by Dose Level. 36 Table 10.2.1.2 Age Median and Range by Dose Level. 37 Table 10.2.1.3 Gender by Dose Level. 37 Table 10.2.1.4 Race by Dose Level. 37 Table 10.2.1.5 Pregnancy Tests by Dose Level. 37 Table 10.2.1.6 Physical Examination Result by Dose Level. 38 Table 10.2.1.7 Physical Examination Parameters by Dose Level. 38 Table 10.2.1.8 ECOG Performance Status by Dose Level at Baseline. 38 Table 10.2.1.9 Vital Signs Parameters by Dose Level. 38 Table 10.2.1.10 ECG Result by Dose Level. 35 Table 10.2.1.11 ECG Parameters by Dose Level. 35 Table 10.2.1.12 Median LVEF for Patients with Previous Treatment with Anthracyclines by Dose Level. 40 Table 10.2.2.1 Time from Diagnosis to First Infusion. 40 Table 10.2.2.2 Time from last PD to First Infusion. 40 Table 10.2.2.3 TTP of Last Prior Therapy. 40 Table 10.2.2.3 Two of Sites Involved by Tumor type and Dose Level. 41 Table 10.2.3.1 No of Sites Involved by Tumor type and Dose Level. 41 Table 10.2.3.2 Summary Statistics. No of Sites Involved by Tumor type Dose Level. 42 Table 10.2.3.3 Frequency of Patients Classified by Sites Involved by Tumor ty | Table 10.1.3.1 Supportive Listing Relevant Protocol Deviations | 36 |
| Table 10.2.1.2 Age Median and Range by Dose Level | | |
| Table 10.2.1.4 Race by Dose Level | Table 10.2.1.2 Age Median and Range by Dose Level | 37 |
| Table 10.2.1.5 Pregnancy Tests by Dose Level | Table 10.2.1.3 Gender by Dose Level | 37 |
| Table 10.2.1.6 Physical Examination Result by Dose Level | Table 10.2.1.4 Race by Dose Level | 37 |
| Table 10.2.1.6 Physical Examination Result by Dose Level | Table 10.2.1.5 Pregnancy Tests by Dose Level | 37 |
| Table 10.2.1.7 Physical Examination Parameters by Dose Level | | |
| Table 10.2.1.8 ECOG Performance Status by Dose Level at Baseline | | |
| Table 10.2.1.10 ECG Result by Dose Level | | |
| Table 10.2.1.11 ECG Parameters by Dose Level | Table 10.2.1.9 Vital Signs Parameters by Dose Level | 38 |
| Table 10.2.1.12 Median LVEF for Patients with Previous Treatment with Anthracyclines by Dose Level | Table 10.2.1.10 ECG Result by Dose Level | 39 |
| by Dose Level | Table 10.2.1.11 ECG Parameters by Dose Level | 39 |
| Table 10.2.2.1 Time from Diagnosis to First Infusion | | |
| Table 10.2.2.3 TTP of Last Prior Therapy | Table 10.2.2.1 Time from Diagnosis to First Infusion | 40 |
| Table 10.2.2.3 TTP of Last Prior Therapy | Table 10.2.2.2 Time from last PD to First Infusion | 40 |
| Table 10.2.2.5 Summary of Cancer History per Patient and Tumor type | | |
| Table 10.2.3.1 No of Sites Involved by Tumor type and Dose Level | Table 10.2.2.4 Tumor type by Dose Level | 41 |
| Table 10.2.3.2 Summary Statistics. No of Sites Involved by Tumor type Dose Level | Table 10.2.2.5 Summary of Cancer History per Patient and Tumor type | 41 |
| Table 10.2.3.3 Frequency of Patients Classified by Sites Involved by Tumor type and Dose Level | Table 10.2.3.1 No of Sites Involved by Tumor type and Dose Level | 41 |
| Level | Table 10.2.3.2 Summary Statistics. No of Sites Involved by Tumor type Dose Level | 41 |
| Table 10.2.3.4 Listing of Sites per Patient.42Table 10.2.3.5 Bulky disease by Tumor type and Dose Level.42Table 10.2.3.6 Median sum of diameter of target lesions (mm).42Table 10.2.4.1 Previous Treatment Summary by Dose Level.42Table 10.2.4.2 Previous Systemic Therapy by Dose Level/Tumor type.42Table 10.2.5.1 Previous Surgery by Dose Level (Curative/Palliative).43Table 10.2.6.1 Previous Radiotherapy by Dose Level.43Table 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1 & 4) by Dose | | |
| Table 10.2.3.6 Median sum of diameter of target lesions (mm).42Table 10.2.4.1 Previous Treatment Summary by Dose Level.42Table 10.2.4.2 Previous Systemic Therapy by Dose Level/Tumor type.42Table 10.2.5.1 Previous Surgery by Dose Level (Curative/Palliative).43Table 10.2.6.1 Previous Radiotherapy by Dose Level.43Table 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1 & 4) by Dose | | |
| Table 10.2.4.1 Previous Treatment Summary by Dose Level.42Table 10.2.4.2 Previous Systemic Therapy by Dose Level/Tumor type.42Table 10.2.5.1 Previous Surgery by Dose Level (Curative/Palliative).43Table 10.2.6.1 Previous Radiotherapy by Dose Level.43Table 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1 & 4) by Dose | Table 10.2.3.5 Bulky disease by Tumor type and Dose Level | 42 |
| Table 10.2.4.1 Previous Treatment Summary by Dose Level.42Table 10.2.4.2 Previous Systemic Therapy by Dose Level/Tumor type.42Table 10.2.5.1 Previous Surgery by Dose Level (Curative/Palliative).43Table 10.2.6.1 Previous Radiotherapy by Dose Level.43Table 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1 & 4) by Dose | Table 10.2.3.6 Median sum of diameter of target lesions (mm) | 42 |
| Table 10.2.5.1 Previous Surgery by Dose Level (Curative/Palliative) | Table 10.2.4.1 Previous Treatment Summary by Dose Level | 42 |
| Table 10.2.5.1 Previous Surgery by Dose Level (Curative/Palliative) | | |
| Table 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1 & 4) by Dose | | |
| | | 43 |

| Table 10.2.7.2 No of Lines of Prior Anticancer Therapy for Advanced Disease by Dose<br>Level/Tumor type4 |
|---|
| Table 10.2.7.3 Summary Statistics. No of Lines of Prior Anticancer Therapy by Dose<br>Level/Tumor type44 |
| Table 10.2.7.4 No of Agents of Prior Anticancer Therapy by Dose Level/Tumor type 4- |
| Table 10.2.7.5 No of Agents of Last Prior Anticancer Therapy before PM01183 treatment by Dose Level/Tumor type44 |
| Table 10.2.7.6 Summary Statistics. No of Agents of Prior Anticancer Therapy by Dose<br>Level/Tumor type4 |
| Table 10.2.7.7 Listing of Agents of Prior Anticancer Therapy by Dose Level4 |
| Table 10.2.7.8 Agents of Prior Anticancer Therapy by Dose Level/Tumor type4. |
| Table 10.2.7.9 CTFI by Dose Level/Cohort/Tumor type4 |
| Table 10.2.7.10 Summary Statistics: CTFI by Dose Level/Cohort/Tumor type4 |
| Table 10.2.7.11 Patients Previously Treated with Anthracyclines by Dose Level4 |
| Table 10.2.7.12 Summary Statistics: Cumulative Dose in Patients Previously Treated with Anthracyclines by Dose Level. 4: |
| Table 10.2.8.1 Hematological Abnormalities at Baseline by Dose Level40 |
| Table 10.2.8.2 Median and Range for Hematological Parameters at Baseline by Dose Level40 |
| Table 10.2.8.3 Supportive Listing: Patients with grade >1 Hematological Abnormalities at Baseline40 |
| Table 10.2.8.4 Patients with Missing Hematological Evaluations at Baseline40 |
| Table 10.2.9.1 Biochemical Abnormalities at Baseline by Dose Level4 |
| Table 10.2.9.2 Median and Range for Biochemical Parameters at Baseline by Dose Level. 4 |
| Table 10.2.9.3 Supportive Listing: Patients with Grade >1 Biochemical Abnormalities at Baseline4 |
| Table 10.2.9.4 Patients with Missing Biochemical Evaluations at Baseline4 |
| Table 10.2.10. 1 Coagulation Abnormalities at Baseline by Dose Level4 |
| Table 10.2.10. 2 Median and Range for Coagulation Parameters at Baseline by Dose Level |
| Table 10.2.10. 3 Supportive Listing: Patients with Grade >1 Coagulation Abnormalities at Baseline |
| Table 10.2.10. 4 Patients with Missing Coagulation Evaluations at Baseline48 |
| Table 10.2.11. 1 Metabolic Abnormalities at Baseline by Dose Level4 |
| Table 10.2.11. 2 Median and Range for Metabolic Parameters at Baseline by Dose Level. |
| ······································ |

| Table 10.2.11. 3 Supportive Listing: Patients with grade >1 Metabolic Ab Baseline | |
|---|---|
| Table 10.2.11. 4 Patients with Missing Metabolic Evaluations at Baseline | 49 |
| Table 10.2.12. 1 Signs and Symptoms by Dose Level | 49 |
| Table 10.2.12. 2 Listing of Adverse Events at Baseline Grade >1 | |
| Table 10.2.13. 1 Concomitant Medication Starting Pre-Study (ATC Level Dose Level | |
| Table 10.2.13. 2 Concomitant Medication Starting Pre-Study (RBC and Itransfusions/EPO) | |
| Table 10.2.13. 3 Supportive Listing: RBC and Platelet transfusions/EPO | (Pre-Study) 50 |
| Table 10.2.13. 4 No of patients with Opioids Treatment at Baseline by Dos | se Level50 |
| Table 10.2.13. 5 Median number of No of Opioids per patient by Dose Lev | el 50 |
| Table 10.2.13. 6 No of patients with Steroids treatment at baseline by dose | Level 50 |
| Table 10.2.13. 7 Known CYP 3A4 Inducers/Inhibitors/Substrates Concom<br>BL | - |
| Table 10.2.13. 8 Listing of CYP 3A4 Inducers/Inhibitors/Substrates Conce | |
| Table 11.1.1.1 No of Cycles Administered by Dose Level | 52 |
| Table 11.1.1.2 Median and Range of Cycles Administered by Dose Level. | 52 |
| Table 11.1.1.3 Cumulative Dose by Dose Level | |
| Table 11.1.1.4 Dose Intensity by Dose Level | 53 |
| Table 11.1.1.5 Relative Dose Intensity by Dose Level | 53 |
| Table 11.1.1.6 Drug Administration: Patients that Reached the Maximal of 450 mg/m <sup>2</sup> | |
| Table 11.1.2.1 No of Patients with Delayed Cycles by Dose Level | 54 |
| Table 11.1.2.2 No of Patients with Dose Delayed by Dose Level According | |
| Table 11.1.2.3 No of Cycles Delayed Per Patient by Dose Level | |
| Table 11.1.2.4 No of Cycles Delayed Per Patient by Dose Level. Summary | Statistics 54 |
| Table 11.1.2.5 Number of Cycles with Drug Related Delay per Patient by | Dose Level 55 |
| Table 11.1.2.6 Number of Cycles with Drug Related Delay per Patient by I Summary Statistics. | |
| Table 11.1.2.7 Length of Delay According to relationship by Dose Level. Statistics | |
| Table 11.1.2.8 Listing of Patient with Dose Delays | 56 |
| Table 11.1.2.9 Supportive Listing: Dose Delays Excluding Administrative | e Reasons 56 |

| Table 11.1.2.10 No. of Patients with Doxorubicin Omissions by Dose Level 56 |
|---|
| Table 11.1.2.11 No of Patients with Doxorubicin Cycles Omission by Dose Level 50 |
| Table 11.1.2.12 Listing of Doxorubicin Dose Omissions56 |
| Table 11.1.2.13 Listing of Cycles Delays due to Hematological Abnormalities56 |
| Table 11.1.2.14 Listing of Cycles Delays due to Non-Hematological Adverse Events 57 |
| Table 11.1.3.1 No of Patients with PM01183 Dose Reduction by Dose Level57 |
| Table 11.1.3.2 No of Patients with PM01183 Cycles Dose Reduction by Dose Level 57 |
| Table 11.1.3.3 Reasons for PM01183 Dose Reduction by Dose Level |
| Table 11.1.3.4 Listing of PM01183 Dose Reductions |
| Table 11.1.3.5 Listing of Dose Reductions due to Hematological Abnormalities58 |
| Table 11.1.3.6 Listing of Dose Reductions due to Non-Hematological Adverse Events 58 |
| Table 11.1.4. 1 Listing of Patients with Dose Interruption and Re-administration 58 |
| Table 11.2.1.1 Summary of Patients with DLT by Dose Level |
| Table 11.2.1.2 Characteristics of Patients with DLT by Dose Level |
| Table 11.3.1.1 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events. Worst Grade by Patient and Dose Level59 |
| Table 11.3.1.2 PM01183-Only Related (or Relationship Unknown) Adverse Events. Worst Grade by Patient and Dose Level59 |
| Table 11.3.1.3 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events. Worst Grade by Patient and Dose Level. |
| Table 11.3.1.4 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events in the First Cycle by Patient and Dose Level |
| Table 11.3.1.5 PM01183-Only Related (or Relationship Unknown) Adverse Events in the First Cycle by Patient and Dose Level |
| Table 11.3.1.6 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events in the First Cycle by Patient and Dose Level |
| Table 11.3.1.7 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events. Worst Grade Per Cycle by Dose Level59 |
| Table 11.3.1.8 PM01183-Only Related (or Relationship Unknown) Adverse Events. Worst Grade Per Cycle by Dose Level59 |
| Table 11.3.1.9 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events. Worst Grade Per Cycle by Dose Level |
| Table 11.3.1.10 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown)<br>Adverse Events Observed in ≥10% of Patients Treated by Dose Level |
| Table 11.3.1.11 PM01183-Only Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated by Dose Level59 |

| Table 11.3.1.12 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated by Dose Level5. |
|---|
| Table 11.3.1.13 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown, Adverse Events Observed in ≥ 10% of Patients Treated. Worst grade per Cycle by Dose Level |
| Table 11.3.1.14 PM01183-Only Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated. Worst grade per Cycle by Dose Level5 |
| Table 11.3.1.15 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events<br>Observed in ≥10% of Patients Treated. Worst grade per Cycle by Dose Level5 |
| Table 11.3.1.16 Adverse Events Regardless of Relationship. Worst Grade by Patient by Dose Level. 5 |
| Table 11.3.1.17 Adverse Events Regardless of Relationship in the First Cycle by Patient and Dose Level. 5 |
| Table 11.3.1.18 Adverse Events Regardless of Relationship. Worst Grade per Cycle by Dose Level. 5 |
| Table 11.3.1.19 Adverse Events Observed in $\geq 10\%$ of Patients Treated by Dose Level 5 |
| Table 11.3.1.20 Adverse Events Observed in ≥ 10% of Patients Treated. Worst grade per Cycle by Dose Level5 |
| Table 11.3.1.21 Supportive Listing: Drug Related (or Relationship Unknown) Adverse Events Grade 3-4 by Dose Level6 |
| Table 11.3.1.22 Time to course to Alopecia Grade >16 |
| Table 11.4.1.1 Patients who Died While on Treatment6 |
| Table 11.4.1.2 Patients Who Died Within 30 Days of Last Drug Administration 6 |
| Table 11.4.1.3 Listing of All Deaths6 |
| Table 11.4.2.1 All SAEs |
| Table 11.5.1.1 Hematological Abnormalities: Worst Grade per Patient by Dose Level 6 |
| Table 11.5.1.2 Hematological Abnormalities: Worst Grade per Cycle by Dose Level 6 |
| Table 11.5.1.3 Hematological Abnormalities: Worst Grade per patient in the First Cycle by Dose Level |
| Table 11.5.1.4 Supportive Listing: Patients with Grade 4 Hematological Abnormalities 6 |
| Table 11.5.1.5 Patients with Missing Hematological Evaluations |
| Table 11.5.1.6 Shift of Hematological Abnormalities. Baseline Grade vs. Worst Grade on First Cycle6. |
| Table 11.5.1.7 Shift of Hematological Abnormalities. Baseline Grade vs. Worst Grade on Treatment |
| Table 11.5.1.8 Listing of Patients with Hematological Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline6. |
| Table 11.5.1.9 Summary of Characteristics of wpp Hematological Abnormailities G3-4 6. |

| Table 11.5.1.10 Summary of Hematological Abnormalities Grade 4 and specific<br>Transfusions/treatment | 63 |
|---|---|
| Table 11.5.1.11 Anemia wpp/wpc and Use of EPO per Dose Level in Cycle >1 | 63 |
| Table 11.5.1.12 Patients with Anemia Grade 3/4 and Use of EPO in Cycle >1 | 63 |
| Table 11.5.1.13 Platelet Count Time Course Pattern (summary) | 63 |
| Table 11.5.1.14 Platelet Count Time Course Pattern | 64 |
| Table 11.5.1.15 Thrombocytopenia wpp/wpc and Use of Transfusions per Dose Level in Cycle>1 | 65 |
| Table 11.5.1.16 Patients with Thrombocytopenia Grade 3/4 and Use of Transfusions in Cycle >1 | 65 |
| Table 11.5.1.17 Summary of Hematological Abnormalities Grade 4 and Specific Transfusions | |
| Table 11.5.1.18 Neutrophil Count Time Course Pattern (summary) | |
| Table 11.5.1.19 Platelet Count Time Course Pattern | 66 |
| Table 11.5.1.20 Neuthropenia wpp/wpc and Use of Prophylactic CSF per Dose Level in Cycle>1 | 67 |
| Table 11.5.1.21 Patients with Neutrophenia Grade 3/4 and Use of Prophylactic CSF in Cycle >1 | |
| Table 11.5.2.1 Biochemical Abnormalities: Worst Grade per Patient by Dose Level | |
| Table 11.5.2.2 Biochemical Abnormalities: Worst Grade per Cycle by Dose Level | 67 |
| Table 11.5.2.3 Biochemical Abnormalities: Worst Grade per Patient in the first Cycle by Dose Level | |
| Table 11.5.2.4 Patients with Missing Biochemical Evaluation | |
| Table 11.5.2.5 Shift of Biochemical Abnormalities. Baseline Grade vs. Worst Grade on First Cycle | |
| Table 11.5.2.6 Shift of Biochemical Abnormalities. Baseline Grade vs. Worst Grade on Treatment | 68 |
| Table 11.5.2.7 Listing of patients with Biochemical Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline | 69 |
| Table 11.5.2.8 Summary of Characteristics of wpp Biochemical Abnormalities G3-4 | 69 |
| Table 11.5.2.9 AST/ALT Count Time Course Pattern (summary) | 69 |
| Table 11.5.2.10 AST/ALT Count Time Course Pattern | 70 |
| Table 11.5.3. 1 Other Metabolic Abnormalities: Worst Grade per Patient by Dose Level. | 70 |
| Table 11.5.3. 2 Other Metabolic Abnormalities: Worst Grade per Cycle by Dose Level | 70 |
| Table 11.5.3. 3 Other Metabolic Abnormalities: Worst Grade per Patient in the first Cycle by Dose Level. | |
| Table 11.5.3. 4 Patients with missing Metabolic Evaluations. | |

| Table 11.5.3. 5 Shift of Metabolic Abnormalities. Baseline Grade vs. Worst Grade on First Cycle7 |
|---|
| Table 11.5.3. 6 Shift of Metabolic Abnormalities. Baseline Grade vs. Worst Grade on Treatment |
| Table 11.5.3. 7 Listing of Patients with Metabolic Abnormailities >G2 and Experience Grade Increase (wpp) from Baseline |
| Table 11.5.3. 8 Supportive Listing: Patients with Grade ≥3 Metabolic Abnormalities 7. |
| Table 11.5.4. 1 Coagulation Abnormalities: Worst Grade per Patient by Dose Level 7. |
| Table 11.5.4. 2 Coagulation Abnormalities: Worst Grade per Cycle by Dose Level |
| Table 11.5.4. 3 Coagulation Abnormalities: Worst Grade per Patient in the first Cycle by Dose Level |
| Table 11.5.4. 4 Shift of Coagulation Abnormalities. Baseline Grade vs. Worst Grade on First Cycle. |
| Table 11.5.4. 5 Shift of Coagulation Abnormalities. Baseline Grade vs. Worst Grade on Treatment |
| Table 11.5.4. 6 Listing of Patients with Coagulation Abnormalities >G2 and Experience Grade Increase from Baseline7. |
| Table 11.5.4. 7 Patients with missing Metabolic Evaluations |
| Table 11.6.1.1 Physical examination during the Study by Cycle and Dose Level7 |
| Table 11.6.1.2 Performance Status during the Study by Cycle and Dose Level7 |
| Table 11.6.1.3 Weight Change during the Study by Dose Level7 |
| Table 11.6.2 1 ECG during the Study by Dose Level |
| Table 11.6.2 2 ECG during the Study by Dose Level |
| Table 11.6.2 3 QTcF Values during the Study by Dose Level |
| Table 11.6.2 4 QTcF (msec) Change per Patient during the Study by Dose Level |
| Table 11.6.2 5 Shift of QTc. Baseline Grade vs. Worst Grade on Treatment7 |
| Table 11.6.2 6 QTcF Values during the Study by Doxorubicin Cumulative Dose7 |
| Table 11.6.2 7 Listing of Patients with Grade $\geq$ 2 QTc Interval Prolonged7 |
| Table 11.6.3 1 LVEF (%) Change per Patient during the Study by Dose Level7 |
| Table 11.6.3 2 Median LVEF Values (%) during the Study by Doxorubicin Cumulative Dose. 7 |
| Table 11.6.3 3 Shift of LVEF. Baseline vs. Worst Grade on Treatment7 |
| Table 11.6.3 4 Listing of Patients with Grade $\geq$ 2 LVEF Decrease7 |
| Table 11.7.1.1 Concomitant Medication during Study (ATC Level 1 and 4) by Dose Level. |
| Table 11.7.1.2 EPO/RBC and PlateletsTransfusions/CSF7 |

| Table 11.7.1.3 Patients with EPO/RBC and Platelets Transfusions/CSF | 78 |
|---|---|
| Table 11.7.1.4 Prophylactic Medication during Study | 79 |
| Table 11.7.1.5 Patients with Nausea and /or Vomiting G3/4 and Use of Antiemetics in Cycle >1 | |
| Table 11.7.1.6 No of Patients with Opioids Treatment During Treatment by Dose Level. | 79 |
| Table 11.7.1.7 Median Number of No of Opioids per Patient During Treatment by Dose<br>Level | ,<br>79 |
| Table 11.7.1.8 No of Patients with Steroids Treatment During Treatment by Dose Level. | 80 |
| Table 11.7.1.9 Known CYP 3A4 Inducers/Inhibitors/Substrates Concomitant Therapies BL | |
| Table 11.7.1.10 Listing of CYP 3A4 Inducers/Inhibitors/Substrates Concomitant Therap<br>During Treatment | pies |
| Table 12.1.1.1 Overall response by Dose Level: Treated Patients | 81 |
| Table 12.1.1.2 Overall response by Tumor type and Dose Level: Treated Patients | 81 |
| Table 12.1.1.3 Overall response by Dose Level: Evaluable Patients | 82 |
| Table 12.1.1.4 Overall Response by Tumor type and Dose Level: Evaluable Patients | 82 |
| Table 12.1.1.5 SD ≥ 4 months by Dose Level: Evaluable Patients | 82 |
| Table 12.1.1.6 Tumor Marker Evolution During Study | 82 |
| Table 12.1.1.7 Characteristics of Patients with Clinical Benefit* | 82 |
| Table 12.1.1.8 Characteristics of Patients with Clinical Benefit based on any Specific Tumor Marker Criteria | |
| Table 12.1.1.9 Progression-Free Survival: Evaluable Patients | |
| Table 12.1.1.10 Duration of Response | |
| Table 12.1.1.11 Overall survival. | |
| Figure 13.1 1 Pattern of Hematological/non Hematological DLTs in Individual Patient | s. 84 |
| Figure 13.1 2 Transaminase Series in Individual Patients | |
| Figure 13.1 3 Barcharts of Adverse Events or Laboratory Abnormalities by Dose Level/Cohort | 85 |
| Figure 13.1 4 Barcharts of Adverse Events or Laboratory Abnormalities by Dose<br>Level/Cohort/Tumor type/ or Other Clinical Relevant Variable | 85 |
| Figure 13.1 5 Hematology/Transaminase Worst Severity by Cycle | 86 |
| Figure 13.1 6 LVEF/QTcF Boxplot by Dose Level | 86 |
| Figure 13.1 7 Boxplot QTcF Worst Value by Cycle | 87 |
| Figure 13.1 8 Duration of Response | |
| Figure 13.1 9 Progression-free Survival by Dose level/Cohort/Tumor type/ or Other<br>Clinical Relevant Variable | |

| Figure 13.1 10 Overall Survival | 88 |
|---|---|
| Figure 13.1 11 Waterfall Graphs | 89 |
| Figure 13.1 12 Spider plot: Evolution of RECIST v.1.1 Assessments | 89 |
| Figure 13.1 13 Best RECIST v.1.1 Efficacy Assessment in Evaluable pts per Ti | |
| Figure 13.1 14 Treatment Exposure and Reasons for Discontinuation per Tum | |
| Figure 13.1 15 Best RECIST v.1.1 Response According to Line of Treatment | 90 |
| Figure 13.1 16 Last Prior Treatment Response (TTP) vs PM001183/Combo res | |
| Figure 13.1 17 Number of Cycles, Reason for Treatment Discontinuation for F<br>Response or Clinical Benefit | |
| Figure 13.1 18 Efficacy and Individual TTP in Selected Patients by BSA/CTF1 Treatment Discontinuation | |
| Figure 13.1 19 Number of Cycles, Reason for Treatment Discontinuation and Patients who Received PM001183 Alone | |
| Listing 14.1 Patient Registration | 93 |
| Listing 14.2 Demography | 93 |
| Listing 14.3 Patient Disposition | 93 |
| Listing 14.4 Protocol Deviations | 93 |
| Listing 14.5 Patient Populations | 93 |
| Listing 14.6 Selection Criteria | 93 |
| Listing 14.7 Medical History | 93 |
| Listing 14.8 Cancer History. | 93 |
| Listing 14.9 Current Disease | 93 |
| Listing 14.10 Prior Surgery | 93 |
| Listing 14.11 Prior Radiotherapy | 93 |
| Listing 14.12 Prior Anticancer Therapy | 93 |
| Listing 14.13 Signs and Symptoms. | 93 |
| Listing 14.14 Tumor Assessment (Target Lesions) | 93 |
| Listing 14.15 Tumor Assessment (Non - Target Lesions) | 93 |
| Listing 14.16 Tumor Assessment (New Lesions) | 93 |
| Listing 14.17 Radiological Response (RECIST v.1.1). | 93 |
| Listing 14.18 Clinical Evaluation Response | 93 |
| Listing 14.19 Tumor Marker Evaluation Response | 93 |
| Listing 14.20 Overall Cycle Response | 93 |

| Listing 14.21 Treatment Exposure | <i>93</i> |
|---|---|
| Listing 14.22 Hematology Laboratory Results | 93 |
| Listing 14.23 Clinical Chemistry and Coagulation Laboratory Results | 93 |
| Listing 14.24 Physical Examination and Performance Status (PS) | 93 |
| Listing 14.25 Vital Signs | 93 |
| Listing 14.26 ECG Results | 93 |
| Listing 14.27 Left Ventricular Ejection Fraction (LVEF) Results | 93 |
| Listing 14.28 Other Tests and Procedures Results | 93 |
| Listing 14.29 Adverse Events | 93 |
| Listing 14.30 Concomitant Therapy | 93 |
| Listing 14.31 End of Treatment | 94 |
| Listing 14.32 Follow-up | 94 |
| Listing 14.33 Follow-up: Antitumor therapy | 94 |
| Listing 14.34 Death Report | 94 |
| Listing 14.35 Best Study Overall Response | 94 |
| Listing 14.36 Off Study | 94 |
| Listing 14.37 Signature Report | 94 |
| A footnote has been added | 115 |
| Table 10.2.1.1. Age at Entry by Dose Level | 115 |
| Table 10.2.7.9 CTFI by Dose Level/Cohort/Tumor typetype | 115 |
| Table 10.2.7.10 Summary Statistics: CTFI by Dose Level/Cohort/Tumor type | |
| Table12.1.1.10 Duration of Response | 117 |
| Table 12.1.1.11 Overall survival. | 118 |

# 10. Appendix I. Patients Disposition.

All statistical outputs will be displayed according to Dose level (grouped)/Cohort/Cancer type or primary site/CSF use or not/other clinical relevant variable, whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

## 10.1. General Characteristics.

## 10.1.1. Patients Treated, Eligible and Evaluable.

Table 10.1.1.1 Patient Accrual by Institution and Dose Level.

| | D | DLI | | DLII | | • • • | | DL n | | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % | N | % |
| Institution 1 | | | | | | | | | | |
| Institution 2 | | | | | | | | | | |
| ••• | | | | | | | | | | |
| Total | | | | | | | | | | |
| Note: Percentages based on number of patients l | by dose level. | | | | | | | | | |

Table 10.1.1.2 Disposition of Patients.

Date information

Date of first consent

Date of first dose

Date of last consent

Date of first dose of last patient

Date of last dose

Date of last follow up\*

Note: (\*) Last follow up date, examination date or procedure before study closure.

Table 10.1.1.3 Time on Treatment by Dose Level.

| Median and Range of Time on treatment (weeks) | DLI | DLII | <br>DLn | Total |
|-----------------------------------------------|-----|------|---------|-------|
| N | | | | |
| Mean | | | | |
| Median | | | | |
| Min | | | | |
| Max | | | | |
| STD | | | | |

Table 10.1.1.4 Number of Patients Evaluable for Analysis.

| Number of included | , | Treated | Patient | 5 | Evaluable for DLT | | | | Evaluable for Safety | | | | Evaluable for<br>Efficacy* | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| patients | Y | es | N | lo | Y | es | N | lo | Y | 'es | N | lo | Yes | No |
| · | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

DLI

DLn

\_\_\_\_\_\_

Notes: (\*) Efficacy by RECIST. A listing of patients not-evaluable by RECIST v.1.1 will be provided.

Table 10.1.1.5 Listing of Not Evaluable Patients.

| Table 10.1.1.5 Elisting 01 | Tiot Evaluable 1 | aticits. | |
|----------------------------|------------------|----------|-----------|
| Not Evaluable for | Dose level | Patient | Reason(s) |

DLT

Safety

Efficacy

| | Not Evaluable for | Dose level | Patient | Reason(s) |
|-------|-------------------|------------|---------|-----------|
| • • • | | • | | |

## 10.1.2. Treatment Discontinuations.

Table 10.1.2.1 Treatment Discontinuation by Dose Level\*.

| | D | DLI | | DLII | | • • • | | DLn | | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % | N | % |
| Progressive disease | | | | | | | | | | |
| Treatment non-related AE | | | | | | | | | | |
| Treatment related AE | | | | | | | | | | |
| Patient refusal | | | | | | | | | | |
| Death | | | | | | | | | | |
| Investigator's decision | | | | | | | | | | |
| Other ** | | | | | | | | | | |
| Total | | | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) Reasons for treatment discontinuation for patients who discontinued while the combination or PM alone will be provided, if required. (\*\*) If applicable, a supporting listing 10.1.2.1.a will be provided and reasons for treatment discontinuation may suffer recategorization after clinical review.

Table 10.1.2.2 Treatment Discontinuation Details.

| Dose level | Patient No | Last cycle infused | Treatment discontinuation reason | Details |
|---|---|---|---|---|
| Table 10.1.2.3 Reasons for Treatment Discontinuations by Cycle and Dose Level. | | | | |

| Treatment discontinuation | | I | DLI | | DLII | | • • • | | DL n | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % | N | % | N | % |
| Progressive disease | Cycle 1 | | | | | | | | | | |
| | Cycles 2-3 | | | | | | | | | | |
| | Cycles≥4 | | | | | | | | | | |
| Patient refusal | Cycle 1 | | | | | | | | | | |
| | Cycles 2-3 | | | | | | | | | | |
| | Cycles≥4 | | | | | | | | | | |
| Non treatment-related AE Cycle 1 | | | | | | | | | | | |
| | Cycles 2-3 | | | | | | | | | | |
| | Cycles≥4 | | | | | | | | | | |
| * | Cycle 1 | | | | | | | | | | |
| | Cycles 2-3 | | | | | | | | | | |
| | Cycles≥4 | | | | | | | | | | |
| | Cycle 1 | | | | | | | | | | |
| Total | Cycles 2-3 | | | | | | | | | | |
| | Cycles≥4 | | | | | | | | | | |

Notes: Percentages based on number of patients by dose level. Cycle grouping is only shown as an example.

Table 10.1.2.4 Listing of patients with Discontinuation with PM01183 alone.

| Dose level | Patient No | Last cycle infused | Treatment discontinuation reason | Details |
|---|---|---|---|---|

Table 10.1.2.5 Treatment Discontinuation Due to Adverse Events.

Note: (\*) Adverse event, Cycle, Grade, NCI-CTCAE v.4., Relationship, Action taken, Seriousness criteria, Prior PM01183 dose reduction.

Table 10.1.2.6 Reasons for Treatment Discontinuation Other than Progressive Disease.

| Dose level | Patient No | Last cycle infused | Off Study reason | Specify |
|---|---|---|---|---|
|---|---|---|---|---|

Table 10.1.2.7 Reasons for Study Discontinuation by Dose Level.

| Traction and discounting action | Dl | LI | DI | | • • | • | DL n | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| I reatment discontinuation | N | 0/0 | N | 0/0 | N | 0/0 | N | 0/0 | N | 0/0 |

Study completion

Patient follow-up completed

Patient refusal

Death

Never treated

Lost to follow up

Other\*

Total

Notes: Percentages based on number of patients by dose level. (\*) If applicable, a supporting listing 10.12.6.a will be showed.

#### 10.1.3. Protocol Deviations.

Table 10.1.3.1 Supportive Listing Relevant Protocol Deviations.

| Dose level | Patient No | Protocol deviation type | Specify |
|------------|------------|-------------------------|---------|
| | | , | |

### 10.2. Patient Characteristics.

All statistical outputs will be displayed according to Dose level (grouped)/Cohort/Cancer type or primary site/CSF use or not/other clinical relevant variable, whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

### 10.2.1. Patient Characteristics at Baseline.

Table 10.2.1.1 Age at Entry by Dose Level.

| A ora at antra i | DLI DLII | | • • • | | DL n | | Total | | | |
|------------------|----------|---|-------|---|------|---|-------|---|---|---|
| Age at entry | N | % | N | % | N | % | N | % | N | % |
| | DI | LI | DLII | | • • • | ] | OL n | To | otal |
|---|---|---|---|---|---|---|---|---|---|
| Age at entry | N | % | N ' | % l | N % | o N | % | N | % |
| 8-45 years | | | | | | | | | |
| 6-55 years | | | | | | | | | |
| < 76* years | | | | | | | | | |
| Fotal | 1 6 6 1 1 | 1 1 1 (* | A.F. 1 ( | | | | | | |
| Note: Percentages based on n | iumber of patients by c | lose level. (* | ) Example categor | 1es. | | | | | |
| Table 10.2.1.2 Age | Median and Ra | nge by I | Oose Level. | | | | | | |
| Age median and range | | DLI | DLII | | | | DL n | To | otal |
| N | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | DEI | | | | DE II | | Outi |
| Median | | | | | | | | | |
| Min | | | | | | | | | |
| Max | | | | | | | | | |
| STD | | | | | | | | | |
| Гable 10.2.1.3 Geno | der by Dose I e | a1 | | | | | | | |
| Tuble 10.2.1.5 Gene | DLI | V C1. | DLII | | | DL | | To | to1 |
| Gender — | N % | NT. | % | N | % | N DL | <u>%</u> | N 10 | |
| | N % | N | %0 | IN | %0 | IN | %0 | IN | % |
| Male | | | | | | | | | |
| Female | | | | | | | | | |
| Fotal | | | | | | | | | |
| Гаble 10.2.1.4 Race | by Dose Level | l <b>.</b> | | | | | | | |
| | by Dose Level | | DLII | • | •• | DL | , n | То | tal |
| | DLI | | | | | | | | |
| Gender — | | N | DLII % | N | | DI<br>N | . n | To<br>N | |
| Gender — | DLI | | | | | | | | |
| Gender —<br>Caucasian | DLI | | | | | | | | |
| Gender —<br>Caucasian<br><br>Total | DLI<br>N % | N | | | | | | | |
| Gender —<br>Caucasian<br><br>Total | DLI<br>N % | N | | | | | | | |
| Gender — Caucasian Total Note: Percentages based on n | DLI N % | N<br>lose level. | % | | | | | | |
| Gender — Caucasian Total Note: Percentages based on n | DLI N % number of patients by on | N<br>lose level. | %<br>evel. | | | N | % | N | % |
| Gender — Caucasian Fotal Note: Percentages based on n Fable 10.2.1.5 Preg | DLI N % number of patients by on the patients by one patients by o | N<br>lose level.<br>Dose Le | %<br>evel.<br>DLII | N | % | N<br>DI | %<br>. n | N | %<br>tal |
| Gender — Caucasian Total Note: Percentages based on n Table 10.2.1.5 Preg | DLI N % number of patients by on | N<br>lose level. | %<br>evel. | N | % | N | % | N | %<br>tal |
| Gender — Caucasian Total Note: Percentages based onn Table 10.2.1.5 Preg | DLI N % number of patients by on the patients by one patients by o | N<br>lose level.<br>Dose Le | %<br>evel.<br>DLII | N | % | N<br>DI | %<br>. n | N | %<br>tal |
| Gender — Caucasian Total Note: Percentages based onn Table 10.2.1.5 Preg Result — Not applicable* | DLI N % number of patients by on the patients by one patients by o | N<br>lose level.<br>Dose Le | %<br>evel.<br>DLII | N | % | N<br>DI | %<br>. n | N | %<br>tal |
| Gender — Caucasian Total Note: Percentages based onn Table 10.2.1.5 Preg Result — Not applicable* Negative | DLI N % number of patients by on the patients by one patients by o | N<br>lose level.<br>Dose Le | %<br>evel.<br>DLII | N | % | N<br>DI | %<br>. n | N | %<br>tal |
| Table 10.2.1.4 Race Gender — Caucasian Total Note: Percentages based onn Table 10.2.1.5 Preg Result — Not applicable* Negative Positive Total | DLI N % number of patients by on the patients by one patients by o | N<br>lose level.<br>Dose Le | %<br>evel.<br>DLII | N | % | N<br>DI | %<br>. n | N | % |
| Gender — Caucasian Fotal Note: Percentages based on n Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal | DLI N % number of patients by on the patients by the patients | N<br>lose level.<br>Dose Le | % evel. DLII % | N | % | N<br>DL<br>N | %<br>n | To N | %<br>tal |
| Gender — Caucasian Fotal Note: Percentages based on n Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal | DLI N % number of patients by on the patients by the patients | N<br>lose level.<br>Dose Le | % evel. DLII % | N | % | N<br>DL<br>N | %<br>n | To N | %<br>tal |
| Gender — Caucasian Fotal Note: Percentages based onn Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal Note: Percentages based onn | DLI N % number of patients by on the patients by DLI N % number of premenopal | N lose level. Dose Le N | % evel. DL II % by dose level. (*) A | N N A supporting | % | N<br>DL<br>N | %<br>n | To N | %<br>tal |
| Gender — Caucasian Fotal Note: Percentages based onn Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal Note: Percentages based onn | DLI N % number of patients by on ancy Tests by DLI N % number of premenoparatical Examination | N lose level. Dose Le N usal patients | % Evel. DL II % by dose level. (*) A | N N A supporting | % | DL<br>N | . n % | N To N | % of the second |
| Gender — Caucasian Fotal Note: Percentages based onn Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal Note: Percentages based onn Fable 10.2.1.6 Phys | DLI N % number of patients by on ancy Tests by DLI N % number of premenoparatical Examination | N lose level. Dose Le N usal patients | % evel. DL II % by dose level. (*) A | N N A supporting | % | DL<br>N | %<br>n | N To N | %<br>tal |
| Gender — Caucasian Fotal Note: Percentages based onn Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal Note: Percentages based onn Fable 10.2.1.6 Phys | DLI N % number of patients by on ancy Tests by DLI N % number of premenoparatical Examination | N lose level. Dose Le N usal patients | by dose level. (*) At the property of the prop | N N A supporting | % % listing 10.1.2.4 | DL<br>N | n % will be showe | To N | tal % |
| Gender — Caucasian Total Note: Percentages based on n Table 10.2.1.5 Preg Result — Not applicable* Negative Positive Total Note: Percentages based on n Table 10.2.1.6 Phys Physical Examination | DLI N % number of patients by on the patients by DLI N % number of premenopal ical Examination D | N lose level. Dose Le N usal patients | % Evel. DL II % by dose level. (*) A | N N A supporting | % % listing 10.1.2.4 | DL<br>N | . n % | N To N | % of the second |
| Gender — Caucasian Fotal Note: Percentages based onn Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal Note: Percentages based onn Fable 10.2.1.6 Phys Physical Examination Normal | DLI N % number of patients by on the patients by DLI N % number of premenopal ical Examination D | N lose level. Dose Le N usal patients | by dose level. (*) At the property of the prop | N N A supporting | % % listing 10.1.2.4 | DL<br>N | n % will be showe | To N | tal % |
| Gender — Caucasian Fotal Note: Percentages based on n Fable 10.2.1.5 Preg Result — Not applicable* Negative Positive Fotal Note: Percentages based on n Fable 10.2.1.6 Phys Physical Examination | DLI N % number of patients by on the patients by DLI N % number of premenopal ical Examination D | N lose level. Dose Le N usal patients | by dose level. (*) At the property of the prop | N N A supporting | % % listing 10.1.2.4 | DL<br>N | n % will be showe | To N | tal % |

Table 10.2.1.7 Physical Examination Parameters by Dose Level. DLI DL n Total . . . Weight (kg). N Mean Median Min Max STD N Mean Median Min Max STD Notes: (\*) Height (cm) and body surface area (BSA) (DuBois formula). Table 10.2.1.8 ECOG Performance Status by Dose Level at Baseline. DLI DLII DL n Total PS(ECOG) N % N % N % % % N N 0 1 Total Note: Percentages based on number of patients by dose level. Table 10.2.1.9 Vital Signs Parameters by Dose Level. Vital signs DLI DLII. . . DL n Total Heart rate (beats/minute) N Mean Median Min Max **STD** BPS (mmHg) N Median Min Max **STD** BPD (mmHg) N Mean Median Min Max STD Temperature (°C) N

Mean

| Vital signs | DLI | DLII | | DL n | Total |
|---|---|---|---|---|---|
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| Table 10.2.1.10 ECG Res | ult by Dose Level. | | | | |
| | DLI | DLII | • • • | DL n | Total |
| Physical Examination | N % | N % | N % | N % | N % |
| Normal | | | | | |
| Abnormal* | | | | | |
| Total | | | | | |
| Notes: Percentages based on number of | of patients by dose level. (*) | If abnormal, a supportive | listing will show detailed | information. | |
| Table 10.2.1.11 ECG Para | ameters by Dose L | evel. | | | |
| ECG | DLI | DLII | • • • | DL n | Total |
| PR interval (msec) | | | | | |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| QT interval (msec) | | | | | |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max<br>STD | | | | | |
| RR interval (msec) | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| QRS interval (msec) | | | | | |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| QTcF*(msec) | | | | | |
| N<br>Maga | | | | | |
| Mean<br>Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| Note: (*) Fridericia method. | | | | | |
| ( ) I I I I I I I I I I I I I I I I I I | | | | | |

Table 10.2.1.12 Median LVEF for Patients with Previous Treatment with Anthracyclines by Dose Level.

| LVEF | DLI | DLII | ••• | DL n | Total |
|--------------------|-----|------|-----|------|-------|
| Anthracyclines | | | | | |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| Non Anthracyclines | | | | | |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| Total | | | | | |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |

# 10.2.2. Cancer History.

Table 10.2.2.1 Time from Diagnosis to First Infusion.

| Time from Diagnosis to First Infusion | D | LI | D | LII | • | • • | D | Ĺn | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| (years) | N | % | N | % | N | % | N | % | N | % |
| N | | | | | | | | | | |
| Mean | | | | | | | | | | |
| Median | | | | | | | | | | |
| Min | | | | | | | | | | |
| Max | | | | | | | | | | |
| STD | | | | | | | | | | |

Table 10.2.2.2 Time from last PD to First Infusion.

| Time from Last PD to First Infusion | D | LI | DI | LΠ | | • | Dl | Ln | To | tal |
|---|---|---|---|---|---|---|---|---|---|---|
| (months) | N | % | N | % | N | % | N | % | N | % |
| N | | | | | | | | | | |
| Mean | | | | | | | | | | |
| Median | | | | | | | | | | |
| Min<br>Max | | | | | | | | | | |
| Max | | | | | | | | | | |
| STD | | | | | | | | | | |

Table 10.2.2.3 TTP of Last Prior Therapy.

| TTP in months of last Prior Therapy | DLI | | DLII | | • • • | | DLn | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| TTP in months of last Prior Therapy | N | % | N | % | N | % | N | % | N | % |

| TTD in months of lost Drien Thomas | D | LI | D | LΠ | | | D | Ln | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| TTP in months of last Prior Therapy | N | % | N | % | N | % | N | % | N | % |
| N | | | | | | | | | | <u>.</u> |
| Mean | | | | | | | | | | |
| Median | | | | | | | | | | |
| Min | | | | | | | | | | |
| Max | | | | | | | | | | |
| STD | | | | | | | | | | |

Table 10.2.2.4 Tumor type by Dose Level.

| Tumont ma* | D | LI | Dl | LΠ | • • | | DI | _ n | To | otal |
|-------------|---|----|----|----|-----|---|----|-----|----|------|
| Tumor type* | N | % | N | % | N | % | N | % | N | % |
| Breast | | | | | | | | | | |
| * | | | | | | | | | | |
| Total | | | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) CRF categories will be shown and categories will be susceptible of clinical coding, if requested. A supportive table 10.22.6.a will be provided for subcategories. (e.g. sarcomas).

Table 10.2.2.5 Summary of Cancer History per Patient and Tumor type.

| Oose | Histology |
|------|-----------|

Notes: (\*) Stage at diagnosis, Histology grade, Date of first diagnosis, Current stage (date), date of last PD before study entry, TTP to prior therapy, best response to last prior therapy. Also characteristics of patients by specific turnor type, e.g. smoker, etc. . . If required, tabulations for specific categories will be shown as Supportive tables.

#### 10.2.3. Sites Involved.

Table 10.2.3.1 No of Sites Involved by Tumor type and Dose Level.

| T | No of Citos | D | LI | D | LII | • • | • • | D | Ln | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Tumor Type* | NOOI SILES | N | % | N | % | N | % | N | % | N | % |
| Breast | 1 Sites | | | | | | | | | | |
| | 2 Sites | | | | | | | | | | |
| | >2 | | | | | | | | | | |
| * | 1 Sites | | | | | | | | | | |
| | 2 Sites | | | | | | | | | | |
| | >2 | | | | | | | | | | |
| | Total | | | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) Coded tumor types.

Table 10.2.3.2 Summary Statistics. No of Sites Involved by Tumor type Dose Level.

| Tumor Type* | Median, range and STD for<br>No. of sites involved | DLI | DLII | ••• | DLn | Total |
|---|---|---|---|---|---|---|
| Breast | N** | | | | | _ |
| * | | | | | | |

Notes: (\*) Coded tumor types. (\*\*) N, mean, STD, median and range.

| Table 10.2.3.3 | Frequency of Patients | Classified by Sites Involved by | y Tumor type and Dose Level. |
|---|---|---|---|
|---|---|---|---|

| TumonTumo* | Cita** | D | LI | D | LII | • | • • | Dl | L n | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Tumor Type* | Site** | N | % | N | % | N | % | N | % | N | % |
| Breast | CNS<br>Liver | | | | | | | | | | |
| * | | | | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\* and \*\*\*) Coded tumor types and sites will be recoded, if required.

Table 10.2.3.4 Listing of Sites per Patient.

| Dose | Patient | Transactions* | Towart/Nian towart | Mathad | Diamatan (mm) |
|---|---|---|---|---|---|
| level | No | Tumor type* | Target/Non target | Method | Diameter (mm) |

Note: (\*) Coded tumor types.

Table 10.2.3.5 Bulky disease by Tumor type and Dose Level.

| Tumor type* | Maximum | D | LI | DLII | | ••• | | DL n | | Total | |
|-------------|----------|---|----|------|---|-----|---|------|---|-------|---|
| Turnor type | diameter | N | % | N | % | N | % | N | % | N | % |
| Breast | ≥50 mm | | | | | | | | | | |
| | < 50 mm | | | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) Coded tumor types.

Table 10.2.3.6 Median sum of diameter of target lesions (mm).

| Tumortype* | Median and range for sum of target lesions (mm) | DLI | DLII | <br>DLn | Total |
|---|---|---|---|---|---|
| Breast | N** | | | | |
| ••••• | | | | | |

Notes: (\*) Coded tumor types (\*\*) N, mean, STD, median and range.

#### 10.2.4. Previous Treatment Summary.

Table 10.2.4.1 Previous Treatment Summary by Dose Level.

| Previous Treatment | DL | Ι | DI | LΠ | | • | DI | _ n | To | otal |
|--------------------|----|---|----|----|---|---|----|-----|----|------|
| Previous Treatment | N | % | N | % | N | % | N | % | N | % |

Systemic Therapy

Surgery\*

Radiotherapy

Systemic Therapy + Surgery\*

Systemic Therapy + Radiotherapy

Systemic Therapy + Surgery\*+

Radiotherapy

Total

Notes: Percentages based on number of patients by dose level. (\*) Curative/Palliative.

Table 10.2.4.2 Previous Systemic Therapy by Dose Level/Tumor type.

| Tumor type | Previous Treatment | DLI | DLII | • • • | DL n | Total |
|------------|--------------------|-----|------|-------|------|-------|

| | • | N | % | N | % | N | % | N | % | N | % |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Breast | Chemotherapy<br>Biological therapy<br>Hormonal therapy<br> | | | | | | | | | | |
| | Total | | | | | | | | | | |

Note: (\*) Adjuvant and /or necadjuvant therapies are not included in this table, if required a supportive table for this therapies will be shown.

### 10.2.5. Previous Surgery.

Table 10.2.5.1 Previous Surgery by Dose Level (Curative/Palliative).

| Durania va Compour | D | LI | D | LII | • | • • | Dl | _ n | Total | |
|--------------------|---|----|---|-----|---|-----|----|-----|-------|---|
| Previous Surgery | N | % | N | % | N | % | N | % | N | % |
| No | | | | | | | | | | |
| Yes | | | | | | | | | | |
| Total | | | | | | | | | | |

Note: Percentages based on number of patients by dose level.

### 10.2.6. Previous Radiotherapy.

Table 10.2.6.1 Previous Radiotherapy by Dose Level.

| Previous | D | LI | D | LII | • | | DI | _ n | To | otal |
|--------------|---|----|---|-----|---|---|----|-----|----|------|
| Radiotherapy | N | % | N | % | N | % | N | % | N | % |
| No | | | | | | | | | | |
| Yes | | | | | | | | | | |
| Total | | | | | | | | | | |

Note: Percentages based on number of patients by dose level.

#### 10.2.7. Previous Anticancer Medical Therapy.

Table 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1 & 4) by Dose Level/Tumor type.

| Medication* | D | LI | D | LΠ | | • • | D | Ln | To | otal |
|-------------|---|----|---|----|---|-----|---|----|----|------|
| Medicauon* | N | % | N | % | N | % | N | % | N | % |
| ATC level 1 | | | | | | | | | | |
| ATC level 4 | | | | | | | | | | |
| ••• | | | | | | | | | | |
| ATC level 4 | | | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) A supportive table of Agents of Previous Chemotherapy will be displayed. Adjuvant and/or neoadjuvant therapies are not included in this table; if required, a supportive table for these therapies will be shown.

Table 10.2.7.2 No of Lines of Prior Anticancer Therapy for Advanced Disease by Dose Level/Tumor type.

| N Cl:* | D. | LI | Dl | LII | | • • | D | Ln | To | otal |
|-------------------|----|----|----|-----|---|-----|---|----|----|------|
| No of lines* | N | % | N | % | N | % | N | % | N | % |
| 0 lines | | | | | | | | | | |
| 0 lines<br>1 line | | | | | | | | | | |
| • • • • • | | | | | | | | | | |
| $\geq$ N lines | | | | | | | | | | |

| NICl:* | | DLI | | DLII | | • • • | Γ | <b>)</b> Ln | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| No of lines* | N | % | N | J % | N | % | N | % | N | % |
| Fotal | | | | | | | | | | |
| Notes: Percentages based on numb<br>Agents of Previous Chemotherapy- | | | | | | t therapies are | not included | d in this table | and a suppo | ortive table |
| agenisori revious chemoricapy- | COLLABILITY 1 | nciapies ioi z | Huvancui | Discase Will U | e dispiayed. | | | | | |
| Γable 10.2.7.3 Summary | z Statistie | cs No of | `Lines o | of Prior A | nticancer | Therapy l | ny Dose | I evel/Tu | mor tyne | |
| Median and range for No of | y Statistiv | | Lines | | inticancei | | | | | |
| lines* | | DLI | | DLII | | ••• | L | <b>D</b> Ln | 10 | otal |
| N | | | | | | | | | | |
| Mean | | | | | | | | | | |
| Median | | | | | | | | | | |
| Min | | | | | | | | | | |
| Max | | | | | | | | | | |
| STD | | | | | | | | | | |
| Note: (*) Adjuvant and /or neoadju | vant therapie | s are not incl | uded in this | stable and a s | upportive tab | le of Agents o | f Previous C | hemotherapy | -containing | Theranie |
| Advanced Disease will be displayed | | | | | Tr | | | FJ | | т |
| 1 · J | | | | | | | | | | |
| - 11 10 <b>2 -</b> 1 3 7 - 6 1 | | | | <b></b> 1 | | 1/20 | | | | |
| Table 10.2.7.4 No of Ag | | | | | • | | | | | . 1 |
| No of agents — | DL | | | LII | NT NT | | DL | | To | |
| | N | % | N | % | N | % | N | % | N | % |
| agents | | | | | | | | | | |
| l agent | | | | | | | | | | |
| 2 agents | | | | | | | | | | |
| ≥Nagents | | | | | | | | | | |
| Total | | | | | | | | | | |
| Note: Percentages based on number | ofpatientsb | v dose level. | Any agents | sused more th | an once will o | only add 1 to th | ne total. | | | |
| | 1 | , | J 1.0 | | | <i>J</i> | | | | |
| T.1.1. 10 2 7 5 N C A . | | D. | | | 1 C. | DM011 | 02 4 | 1. D | т | 1/T |
| Table 10.2.7.5 No of Ag | gents of I | Last Prior | Antica | ncer Ther | apy befor | re PM011 | 83 treatn | nent by D | ose Leve | el/Tum |
| type. | | | | | | | | | | |
| No of agents — | DL | | | LII | • • | | DL | | To | |
| 10 of agents | N | % | N | % | N | % | N | % | N | % |
| ) agents | | | | | | | | | | |
| l agent | | | | | | | | | | |
| 2 agents | | | | | | | | | | |
| - 100 | | | | | | | | | | |
| <br>≥Nagents | | | | | | | | | | |
| Fotal | | | | | | | | | | |
| | C 1 | 1 1 1 | A | 1 4 | '11 | . 1 . 1117 / | 1 | | | |
| Note: Percentages based on number | orpatients o | y dose level. | Any agents | s usea more in | an once will o | oniyada i totr | ie totai. | | | |
| Table 10.2.7.6 Summary | y Statistic | cs. No of | Agents | of Prior | Anticance | er Therapy | by Dos | e Level/T | umor typ | e. |
| Median and range for No of | | | | | | 1.7 | | | | |
| <del>-</del> | | DLI | | DLII | | • • • | D | Ln | To | otal |
| agents | | | | | | | | | | |
| N | | | | | | | | | | |
| Mean<br>Median<br>Min | | | | | | | | | | |

Min Max STD

| Dose level Patient N | o Setting Type | | Anticancer Then* | 100 | | | | Progressi | on date |
|---|---|---|---|---|---|---|---|---|---|
| (*) Dose and units; Schedi | ıle, Start—End date an | d Best Resp | onse. | | | | | | |
| ., | | | | | | | | | |
| Table 10.2.7.8 Ag | | | * * * | | • | | | | . 1 |
| Agents* | DL<br>N | <u>1</u> % | DLII<br>N % | N | % | DI<br>N | ∠ n // <sub>%</sub> | N | otal<br>% |
| Platinum | IN | 70 | N % | IN | %0 | IN | %0 | IN | %0 |
| •••• | | | | | | | | | |
| Notes: Percentages based o | on number of nationts | by dose lev | elorbytumortyne Am | zagents used n | none than onc | e will only a | ld 1 to the tot | al (*) Indicat | ed by clini |
| equest e.g: Anti-EGFR tar | - | - | | _ | | e wiii Oriiy ac | ICI IO UIC IOU | al.() likika | ica by Cilli |
| equeste.g.7 init-Eor Real | дассинацися, таха | iks, Ouki ii | ivesugational citags, etc. | •• | | | | | |
| | | | _ | | | | | | |
| Table 10.2.7.9 CT | TFI by Dose Le | vel/Coho | ort/Tumor type | | | | | | |
| | - , | | | | | | | | |
| CTU/TU* | DL | I | DLII | • | • | DI | _ n | To | otal |
| CTFI/TFI* | | <u>%</u> | DLII<br>N % | N | % | DI<br>N | <u>√</u> n /⁄₀ | N To | otal<br>% |
| | DL | | | | | | | | |
| Resistant | DL | | | | | | | | |
| Resistant<br>Sensitive | DL | | | | | | | | |
| Resistant<br>Sensitive | DL | | | | | | | | |
| Resistant<br>Sensitive<br> | DL<br>N | 0/0 | N % | N | % | N | % | N | % |
| Resistant Sensitive Total Note: (*) CTF1 (Chemoth | DL<br>N<br>eraphy Free Interval)/1 | %<br>for SCLC pa | N % atients and TFI (System | N<br>c Chemothera | % py Free Inter | N<br>val) for Endo | % metrial patien | N ts. Calculated | % I from the |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth | DL<br>N eraphy Free Interval)/1 with ATC coded "L0 | %<br>for SCLC pa | N % atients and TFI (System | N<br>c Chemothera | % py Free Inter | N<br>val) for Endo | % metrial patien | N ts. Calculated | % I from the |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth | DL<br>N eraphy Free Interval)/1 with ATC coded "L0 | %<br>for SCLC pa | N % atients and TFI (System | N<br>c Chemothera | % py Free Inter | N<br>val) for Endo | % metrial patien | N ts. Calculated | % I from the |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy v (resistant) and S (sensitive). | DL<br>N exaphy Free Interval)/1 with ATC coded ''L0 | %<br>for SCLC pa<br>11XA" and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Interested of there | N<br>val) for Endo<br>py to the PC | % metrial patien | N ts. Calculated | % I from the I |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy v (resistant) and S (sensitive). Table 10.2.7.10 S | DL<br>N eraphy Free Interval)/1 with ATC coded ''L0 ummary Statist | %<br>for SCLC pa<br>11XA" and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Interested of there | N<br>val) for Endo<br>py to the PC | % metrial patien | N ts. Calculated | % I from the l |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy v (resistant) and S (sensitive). | DL N exaphy Free Interval)/1 with ATC coded '10 ummary Statist | % for SCLC pay IXA'' and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Interested of there | N val) for Endo py to the PC e. | %<br>metrial patien<br>), e.g. for SC | N<br>ts. Calculated<br>LC patients ( | % I from the I |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy v (resistant) and S (sensitive). Table 10.2.7.10 S Tumor type*/Median | DL N exaphy Free Interval)/1 with ATC coded '10 ummary Statist | %<br>for SCLC pa<br>11XA" and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Intered of there umor typ | N val) for Endo py to the PC e. | % metrial patien | N<br>ts. Calculated<br>LC patients ( | % I from the l |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy v (resistant) and S (sensitive). Table 10.2.7.10 S Turnor type*/Median range | DL N exaphy Free Interval)/1 with ATC coded '10 ummary Statist | % for SCLC pay IXA'' and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Intered of there umor typ | N val) for Endo py to the PC e. | %<br>metrial patien<br>), e.g. for SC | N<br>ts. Calculated<br>LC patients ( | % I from the I |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy versistant) and S (sensitive). Table 10.2.7.10 S Turnor type*/Median range | DL N exaphy Free Interval)/1 with ATC coded '10 ummary Statist | % for SCLC pay IXA'' and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Intered of there umor typ | N val) for Endo py to the PC e. | %<br>metrial patien<br>), e.g. for SC | N<br>ts. Calculated<br>LC patients ( | % I from the I |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy viresistant) and S (sensitive). Table 10.2.7.10 S Tumor type*/Median range N Mean | DL N exaphy Free Interval)/1 with ATC coded '10 ummary Statist | % for SCLC pay IXA'' and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Intered of there umor typ | N val) for Endo py to the PC e. | %<br>metrial patien<br>), e.g. for SC | N<br>ts. Calculated<br>LC patients ( | % I from the Categories |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy versistant) and S (sensitive). Table 10.2.7.10 S Tumor type*/Median range N Mean Median | DL N exaphy Free Interval)/1 with ATC coded '10 ummary Statist | % for SCLC pay IXA'' and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Interested of there umor typ | N val) for Endo py to the PC e. | %<br>metrial patien<br>), e.g. for SC | N<br>ts. Calculated<br>LC patients ( | % I from the Categories |
| Resistant Sensitive Total Note: (*) CTFI (Chemoth therapy previous therapy v (resistant) and S (sensitive). Table 10.2.7.10 S | DL N exaphy Free Interval)/1 with ATC coded '10 ummary Statist | % for SCLC pay NIXA'' and | N % atients and TFI (System calculated as the differ | N<br>ic Chemothera<br>ence from the | % py Free Interested of there umor typ | N val) for Endo py to the PC e. | %<br>metrial patien<br>), e.g. for SC | N<br>ts. Calculated<br>LC patients ( | % I from the Categories |

Table 10.2.7.11 Patients Previously Treated with Anthracyclines by Dose Level.

| A settem or valin oak | D | LI | Dl | LII | | • • | D | L n | To | otal |
|-----------------------|---|----|----|-----|---|-----|---|-----|----|------|
| Anthracyclines* | N | % | N | % | N | % | N | % | N | % |
| Yes | | | | | | | | | | |
| No | | | | | | | | | | |
| Total | | | | | | | | | | |

Note: (\*) For those patients previously treated with anthracyclines a supportive listing 10.277.a will be given.

Table 10.2.7.12 Summary Statistics: Cumulative Dose in Patients Previously Treated with Anthracyclines by Dose Level.

| Dose | Levei. | | | | |
|------------------|--------|------|-------|------|-------|
| Median and range | DLI | DLII | • • • | DL n | Total |
| N | | | | | |
| Mean<br>Median | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |

| Median and range | | DLI | DLII | • • • | DL n | Total |
|---|---|---|---|---|---|---|
| STD | | | | | | |
| 0.2.8. Hemat | ological Ev | valuation at | t Baseline. | | | |
| Гable 10.2.8.1 Не | ematological A | Abnormalities | at Baseline by D | Oose Level. | | |
| Abnormality* | | DLI | DLII | | DL n | Total |
| Anemia | | | | | | |
| Grade 1 - 4, n (%) | | | | | | |
| Grade 1 | | | | | | |
| Grade 2 | | | | | | |
| Grade 3 | | | | | | |
| Grade 4 | | | | | | |
| * | | | | | | |
| Grade 1 - 4, n (%) | | | | | | |
| Grade 1 | | | | | | |
| Grade 2 | | | | | | |
| Grade 2<br>Grade 3 | | | | | | |
| Grade 2<br>Grade 3<br>Grade 4<br>Notes: Baseline values obt | | | | ion .Percentages based on nun | nber of patients by dose | level/cohort.(*) A |
| Grade 2<br>Grade 3<br>Grade 4 | | | | ion .Percentages based on nun | nber of patients by dose | level/cohort. (*) A |
| Grade 2<br>Grade 3<br>Grade 4<br>Notes: Baseline values obt<br>Leukopenia, Lymphopen | ia, Neutropenia, and | l Thrombocytopenia | | ion Percentages based on nun<br>eers at Baseline by Do | | level/cohort. (*) A |
| Grade 2<br>Grade 3<br>Grade 4<br>Notes: Baseline values obt<br>Leukopenia, Lymphopen | ia, Neutropenia, and | l Thrombocytopenia | | - | | level/cohort. (*) A Total |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Table 10.2.8.2 Me Parameters* Hemoglobin ( | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Table 10.2.8.2 Ma | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Table 10.2.8.2 Me Parameters* Hemoglobin ( | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obteukopenia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin (s) Mean | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Table 10.2.8.2 Me Parameters* Hemoglobin ( N Mean Median | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obtende penia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin ( Mean Median Min | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obtenukopenia, Lymphopen Fable 10.2.8.2 Marameters* Hemoglobin (Marameterian) Median Min Max | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Fable 10.2.8.2 Ma Parameters* Hemoglobin ( N Mean Median Min Max | ia, Neutropenia, and<br>edian and Rar | l Thrombocytopenia<br>nge for Hemato | ological Paramet | ers at Baseline by De | ose Level. | |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obtective penia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin (s) Mean Median Min Max STD* | ia, Neutropenia, and<br>edian and Rar<br>g/dL) | 1Thrombocytopenia | ological Paramet | ers at Baseline by De | ose Level.<br>DL n | Total |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obtenukopenia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin (s) Mean Median Min Max STD* Notes: Baseline values obtenue solues obtenue services solues s | ia, Neutropenia, and edian and Rar g/dL) stained from last va | ange for Hemato | ological Paramet | ers at Baseline by De | ose Level.<br>DL n | Total |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin (s) Mean Median Min Max STD* Notes: Baseline values ob | ia, Neutropenia, and edian and Rar g/dL) stained from last va | ange for Hemato | ological Paramet | ers at Baseline by De | ose Level.<br>DL n | Total |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obtective penia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin (s) Mean Median Min Max STD* Notes: Baseline values obtective penia, Lymphocytes, WBC, Net | ia, Neutropenia, and edian and Ran g/dL) otained from last valutrophils, Platelets in | alter recorded before in 109/L. | ological Paramet DLII or on the date of first in | ers at Baseline by De | ose Level. DL n number of patients by | Total dose level. (*) A |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin (s) Mean Median Min Max STD* Notes: Baseline values obt Lymphocytes, WBC, Nea | ia, Neutropenia, and edian and Ran g/dL) otained from last valutrophils, Platelets in | alter recorded before in 109/L. | ological Paramet DLII or on the date of first in | ers at Baseline by Do | ose Level. DL n number of patients by | Total dose level. (*) A |
| Grade 2 Grade 3 Grade 4 Notes: Baseline values obt Leukopenia, Lymphopen Fable 10.2.8.2 Me Parameters* Hemoglobin (s) Mean Median Min Max STD* Notes: Baseline values obt Lymphocytes, WBC, Nea | ia, Neutropenia, and edian and Ran g/dL) otained from last valutrophils, Platelets in | alter recorded before in 109/L. | ological Paramet DLII or on the date of first in | ers at Baseline by Do | ose Level. DL n number of patients by | Total dose level. (*) A |

Patient

Table 10.2.8.4 Patients with Missing Hematological Evaluations at Baseline.

Dose level

Lab. test

#### 10.2.9. Biochemical Evaluation at Baseline.

Table 10.2.9.1 Biochemical Abnormalities at Baseline by Dose Level

| Abnormality* | DLI | DLII | • • • | DL n | Total |
|--------------------|-----|------|-------|------|-------|
| AP increase | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |
| * | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |

Notes: Baseline values obtained from last value recorded before or on the date of first infusion. Percentages based on number of patients by dose level. (\*) All biochemical abnormalities susceptible to be graded with NCI-CTCAE v.4.

Table 10.2.9.2 Median and Range for Biochemical Parameters at Baseline by Dose Level.

| Parameters* | DLI | DLII | • • • | DL n | Total |
|-------------|-----|------|-------|------|-------|
| AP | | | | | _ |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |
| * | | | | | _ |
| N | | | | | |
| Mean | | | | | |
| Median | | | | | |
| Min | | | | | |
| Max | | | | | |
| STD | | | | | |

Note: (\*) Baseline values obtained from last value recorded before or on the date of first infusion AP, AST, ALT, LDH, CPK, CPK MB and Amylase in IU/L. Total and direct bilirubin, creatinine, Alpha-1 acid glycoprotein, and LDL in mg/dl. Total proteins in g/dl and C-reactive protein in mg/l.

Table 10.2.9.3 Supportive Listing: Patients with Grade >1 Biochemical Abnormalities at Baseline.

| Dose level | Patient | Lab. test | Cycle | Examination date | Std. value | Grade NCI-<br>CTCAE v.4 |
|---|---|---|---|---|---|---|
| Table 10.2.9.4 Pati | ents with M | lissing Biochen | nical Evaluations | s at Baseline. | | |
| D | ose level | | Patient | | Lab. test | |

Grade NCI-

#### Coagulation Evaluations at Baseline. 10.2.10.

Table 10.2.10. 1 Coagulation Abnormalities at Baseline by Dose Level.

| Abnormality | DLI | DLII | • • • | DL n | Total |
|---|---|---|---|---|---|
| INR increase | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |
| PTT | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |
| Note: Baseline values obtained from | n last value recorded before or | on the date of first infusion | n. Percentages based on | number of patients by dos | e level. |

Table 10.2.10. 2 Median and Range for Coagulation Parameters at Baseline by Dose Level.

| Parameters* | DLI | DLII | <br>DL n | Total |
|-------------------|-----|------|----------|-------|
| INR | | | | |
| N | | | | |
| Mean | | | | |
| Mean<br>Median | | | | |
| Min | | | | |
| Max | | | | |
| Min<br>Max<br>STD | | | | |
| * | | | | |

Notes: (\*) Baseline values obtained from last value recorded before or on the date of first infusion. INR: no units. PTT and PT in seconds.

Table 10.2.10. 3 Supportive Listing: Patients with Grade >1 Coagulation Abnormalities at Baseline.

| Dose level | Dotiont | Lab tost | Cyrolo | Examination data | Std volue | Grade NCI- |
|---|---|---|---|---|---|---|
| Dose level | Patient | Lab. test | Cycle | Examination date | Std. value | CTCAE v.4 |

Table 10.2.10. 4 Patients with Missing Coagulation Evaluations at Baseline.

| Tuble 10.2.10. T Tutlents with Williams Co | bagaiation Evaluations at Basen | 110. |
|---|---|---|
| Dose level | Patient | Lab. test |

#### 10.2.11. Other Metabolic Evaluations at Baseline.

Table 10.2.11. 1 Metabolic Abnormalities at Baseline by Dose Level.

| Abnormality* | DLI | DLII | • • • • | DL n | Total |
|--------------|-----|------|---------|------|-------|

Hypercalcemia

Grade 1 - 4, n (%)

Grade 1

Grade 2

| Abnormality* | | | DLI | | DLII | | | | DL | n | Tot | al |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Grade 3 | | | | | | | | | | | | |
| Grade 4 | | | | | | | | | | | | |
| * | | | | | | | | | | | | |
| Grade 1 - 4, n (%) | | | | | | | | | | | | |
| Grade 1 | | | | | | | | | | | | |
| Grade 2 | | | | | | | | | | | | |
| Grade 3 | | | | | | | | | | | | |
| Grade 4 | | | | | | | | | | | | |
| Notes: Baseline values<br>metabolic abnormalities | | | | | | of first infu | sion. Perce | ntages based o | on numb | er of patients | by dose le | vel. (*) A |
| Гable 10.2.11. 2 | Median | and Rane | ge for l | Metabo | lic Paran | neters at | t Racelir | ne by Dos | e I eve | 1 | | |
| Parameters* | Wiculan | | DLI | victabo | DLII | icicis a | ··· | ic by Dos | DL | | Tot | n1 |
| | | | DLI | | DLII | | | | DL | , II | 100 | aı |
| Calcium<br>N | | | | | | | | | | | | |
| N<br>M | | | | | | | | | | | | |
| Mean<br>Madian | | | | | | | | | | | | |
| Median<br>Mira | | | | | | | | | | | | |
| Min<br>Mov | | | | | | | | | | | | |
| Max<br>STD | | | | | | | | | | | | |
| *<br>Notes: (*) Baseline val | | | | | | | | | | | | |
| TIITIOVI., III giyootides ati | d total chole | sterol in mg/dl | | | | OI IIISCII IIG | | | | | | |
| | | sterol in mg/dl | Landalbi | umin in g/d | L. | | | Abnormal | ities at | Baseline | <del>2</del> . | |
| | | sterol in mg/dl | Landalbi | umining/d | L. | | tabolic . | Abnormal<br>ination date | | Baseline<br>Std. value | Grad | e NCI-<br>AE v.4 |
| Table 10.2.11. 3 | Suppor | sterol in mg/dl | Landalbi | umining/d | L.<br>rith grade | | tabolic . | | | | Grad | |
| Table 10.2.11. 3 Dose level/ | Suppor<br>Pat | sterol in mg/dl | Landalbi<br>ng: Par<br>Lab. tes | umin in g/d<br>tients w | ith grade | e>1 Me | tabolic .<br>Exam | ination date | | | Grad | |
| Table 10.2.11. 3 Dose level/ | Suppor<br>Pat | sterol in mg/dl | Landalbi<br>ng: Par<br>Lab. tes | umin in g/d<br>tients w | ith grade<br>Cycle<br>ic Evalua | e>1 Me | tabolic .<br>Exam | ination date | | | Grad | |
| Table 10.2.11. 3 | Support Pat | sterol in mg/dl | Landalbi<br>ng: Par<br>Lab. tes | umin in g/d<br>tients w | ith grade<br>Cycle<br>ic Evalua | e >1 Me | tabolic .<br>Exam | ination date | | Std. value | Grad | |
| Table 10.2.11. 3 Dose level/ | Support Pat | sterol in mg/dl | Landalbi<br>ng: Par<br>Lab. tes | umin in g/d<br>tients w | ith grade<br>Cycle<br>ic Evalua | e >1 Me | tabolic .<br>Exam | ination date | | Std. value | Grad | |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 | Patients Dose let | sterol in mg/dl | ng: Pa<br>Lab. tes | tients w | ith grade Cycle ic Evalua | e >1 Me | tabolic .<br>Exam | ination date | | Std. value | Grad | |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 | Patients Dose let | sterol in mg/dl | ng: Par Lab. tess | tients west | ith grade Cycle ic Evalua P | e >1 Me | tabolic .<br>Exam | ination date | | Std. value | Grad | |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 10.2.12. Si Table 10.2.12. 1 | Patients Dose let | sterol in mg/dl | ng: Pa Lab. tes sssing N | tients west | ith grade Cycle ic Evalua P | e >1 Me | tabolic .<br>Exam | ination date | | Std. value | Grad<br>CTC | |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 10.2.12. Si Table 10.2.12. 1 MedDRA System | Patients Dose let | sterolinmg/dl rtive Listi ient s with Mis vel d Symp nd Sympt DLI | ng: Pa Lab. tes sssing N | tients west | ith grade Cycle ic Evalua P | e >1 Me | Exam | ination date | | Std. value Lab. test | Grad<br>CTC | |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 10.2.12. Si Table 10.2.12. 1 MedDRA System Organ Class | Patients Dose lev Signs an Gr. 1* | sterol in mg/dl retive Listinient s with Misswel d Symp nd Sympt DLI Gr. 2 Gr. | ng: Par Lab. tess ssing N toms coms by | tients w t Aetabol at Ba | ith grade Cycle ic Evalua P seline. Level. | e >1 Me | Exam Baselin Gr. 3 | ination date | Gr. 1 | Lab. test Tot Gr. 2 | Grad<br>CTC | AE v.4 |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 | Patients Dose lev Signs an Gr. 1* | sterol in mg/dl retive Listinent s with Misswel d Symp nd Sympt DLI Gr.2 | ng: Par Lab. tess ssing N toms coms by | at Ba y Dose | ith grade Cycle ic Evalua P seline. Level. | e>1 Me ations at atient Gr. 2 | Exam Baselin Gr. 3 | ination date | Gr. 1 | Lab. test Tot Gr. 2 | Grad<br>CTC | AE v.4 |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 10.2.12. Si Table 10.2.12. 1 MedDRA System Organ Class | Patients Dose lev Signs an Gr. 1* n % | sterolin mg/dl retive Listi ient s with Mis vel d Symp nd Sympt DLI Gr. 2 ( n % n | Land albumg: Par Lab. tessing Moreoms by Gr. 3 | at Ba y Dose Gr. 4 n % | ith grade Cycle ic Evalua P seline. Level. Gr. 1 n % | e >1 Me ations at atient Gr. 2 n % | Exam Baselin Gr. 3 n % | ination date | Gr. 1<br>n % | Lab. test Tot Gr. 2 n % | Grad<br>CTC | AE v.4 |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 10.2.12. Si Table 10.2.12. 1 MedDRA System Organ Class Preferred Term | Patients Dose lev gns an Signs a Gr. 1* n % | trive Listinent s with Missel d Symp nd Sympt DLI Gr. 2 | Land albumg: Par Lab. tessing Moreoms by Gr. 3 | at Ba y Dose Gr. 4 n % | ith grade Cycle ic Evalua P seline. Level. Gr. 1 n % | e>1 Me ations at atient Gr. 2 n % | Exam Baselin Gr. 3 n % | ination date | Gr. 1<br>n % | Lab. test Tot Gr. 2 n % | Grad<br>CTC | AE v.4 |
| Table 10.2.11. 3 Dose level/ Table 10.2.11. 4 10.2.12. Si Table 10.2.12. 1 MedDRA System Organ Class Preferred Term | Patients Dose lev gns an Signs a Gr. 1* n % donnumbe | trive Listinent s with Missel d Symp d Symp Gr.2 | Land albumg: Par Lab. tessing Moreoms by Gr. 3 | at Ba y Dose Gr. 4 n % | ith grade Cycle ic Evalua P seline. Level. Gr. 1 n % | e>1 Me ations at atient Gr. 2 n % | Exam Baselin Gr. 3 n % tion(e.g. G | ination date | Gr. 1<br>n % | Lab. test Tot Gr. 2 n % | tal<br>Gr. 3<br>n % | AE v.4 Gr. 4 n % |

| Dose level | Patient No | Literal | | MedDRA<br>Preferred Terr | | CTCAE<br>I grade | Start | date | Relation | ship ' | Treate |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Ticiciled Tell | 1 V | rgiauc | | | | | |
| 10.2.13. | Concom | itant and Pr | ophylacti | c Medicat | ion Sta | rting P | Pre-S | tudy | • | | |
| | | nitant Medicatio | | • | | ls 1 and | 4) by | | | | |
| Medication To<br>(ATC level 1) | | on TermMedication<br>vel 2) (ATC lev | | OLI<br>% N | DLII<br>% | N | % | DL<br>N | ∠ n<br>% | N<br>N | otal<br><u>%</u> |
| Note: Percentage | es based on number | of patients by dose lev | vel. | | | | | | | | |
| | | mitant Medicati | | | | Platelet 1 | transfi | usions | /EPO). | | |
| (ATC level 1) | (ATC lev | on TermMedication<br>vel 2) (ATC lev | | OLI<br>% N | DLII<br>% | <br>N | % | DI<br>N | ∠n<br>% | To<br>N | otal<br>% |
| Platelet transfi<br>RBC transfus | | | | | | | | | | | |
| <br>Note: Percentage | es based on number | of patients by dose lev | vel. | | | | | | | | |
| | | rtive Listing: R | | | | | | Ct. 4 | Г 1 | D | C |
| | 13. 3 Supportent No Cycle | | BC and Plate<br>Literal Term | elet transfusi<br>ATC4 ATC | | | ıdy).<br> | Start<br>date | End<br>date | | son for<br>Jse |
| Dose Patie | | | | | | | | | | | son fo<br>Jse |
| Dose Patie | | | | | | | | | | | |
| Dose Patie<br>Level | ent No Cycle | Туре | Literal Term | ATC4 ATC | C2 ATC1 | Route | | | | | |
| Dose Pation Level Γable 10.2. | ent No Cycle | Type | Literal Term | ATC4 ATC | C2 ATC1 | Route | 1. | date | | J | Jse |
| Dose Patie<br>Level | ent No Cycle | Туре | Literal Term | ATC4 ATC | ne by Do | Route<br>se Leve | l. DL | date | | Tota | Jse |
| Dose Pation Level Γable 10.2. Opioids* | ent No Cycle | Type atients with Opi DLI | Literal Term ioids Treatm DLI | ATC4 ATC | ne by Do | Route<br>se Leve | l. DL | date<br>n | date | Tota | Jse<br>I |
| Dose Pation Level Γable 10.2. Opioids* | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | Literal Term<br>ioids Treatm<br>DLI<br>N | ATC4 ATC | ne by Do | Route<br>se Leve | l. DL | date<br>n | date | Tota | Jse<br>I |
| Dose Pation Level Γable 10.2. Opioids* | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI | Literal Term<br>ioids Treatm<br>DLI<br>N | ATC4 ATC | ne by Do | Route<br>se Leve | l. DL | date<br>n | date | Tota | Jse<br>I |
| Dose Pation Level Γable 10.2. Opioids* Note: (*) ATC of | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | ioids Treatm DLI N | ATC4 ATC | ne by Do % al request. | Route<br>se Leve | l. DL | date<br>n | date | Tota | Jse |
| Dose Pation Level Γable 10.2. Opioids* Note: (*) ATC of | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | Literal Term oioids Treatm DLI N will be selected and of Opioids p | ATC4 ATC | ne by Do % al request. | Route<br>se Leve | I. DL1 | date n % | date | Tota | I % |
| Dose Pation Level Fable 10.2. Opioids* Note: (*) ATC of the control of | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | Literal Term oioids Treatm DLI N will be selected and of Opioids p | ATC4 ATC | ne by Do % al request. | Route<br>se Leve | I. DL1 | date<br>n | date | Tota | I % |
| Table 10.2. Opioids* Note: (*) ATC of the control of the co | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | Literal Term oioids Treatm DLI N will be selected and of Opioids p | ATC4 ATC | ne by Do % al request. | Route<br>se Leve | I. DL1 | date n % | date | Tota | I % |
| Dose Pation Level Γable 10.2. Opioids* Note: (*) ATC of the strength | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | Literal Term oioids Treatm DLI N will be selected and of Opioids p | ATC4 ATC | ne by Do % al request. | Route<br>se Leve | I. DL1 | date n % | date | Tota | I % |
| Dose Pation Level Fable 10.2. Opioids* Note: (*) ATC of the strength of th | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | Literal Term oioids Treatm DLI N will be selected and of Opioids p | ATC4 ATC | ne by Do % al request. | Route<br>se Leve | I. DL1 | date n % | date | Tota | I % |
| Dose Pation Level Fable 10.2. Opioids* Note: (*) ATC of the state of the s | ent No Cycle 13. 4 No of pa | Type atients with Opi DLI N % | Literal Term oioids Treatm DLI N will be selected and of Opioids p | ATC4 ATC | ne by Do % al request. | Route<br>se Leve | I. DL1 | date n % | date | Tota | I % |
| Dose Pation Level Fable 10.2. Opioids* Note: (*) ATC of the state of the s | ent No Cycle 13. 4 No of parallessification includir 13. 5 Median | Type atients with Opi DLI N % ngopioids and terms w number of No o | ioids Treatm DLI N will be selected and | ATC4 ATC | ne by Do % al request. Dose Le | Route<br>se Leve | I. DL1 | date n % | date | Tota | I % |
| Table 10.2. Opioids* Note: (*) ATC of the ATC of t | ent No Cycle 13. 4 No of parallelessification including | Type atients with Opi DLI N % ngopioids and terms with opi DLI DLI | ioids Treatm DLI N vill be selected and | ATC4 ATC | ne by Do % al request. Dose Le | Route se Level | I. DL1 | date n % | date | Tota | I % |
| Dose Pation Level Fable 10.2. Opioids* Note: (*) ATC of the state of the s | ent No Cycle 13. 4 No of parallelessification including | Type atients with Opi DLI N % ngopioids and terms w number of No o | ioids Treatm DLI N vill be selected and | ent at Baseli I % N Iprovided by clinica er patient by DL II | ne by Do % al request. Dose Le | Route se Level | I. DL1 | n % | date | Tota | l % |

| Ctouri dak | I | OLI | DL | II | | • | D | L <b>n</b> | To | ıtal |
|---|---|---|---|---|---|---|---|---|---|---|
| Steroids* | N | % | N | % | N | % | N | % | N | % |
| ••• | | | | | | | | | | |
| Note: (*) The ATC classif | ication, includings | steroids and term | rs, will be sele | cted and pro | ovided by clini | cal request. | | | | |
| Гable 10.2.13. 7 К | Lnown CYP ( | 3A4 Induce | ers/Inhibit | ors/Sub | strates Co | ncomitan | t Therap | ies at BL | | |
| CVD 2 A 4* | I | OLI | DL | II | • • | • | D | Ln | To | otal |
| CYP 3A4* | N | % | N | % | N | % | N | % | N | % |
| Inhibitor | | | | | | | | | | |
| ••• | | | | | | | | | | |
| Notes: (*) Also the possib | ility of displaying | one table for ea | ch category Ir | nducers/Inhi | bitors or subst | rates. Some r | nedication v | vill be exclud | ed by clinical | l request |
| Dexamethasone). | | | | | | | | | | |
| Table 10.2.13. 8 L | isting of CY | P 3A4 Indu | acers/Inhi | bitors/Si | ubstrates ( | Concomit | ant Ther | apies at I | BL. | |
| _ | Type* | Literal Tem | n ATC | ATC2 | ATC1 | Star | End | Reason for | rUse SS/A | AE Spec |
| Dose Patno | - 71 | | | | | | | | | |

Notes: (\*) Also the possibility of display onetable for each category Inducers/Inhibitors or substrates. Some medication will be excluded by clinical request (e.g. Dexamethasone).

## 11. Appendix II. Safety Evaluation.

All statistical outputs in this section, whenever applicable, will be displayed according to the discontinuation of the combination treatment. Treatment exposure, delays, omissions and reductions will be shown considering the whole study treatment and/or before and after discontinuation, if appropriate.

Dose level may suffer categorization (e.g.  $RD \le or RD$ , Cohorts/Cancer type or primary site/CSF use or not/other clinical relevant variable), if required and if an adequate number of patients is represented.

Each specific table and listing will have a comprehensive header identifying the group/cohort of treatment, whenever necessary.

Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

## 11.1.Extent of Exposure.

#### 11.1.1. Cumulative Dose, Dose Intensity and Relative Dose Intensity.

Table 11.1.1.1 No of Cycles Administered by Dose Level.

| | | | | Patients |
|---|---|---|---|---|
| Dagalaval | | No. of | No. of patients | No. of patients |
| Dose level | cyc | les infused | with PM01183+Doxo | with PM01183 alone |
| | 1 Cycle | | | |
| I | 1 Cycle<br>2 Cycles | | | |
| П | 1 Cycle | | | |
| 11 | 2 Cycles | | | |
| ••• | | | | |
| | 1 Cycle | | | |
| N | 2 Cycles | | | |
| | 1 Cycle | | | |
| Total | 2 Cycles | | | |
| 10121 | | | | |
| | N Cycles | | | |

Table 11.1.1.2 Median and Range of Cycles Administered by Dose Level.

| Drug | Median range and STD of<br>cycles administered | DLI | DLII | <br>DL n | Total |
|---|---|---|---|---|---|
| PM01183+Doxorubicin | N* | | | | |
| PM01183 alone | N* | | | | |
| Total | N* | | | | |

Note: (\*) N, median, mean, range, and STD.

Table 11.1.1.3 Cumulative Dose by Dose Level.

| Drug | Cumulative dose | DLI | DLII | <br>DL n | Total |
|-------------|-----------------|-----|------|----------|-------|
| | N | | | | |
| | Mean | | | | |
| PM01183 | Median | | | | |
| (mg) | Min | | | | |
| | Max | | | | |
| | STD | | | | |
| | N | | | | |
| | Mean | | | | |
| Doxorubicin | Median | | | | |
| $(mg/m^2)$ | Min | | | | |
| , , | Max | | | | |
| | STD | | | | |

Table 11.1.1.4 Dose Intensity by Dose Level.

| Drug | Dose intensity | DLI | DLII | • • • | DL n | Total |
|--------------|----------------|-----|------|-------|------|-------|
| | N | | | | | |
| | Mean | | | | | |
| PM01183* | Median | | | | | |
| (mg/week) | Min | | | | | |
| | Max | | | | | |
| | STD | | | | | |
| | N | | | | | |
| | Mean | | | | | |
| PM01183* | Median | | | | | |
| (mg/m²/week) | Min | | | | | |
| | Max | | | | | |
| | STD | | | | | |
| | N | | | | | |
| | Mean | | | | | |
| Doxorubicin | Median | | | | | |
| (mg/m²/week) | Min | | | | | |
| | Max | | | | | |
| | STD | | | | | |

<sup>(\*)</sup> Results of dose intensity may be grouped and presented in mg/m²/week for patients treated in the Cohort A, if appropriate.

Table 11.1.1.5 Relative Dose Intensity by Dose Level.

| Drug | Relative dose intensity (%) | DLI | DLII | <br>DL n | Total |
|---|---|---|---|---|---|
| PM01183 | N<br>Mean<br>Median<br>Min<br>Max<br>STD | | | | |
| Doxorubicin | N<br>Mean<br>Median<br>Min<br>Max<br>STD | | | | |

| Table 11.1.1.6 Drug Administration: Patients that Reached the Maximal Cumulative Dose of 450 mg/m <sup>2</sup> . |
|---|
|---|

| Dose level | Patient No | No. of Cycles<br>PM01183 | No. of Cycles<br>Doxorubicin | Delay | Delay specify | * |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

Note: (\*) Delays, omissions, reductions and specify.

## 11.1.2. Cycle Delays and Omissions.

Table 11.1.2.1 No of Patients with Delayed Cycles by Dose Level.

| No of patients with delayed | D | DLI | | DLII | | • • • | | DL n | | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| cycles | N | % | N | % | N | % | N | % | N | % |

No

Yes

Any DR\*

All NDR\*\*

Total

Notes: Percentages based on number of patients by dose level. (\*) Drug related (\*\*) Non-drug related.

Table 11.1.2.2 No of Patients with Dose Delayed by Dose Level According to Relationship.

| No of | av valas dalav vad | Γ | DLI | DI | LII | • • • | | DL n | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 110 01 0 | cycles delayed | N | % | N | % | N | % | N | % | N | % |
| No | | | | | | | | | | | |
| Yes | Drug Related | | | | | | | | | | |

Hematological Non Hematological Both

Non Drug Related

Total

Note: Percentages based on number of cycles susceptible of delay by dose level.

Table 11.1.2.3 No of Cycles Delayed Per Patient by Dose Level.

| No motionto ve itle . | DLI | | DLII | | • • • | | D | DL n | | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| No patients with: | N | % | N | % | N | % | N | % | N | % |
| No cycle delayed | | | | | | | | | | |
| 01 cycle delayed | | | | | | | | | | |
| 02 cycles delayed | | | | | | | | | | |
| ••• | | | | | | | | | | |
| N cycles delayed | | | | | | | | | | |
| Total | | | | | | | | | | |

Note: Percentages based on number of patients by dose level.

Table 11.1.2.4 No of Cycles Delayed Per Patient by Dose Level. Summary Statistics.

| No patients with delays | DLI | DLII | • • • | DL n | Total |
|-------------------------|-----|------|-------|------|-------|
| N | | | | | |
| Median | | | | | |
| Min<br>Max | | | | | |
| Max | | | | | |
| STD | | | | | |

Table 11.1.2.5 Number of Cycles with Drug Related Delay per Patient by Dose Level. DLI DLII DL n Total No cycles with: N % N % N % N % % N No cycle delayed 01 cycle delayed 02 cycles delayed N cycles delayed Total Table 11.1.2.6 Number of Cycles with Drug Related Delay per Patient by Dose Level. Summary Statistics. No cycles with delays DLI DLII DL n Total N Median Min Max STD Table 11.1.2.7 Length of Delay According to relationship by Dose Level. Summary Statistics. Relationship Total DLI DLII DL n Hematological N Mean Median Min Max STD Non Hematological N Mean Median Min Max **STD** Both N Mean Median Min Max **STD** Total N Mean Median Min Max STD

| Dose level | Patient No | Cycle | Date | Intended dose | Total dose | Length of<br>Delay | Delay<br>Reason | Delay s <sub>l</sub> | ecify |
|---|---|---|---|---|---|---|---|---|---|
| Γable 11.1. | 2.9 Supporti | ve Listing: 1 | Dose Dela | nys Excluding A | dministrativ | e Reasons. | | | |
| Dose level | Patient No | Cycle | Date | Intended dose | Total dose | Length of<br>Delay | Delay<br>Reason | Delay s <sub>l</sub> | ecify |
| Note: (*) Exclud | ling administrative | reasons. | | | | | | | |
| Гable 11.1. | 2.10 No. of l | | | oicin Omissions | by Dose Le | | | | |
| | s with any dosag | | LI | DLII | • • • | | DL n | Tot | |
| omitted | | N | % | N % | N | % N | % | N | % |
| Omitted | | | | | | | | | |
| Maintained | | | | | | | | | |
| Total | es based on numbe | | | | | | | | |
| | 2.11 No of Powith cycles | atients with | Doxorub | icin Cycles Omi | ission by Do | | L n | Tota | 1 |
| No of patients<br>omitted<br>No omission<br>cycle | | DLI | Doxorub<br>% N | DLII | · | D | L n<br>% | Tota<br>N | 1 % |
| No of patients omitted No omission cycle cycles Fotal | s with cycles | DLI<br>N | % N | DLII | | D | | | |
| No of patients omitted No omission I cycle 2 cycles Fotal Note: Percentag | | DLI<br>N s | % N ose level. | DLII N % Omissions. | | DA On | % nission | | % |
| To of patients mitted To omission cycle cycles Cotal Total Table 11.1. Dose lev | es based on number 2.12 Listing el Patien 2.13 Listing | DLI<br>N Seriof patients by door of Doxorub<br>t No Cy | oselevel. | Omissions. DA Start DA in Date to Hematologic ober of Cycle number of with dose | nfusion omittee | Di<br>N<br>d? DA On<br>reas | nission<br>on | N | <u>%</u> |

Notes: (\*/\*\*) Also Leukopenia /CSF, Anemia / EPO, Thrombocytopenia / platelet transfusions. Narratives with the information contained in the tables will be provided instead of tables only if a low number of dose delays occur.

| Dose level | Patient No | Total numl<br>cycles rece | with dose | delays Cy | cle numbers wi<br>lelays not due to | | cle numbers witho<br>lequate prophylaxis |
|---|---|---|---|---|---|---|---|
| Notes: (*)Adverse event. N | farratives with the in | nformation contained i | n the tables will be pro | vided instead | oftables only if a lo | w number of do | ose delays are found. |
| 11.1.3. Dose R | eductions. | | | | | | |
| Гable 11.1.3.1 No | of Patients w | rith PM01183 I | Dose Reduction | hy Dose | I evel | | |
| No of patients with an | | DLI | DLII | | | DL n | Total |
| nodified | | N % | N % | N | % N | | N % |
| Reduced | | | | | | | |
| No reduced | | | | | | | |
| Total . | | | | | | | |
| Note: Percentages based or | n number of patient | s by dose level. | | | | | |
| Table 11.1.3.2 No | | | | duction b | | | |
| No of patients with cy | | LI | DLII | | | DL n | Total |
| educed | N | % N | % | N | % N | % | N % |
| reduction | | | | | | | |
| 2 reductions | | | | | | | |
| Гotal | | | | | | | |
| Note: Percentages based or | number of patient | s by dose level. | | | | | |
| C | • | | | | | | |
| Гable 11.1.3.3 Re | asons for PM | 01183 Dose Re | eduction by Dos | se Level. | | | |
| | | DLI | DLII | | • | DL n | Total |
| No of patients with cy | cies reduced | N % | N % | N | % N | <b>1</b> % | N % |
| No dose reduction | | | | | | | |
| Hematological | | | | | | | |
| Non-hematological | | | | | | | |
| Both (hematological a | nd non- | | | | | | |
| nematological)<br>Other | | | | | | | |
| Total | | | | | | | |
| | number of patients | s by dose level. | | | | | |
| Note: Percentages based or | • | - | | | | | |
| Note: Percentages based or | | | | | | | |
| - | ting of PM01 | 183 Dose Redi | actions. | | | | |
| Гable 11.1.3.4 Lis | ting of PM01 | DA Start | uctions. DA infusion | ۰ ۵/ ۵ | reduction [ | DA Reduce | Specify |

| Dose level | Patient N | NO. | number of<br>s received | Cycle numbers with dose reduction due to* | Cycle<br>reduc | numbers with a<br>tion not due to . | dose<br>* Cycle nu | mbers with* |
|---|---|---|---|---|---|---|---|---|
| Notes: (*/**) Also Leukoj | penia/CSF, Anemi | ia/EPO, Thromb | ocytopenia/p | olatelet transfusions. | | | | |
| Гable 11.1.3.6 Li | sting of Dose | e Reductions | s due to N | on-Hematologic | cal Ad | verse Events | | |
| Dose level | Patient N | NO. | number of<br>s received | Cycle numbers with dose reduction due to* | | numbers with a<br>tion not due to . | | umbers withou<br>ate prophylaxis |
| lote: (*) Adverse event. 1.1.4. Dose I | nterruptio | on and Re | -admini | istration. | | | | |
| Γable 11.1.4.1 L | isting of Pati | ents with Do | ose Interru | • | dminis | tration. | | |
| Table 11.1.4.1 L Dose level Patient | | ents with Do<br>Infusion Day<br>1/Day 8 | | uption and Re-active Was infusion interrupted? Reason | | tration. Intended dose | Total dose | Total Volum |
| Dose level Patient 11.2.Dose-La | imiting T | Infusion Day 1/Day 8 Toxicities oxicities. | Drug | Was infusion interrupted? Reason | | | Total dose | Total Volum |
| Dose level Patient | imiting T | Infusion Day 1/Day 8 Coxicities oxicities. | Drug | Was infusion interrupted? Reason | | | Total dose Patients with | |

## 11.3. Adverse Events (AEs).

#### 11.3.1. Display of Adverse Events.

All adverse events tables will be listed by cohort and dose level (or most adequate dose grouping/tumor type/other clinical relevant variable or according to the discontinuation of the combination treatment, if required).

- Table 11.3.1.1 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events. Worst Grade by Patient and Dose Level.
- Table 11.3.1.2 PM01183-Only Related (or Relationship Unknown) Adverse Events. Worst Grade by Patient and Dose Level.
- Table 11.3.1.3 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events. Worst Grade by Patient and Dose Level.
- Table 11.3.1.4 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events in the First Cycle by Patient and Dose Level.
- Table 11.3.1.5 PM01183-Only Related (or Relationship Unknown) Adverse Events in the First Cycle by Patient and Dose Level.
- Table 11.3.1.6 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events in the First Cycle by Patient and Dose Level.
- Table 11.3.1.7 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events. Worst Grade Per Cycle by Dose Level.
- Table 11.3.1.8 PM01183-Only Related (or Relationship Unknown) Adverse Events. Worst Grade Per Cycle by Dose Level.
- Table 11.3.1.9 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events. Worst Grade Per Cycle by Dose Level.
- Table 11.3.1.10 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated by Dose Level.
- Table 11.3.1.11 PM01183-Only Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated by Dose Level.
- Table 11.3.1.12 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated by Dose Level.
- Table 11.3.1.13 Combination (PM01183-Doxorubicin) Related (or Relationship Unknown) Adverse Events Observed in ≥ 10% of Patients Treated. Worst grade per Cycle by Dose Level.
- Table 11.3.1.14 PM01183-Only Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated. Worst grade per Cycle by Dose Level.
- Table 11.3.1.15 Doxorubicin-Only Related (or Relationship Unknown) Adverse Events Observed in ≥10% of Patients Treated. Worst grade per Cycle by Dose Level.
- Table 11.3.1.16 Adverse Events Regardless of Relationship. Worst Grade by Patient by Dose Level.
- Table 11.3.1.17 Adverse Events Regardless of Relationship in the First Cycle by Patient and Dose Level.
- Table 11.3.1.18 Adverse Events Regardless of Relationship. Worst Grade per Cycle by Dose Level.
- Table 11.3.1.19 Adverse Events Observed in  $\geq$  10% of Patients Treated by Dose Level.
- Table 11.3.1.20 Adverse Events Observed in ≥ 10% of Patients Treated. Worst grade per Cycle by Dose Level.

Tables 11.3.1.1-.20 will have the following pattern but DL and Grade column might be grouped if required.

| MedDRA System Organ | DLI | • • • | DLn | Total |
|---|---|---|---|---|
| Class | Gr.1 Gr.2 Gr.3 Gr.4 | Gr.1 Gr.2 Gr.3 Gr.4 G | Gr.1 Gr.2 Gr.3 Gr.4 | Gr.1 Gr.2 Gr.3 Gr.4 |
| Preferred Term | n % n % n % n % | n % n % n % n % 1 | n % n % n % n % | $n\ \%\ n\ \%\ n\ \%\ n\ \%$ |

Note: Percentages based on number of patients/cycles by dose level.

Table 11.3.1.21 Supportive Listing: Drug Related (or Relationship Unknown) Adverse Events Grade 3-4 by Dose Level.

| Dose level Patient SO | MedDRA<br>C Preferred<br>Term | Literal<br>term | Grade | SAE<br>(Y/N) | Onset<br>Date | Resolved Date | Relationship<br>to Study<br>Drug | Action<br>Taken | Main<br>Consequence |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

Table 11.3.1.22 Time to course to Alopecia Grade >1.

| Doga laval | Dations | Grade at | Cendo | Owart Data | Resolved | Times in days * A stiger Talyan | Main |
|---|---|---|---|---|---|---|---|
| Dose level | Patient | Baseline | Grade | Onset Date | Date | Time in days * Action Taken | Consequence |

<sup>(\*)</sup> Time in days calculated as the difference between Onset date and DA first drug administration.

#### 11.4.Deaths and Other Serious Adverse Events.

#### 11.4.1. Deaths.

Table 11.4.1.1 Patients who Died While on Treatment.

| Dose | Patient | Last cycle | Last infusion | Death | Time from last | Course | Commonts | Time on treatment |
|---|---|---|---|---|---|---|---|---|
| level | No | received | date | date | infusion date (days) | Cause | Comments | (weeks) |
| | | | | | | | | _ |

Note: Patients with death reported as end of treatment reason.

Table 11.4.1.2 Patients Who Died Within 30 Days of Last Drug Administration.

| Dose | Patient | Last cycle | Last infusion | Death | Time from last | Course | Commonts | Time on treatment |
|---|---|---|---|---|---|---|---|---|
| level | No | received | date | date | infusion date (days) | Cause | Comments | (weeks) |

Table 11.4.1.3 Listing of All Deaths.

| Dose Patient Last cycle | Last | | | | | Time on | Time from last |
|---|---|---|---|---|---|---|---|
| - | infusion | Death date | Cause | Comments | Autopsy | treatment | infusion date |
| level No received | date | | | | 1 0 | (weeks) | (days) |

#### 11.4.2. Serious Adverse Events.

All serious adverse events will be listed only for the purpose of reconciliation with the database of pharmacovigilance. The listings provided by the Product Safety department will be used for the clinical study report.

| Table | 11 | 421 | A 11 | SAEs. |
|--------|----|-----|------|-------|
| 1 autc | 11 | | 7111 | DIL. |

| Dose<br>level Patient Cycle System Organ<br>Class | Preferred<br>Term Grade | AE<br>Status | AE<br>relationship | AE consequences | SAE | Onset<br>date | Resolved date |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

## 11.5. Clinical Laboratory Evaluation.

## 11.5.1. Hematological Abnormalities.

Table 11.5.1.1 Hematological Abnormalities: Worst Grade per Patient by Dose Level.

Table 11.5.1.2 Hematological Abnormalities: Worst Grade per Cycle by Dose Level.

Table 11.5.1.3 Hematological Abnormalities: Worst Grade per patient in the First Cycle by Dose Level.

Tables 11.5.1.1-.3 will have the following pattern but DL and Grade columns might be grouped if required.

| Abnormality* | DLI | DLII | • • • | DL n | Total |
|--------------------|-----|------|-------|------|-------|
| Anemia | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |
| **** | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |

Notes: Percentage s based on number of patients by dose level. (\*) Also Leukopenia, Lymphopenia, Neutropenia, and Thrombocytopenia

Table 11.5.1.4 Supportive Listing: Patients with Grade 4 Hematological Abnormalities.

| date | Dose level | Patient | Lab. test | Cycle | Examination date | * |
|------|------------|---------|-----------|-------|------------------|---|
|------|------------|---------|-----------|-------|------------------|---|

Notes: (\*) Include the following: Value at BL, Grade at BL, Onset day, Onset grade, Nadir day, Nadir value, Nadir grade, Recovery day, Recovery value, Recovery grade, Days Grade 4.

Table 11.5.1.5 Patients with Missing Hematological Evaluations.

| Dose level/CSF | Patient | Cycle | Lab. test |
|----------------|---------|-------|-----------|

| Dose level/CSF Patient | Cycle | Lab. test |
|------------------------|-------|-----------|

Table 11.5.1.6 Shift of Hematological Abnormalities. Baseline Grade vs. Worst Grade on First Cycle.

| | | | | | Worst | Grade o | on First | Cycle | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose level | /Parameter* | Baseline Grade | G | r. 1 | G | r. 2 | G | r.3 | Gı | :4 |
| | | | N | % | N | % | N | % | N | % |
| | Anemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| DLI | | 4 | | | | | | | | |
| DLI | | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Anemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| ••• | | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Anemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| T-4-1 | | 4 | | | | | | | | |
| Total | | 0 | | | | | | | | |
| | | 4 | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) Also Leukopenia, Lymphopenia, Neutropenia and Thrombocytopenia.

Table 11.5.1.7 Shift of Hematological Abnormalities. Baseline Grade vs. Worst Grade on Treatment.

| | | | | Wo | orst Gra | nde duri | ng on T | reatme | nt | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose level/ | Parameter* | Baseline Grade | G | r. 1 | G | r. 2 | G | r.3 | Gı | :4 |
| | | | N | % | N | % | N | % | N | % |
| | Anemia | 0 | | | | | | | | |
| DLI | | 4 | | | | | | | | |
| DLI | | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Anemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| ••• | ••• | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Anemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| Total | | 4 | | | | | | | | |
| rotar | | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |

 $Notes: Percentages \ based \ on number \ of patients \ by \ dose \ level. (***) \ Leukopenia, \ Lymphopenia, \ Neutropenia \ and \ Thrombocytopenia.$ 

| Dose level | om Baseline. Patient | Event* | NCI-CTCAE v.<br>at baseline | 4 NCI-CTCAF<br>at Cycle | Ev.4 | Cycle |
|---|---|---|---|---|---|---|
| ble 11.5.1.9 Sum Dose Level | mary of Characte Parameter | eristics of wpp<br>N(%)* | Hematological Ab<br>Mean** | normailities G3-<br>"*Median | | Range** |
| Dose Level | Tatarroor | 1 (70) | Ivicui | TVICARAI | · | range |
| es: (*) Percentages based | on number of patients by | / dose level with grade | e 3-4. (**) Cycle occurrenc | е. | | |
| ble 11.5.1.10 Sur | nmary of Hemat | ological Abnor | malities Grade 4 a | _ | sfusions/treat | ment. |
| Dose level | Patient | Cycles received | Cycle number wit<br>hematological abnom<br>*<br>grade 4 | | • | numbers w<br>se reduction |
| (*) N + | 1 | 4:- /Dl-4-1-4-4- | £ | 0 | | |
| | | | nnsfusion and Anemia/EF<br>per Dose Level in | | | |
| | | | | Worst Grade on Tre | | |
| | EPO/Dose Level | | Gr. 1-2<br>N % | Gr. 3<br>N % | Gr. 4<br>N % | Total<br>N |
| EPO | DLI | | | | | |
| ЦО | | | | | | |
| No EPO | DLI | | | | | |
| NOLIO | | | | | | |
| bla 11 5 1 12 Da | tionts with Anom | via Grada 2/4 ar | nd Uga af EDO in | Cyalo >1 | | |
| Dose Level | Tumor type | Patno | nd Use of EPO in Cycle | Prophylaxis CSF (Y | 7N) | * |
| | Jr · | | | 1 3 2 2 2 (2 | | |
| es: (*) Grade, nadir day to<br>vals in days might chang | | to grade≤3,** duratio | on in days to grade 3**, (** | ) Grade 2 or 1 also if clin | ically indicated (** | **)Numeric |
| ble 11.5.1.13 Pla | atelet Count Time | e Course Patter | n (summary). | | | |

| | Parameter* | | DLI | ••• | DL n |
|---|---|---|---|---|---|
| | | Pla | atelet transfusion | | |
| | | | N Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day grade 4 | 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade >0 | Onset day grade 4 | 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| | | No l | Platelet transfusion | | |
| | | | N Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day grade 4 | 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade >0 | Onset day grade 4 | 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| | | | Totals | | |
| | | | N Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day grade 4 | 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade > 0 | Onset day grade 4 | 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |

Notes: (\*) Also nadir day grade 4, nadir value grade 4, recovery day to grade  $\leq$  3, duration in days to grade  $\leq$  3, duration in days to grade  $\leq$  2, duration in days to grade  $\leq$  2, duration in days to grade  $\leq$  1 and duration in days to grade 1. Grade limits may change under request.

Table 11.5.1.14 Platelet Count Time Course Pattern.

| Parameter* | | | DLI | • • • | | | DL n |
|---|---|---|---|---|---|---|---|
| | P | latelet tr | ansfusion | | | | |
| | Onset day grade 4 | N | % | N | % | N | % |
| | ≤7*** | | | | | | |
| 1 <sup>st</sup> cycle | 8-14 | | | | | | |
| | ≥15 | | | | | | |
| | ≤7 | | | | | | |
| Cycle>1 | 8-14 | | | | | | |
| | ≥15 | | | | | | |
| | ≤7 | | | | | | |
| 1 <sup>st</sup> cycle | 8-14 | | | | | | |
| | ≥15 | | | | | | |
| | ≤7 | | | | | | |
| Cycle>1 | 8-14 | | | | | | |
| | ≥15 | | | | | | |
| | No | Platelet | transfusion | | | | |
| Ons | et day grade 4 | N | % | N | % | N | % |
| | ≤7 | | | | | | |
| | 8-14 | | | | | | |
| | ≥15 | | | | | | |
| | 1st cycle Cycle>1 1st cycle Cycle>1 Ons | Onset day grade 4 1 <sup>st</sup> cycle | Platelet tra Onset day grade 4 N 1st cycle | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Platelet transfusion Onset day grade 4 N % N % N Solid Service S-14 S-15 S- |

| | Paramet | er* | | DLI | • • • | | | DL n |
|---|---------|-------------------|--------|-----|-------|---|---|------|
| | | ≤7 | | | | | | |
| | | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | | Totals | | | | | |
| | | Onset day grade 4 | N | % | N | % | N | % |
| | | ≤7 | | | | | | |
| | | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | ≤7 | | | | | | |
| | | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| * | • | | | | | | | |

Note: (\*) Also nadir day to grade 4, recovery day to grade  $3^{**}$ , duration in days to grade  $3^{**}$ , (\*\*) Grade 2 or 1 also if clinically indicated, (\*\*\*) Numeric intervals in days might change upon request.

Table 11.5.1.15 Thrombocytopenia wpp/wpc and Use of Transfusions per Dose Level in Cycle>1.

| 140.0 1110.1110 1111.0110.000 | | Worst Grade on Treatment*/Cycle* | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Tansfusion/D | Oose Level | Gr. 1-2 | | Gr.3 | | G | r. 4 | To | tal |
| | | N | % | N | % | N | % | N | % |
| DLI<br>Transfusion | | | | | | | | | |
| Hansusion | | | | | | | | | |
| N.T. C. | DLI | | | | | | | | |
| No Transfusion | | | | | | | | | |

<u>Table 11.5.1.16</u> Patients with Thrombocytopenia Grade 3/4 and Use of Transfusions in Cycle >1.

| Dose Level Tumor type Patno Cycle Prophylaxis CSF (Y/N) * |
|-----------------------------------------------------------|
|-----------------------------------------------------------|

Notes: (\*) Grade, nadir day to grade 3/4, recovery day to grade  $\leq$ 3, (\*\*) duration in days to grade 3\*\*, (\*\*) Grade 2 or 1 also if clinically indicated (\*\*\*\*) Numeric intervals in days might change upon request.

Table 11.5.1.17 Summary of Hematological Abnormalities Grade 4 and Specific Transfusions.

| | | | Cycle number with | | |
|---|---|---|---|---|---|
| Dose level | Patient | Cycles received | hematological<br>abnormality* | Cycle numbers with** | Cycle numbers with dose reduction |
| | | | grade 4 | | |

Note: (\*) Also Neutropenia/CSF administration. Thrombocytopenia/Platelets transfusion and Anemia/EPO transfusions.

Table 11.5.1.18 Neutrophil Count Time Course Pattern (summary).

| Table 11.5.1.18 f | Neutrophii Count | i ime Course P | attern (summary). | | |
|---|---|---|---|---|---|
| | Parameter* | | DLI | ••• | DL n |
| | | | CSF use | | |
| | | N | Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day grade 4 | 1 <sup>st</sup> cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade >0 | Onset day grade 4 | 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| | | | No CSF | | |
| | | | N Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day grade 4 | 1 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade >0 | Onset day grade 4 | 1 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| | | | Totals | | |
| | | | N Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day grade 4 | 1 1st cycle | | | |
| | | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade >0 | Onset day grade 4 | 1 1st cycle | _ | _ | |
| | | Cycle>1 | | | |
| | | Total | | | |

Note: (\*) Also nadir day grade 4, nadir value grade 4, recovery day to grade ≤ 3, duration in days to grade 3, recovery day to grade ≤ 2, duration in days to grade ≤ 1, recovery day to grade ≤ 1 and duration in days to grade 1.

Table 11.5.1.19 Platelet Count Time Course Pattern.

| | Parameter* | | | DLI | • • • | | | DL n |
|---|---|---|---|---|---|---|---|---|
| | | | Platelet tr | ansfusion | | | | |
| ( | Onset day grade 4 | | N | % | N | % | N | % |
| Baseline grade 0 | | ≤7 <b>***</b> | | | | | | |
| | 1 <sup>st</sup> cycle | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | ≤7 | | | | | | |
| | Cycle>1 | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| Baseline grade > 0 1st cycle | | ≤7 | | | | | | |
| | 1 <sup>st</sup> cycle | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | ≤7 | | | | | | |
| | Cycle>1 | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | N | o Platelet | transfusion | | | | |
| ( | Onset day grade 4 | | N | 0/ | o N | % | N | % |
| •••• | | ≤7 | | | | | | |
| | | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | - | | | | | | |

| | Parameter* | | DLI ··· | DL n |
|---|------------|-------------|---------|------|
| | | ≤7 | | |
| | | 8-14 | | |
| | | 8-14<br>≥15 | | |
| | | | Totals | |
| | | ≤7 | | |
| | | 8-14 | | |
| | | ≥15 | | |
| | | <b>≤</b> 7 | | |
| | | 8-14 | | |
| | | 8-14<br>≥15 | | |
| * | • | | | |

Notes: (\*) Also nadir day to grade 4, recovery day to grade  $\leq$ 3\*\*, duration in days to grade 3\*\*, (\*\*) Grade 2 or 1 also if clinically indicated, (\*\*\*) Numeric intervals in days might change upon request.

Table 11.5.1.20 Neuthropenia wpp/wpc and Use of Prophylactic CSF per Dose Level in Cycle>1

| | | Worst Grade on Treatment*/Cycle* | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Tansfusion | n/Dose Level | Gr. 1-2 | | Gr.3 | | Gr.4 | | To | tal |
| | | | % | N | % | N | % | N | % |
| CSE | DLI | | | | | | | | |
| CSF | | | | | | | | | |
| No CSF | DLI | | | | | | | | |

Table 11.5.1.21 Patients with Neutrophenia Grade 3/4 and Use of Prophylactic CSF in Cycle >1.

| Dose Level | Tumortype | Patno | Cycle | Prophylaxis CSF (Y/N) | * |
|------------|-----------|-------|-------|-----------------------|---|
|------------|-----------|-------|-------|-----------------------|---|

<sup>(\*)</sup> Grade, nadir day to grade 3/4, recovery day to grade ≤3, (\*\*) duration in days to grade 3\*\*, (\*\*) Grade 2 or 1 also if clinically indicated (\*\*\*) Numeric intervals in days might change upon request.

#### 11.5.2. Biochemical Abnormalities.

AP

Table 11.5.2.1 Biochemical Abnormalities: Worst Grade per Patient by Dose Level.

Table 11.5.2.2 Biochemical Abnormalities: Worst Grade per Cycle by Dose Level.

Table 11.5.2.3 Biochemical Abnormalities: Worst Grade per Patient in the first Cycle by Dose Level.

Tables 11.5.2.1-.3 will have the following pattern but Grade column might be grouped if required.

| Abnormality* | DLI | DLII | • • • | DL n | Total |
|--------------|-----|------|-------|------|-------|

| Abnormality* | DLI | DLII | • • • | DL n | Total |
|--------------------|-----|------|-------|------|-------|
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |
| ** | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) All biochemical abnormalities susceptible to be graded with NCI-CTCAE v.4.

Table 11.5.2.4 Patients with Missing Biochemical Evaluation.

| Table 11.5.2.4 Tatients with With | sing Diochemical Lva. | iuation. | |
|---|---|---|---|
| Dose level | Patient | Cycle | Lab. test |

Table 11.5.2.5 Shift of Biochemical Abnormalities. Baseline Grade vs. Worst Grade on First Cycle.

| | | | | | Wor | st Grad | e on Cy | cle 1 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose le | vel/Parameter | Baseline Grade | G | Gr. 1 | | r. 2 | G | r. 3 | G | r.4 |
| | | | N | % | N | % | N | % | N | % |
| | AP increase | 0 | | | | | | | | |
| DLI | | 4 | | | | | | | | |
| DLI | | 0 | | | | | | | | |
| | AD: | 4 | | | | | | | | |
| | AP increase | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| ••• | | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | AP increase | 0 | | | | | | | | |
| Tr. 4.1 | | 4 | | | | | | | | |
| Total | | 0 | | | | | | | | |
| | | 4 | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) All biochemical abnormalities susceptible to be graded with NCI-CTCAE v.4.

Table 11.5.2.6 Shift of Biochemical Abnormalities. Baseline Grade vs. Worst Grade on Treatment.

| Dose level/Parameter | | | Worst Grade on Treatment | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline Grade | Gr. 1 | | Gr.2 | | Gr.3 | | Gı | r. 4 |
| | | | N | % | N | % | N | % | N | % |
| | AP increase | 0 | | | | | | | | |
| DLI | | ••• | | | | | | | | |
| DLI | | 4 | | | | | | | | |
| | | 0 | | | | | | | | |

| | | ••• |
|-------|-------------|-----|
| | | 4 |
| | AP increase | 0 |
| | | 4 |
| ••• | ••• | 0 |
| | | 4 |
| | AP increase | 0 |
| | | ••• |
| T-4-1 | | 4 |
| Total | | 0 |
| | | 4 |

Notes: Percentages based on number of patients by dose level. (\*) All biochemical abnormalities susceptible to be graded with NCI-CTCAE v.4.

Table 11.5.2.7 Listing of patients with Biochemical Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline.

| Dose level | Dationt | Ex zont* | NCI-CTCAE v4 at | NCI-CTCAE v4 | Curlo |
|------------|---------|----------|-----------------|--------------|-------|
| Dose level | Patient | Event* | baseline | at Cycle | Cycle |

Note: (\*) For nausea and vomiting events, other table will be provided and use or not of antiemetic will be added.

Table 11.5.2.8 Summary of Characteristics of wpp Biochemical Abnormalities G3-4.

| | _ | 3.74 | | 3 5 11 ded. | The state |
|------------|-----------|------|--------|-------------|-----------|
| Dose Level | Parameter | N* | Mean** | Median** | Range** |

Notes: (\*) Percentages based on number of patients by dose level. with grade 3-4. (\*\*) Cycle occurrence.

Table 11.5.2.9 AST/ALT Count Time Course Pattern (summary).

| _ | Parameter* | | DLI | | DL n |
|---|---|---|---|---|---|
| | | | N Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day | 1 <sup>st</sup> cycle | | | |
| | grade 3-4 | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade > 0 | Onset day | 1 <sup>st</sup> cycle | | | |
| | grade 3-4 | Cycle>1 | | | |
| | | Total | | | |
| | | | Totals | | |
| | | | N Median Range | N Median Range | N Median Range |
| Baseline grade 0 | Onset day | 1 <sup>st</sup> cycle | | | |
| _ | grade 3-4 | Cycle>1 | | | |
| | | Total | | | |
| Baseline grade > 0 | Onset day | 1 <sup>st</sup> cycle | | | |
| • | grade 3-4 | Cycle>1 | | | |
| | | Total | | | |

Note: (\*) Also Onset day grade 3-4, Peak day grade 3-4, Peak value grade 3-4, Recovery\* day to grade ≤2, Duration in days to grade 2, Recovery day to grade ≤1, Duration in days to grade 1. Grade limits may change under request.

Table 11.5.2.10 AST/ALT Count Time Course Pattern.

| | Parameter | | | DLI | • • • | | | DL n |
|---|---|---|---|---|---|---|---|---|
| | Onset day<br>grade 3-4 | | N | % | N | % | N | % |
| Baseline grade 0 | | ≤7 <b>**</b> * | | | | | | |
| | 1 <sup>st</sup> cycle | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | ≤7 | | | | | | |
| | Cycle>1 | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| Baseline grade >0 | | ≤7 | | | | | | |
| | 1 <sup>st</sup> cycle | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | ≤7 | | | | | | |
| | Cycle>1 | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | | Tot | als | | | | |
| Ons | set day grade 3- | 4 | N | 9/ | % N | % | N | % |
| | | ≤7 | | | | | | |
| | | 8-14 | | | | | | |
| | | ≥15 | | | | | | |
| | | ≤7 | | | | | | |
| | | 8-14 | | | | | | |
| | | ≥15 | | | | | | |

Notes: (\*) Also Peak day to grade 3-4, recovery day to grade  $2^{**}$ , duration in days to grade  $2^{**}$ , (\*\*) Grade 1 also if clinically indicated (\*\*\*) Numeric intervals in days might change upon request.

#### 11.5.3. Other Metabolic Abnormalities.

Table 11.5.3. 1 Other Metabolic Abnormalities: Worst Grade per Patient by Dose Level.

Table 11.5.3. 2 Other Metabolic Abnormalities: Worst Grade per Cycle by Dose Level.

Table 11.5.3. 3 Other Metabolic Abnormalities: Worst Grade per Patient in the first Cycle by Dose Level.

Tables 11.5.3.1-.3 will have the following pattern but Grade column might be grouped if required.

| Abnormality* | DLI | DLII | • • • | DL n | Total |
|-----------------------|-----|------|-------|------|-------|
| Metabolic abnormality | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |
| * | | | | | |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) All biochemical abnormalities susceptible to be graded with NCI-CTCAE v.4.

Table 11.5.3. 4 Patients with missing Metabolic Evaluations.

| Dose level | Patient | Cycle | Lab. test |
|------------|---------|-------|-----------|

Table 11.5.3. 5 Shift of Metabolic Abnormalities. Baseline Grade vs. Worst Grade on First Cycle.

| | | | | | Wor | st Grade | e on Cy | cle 1 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose leve | el/Parameter | Baseline Grade | Gr. 1 Gr. 2 | | | | G | r. 3 | G | r. 4 |
| | | | N | % | N | % | N | % | N | % |
| | Hypercalcemia | 0 | | | | | | | | |
| DLI | | 4 | | | | | | | | |
| DLI | | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Hypercalcemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| ••• | | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Hypercalcemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| Total | | 4 | | | | | | | | |
| Total | ••• | 0 | • | • | • | • | | • | | |
| | | 4 | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) All metabolic abnormalities susceptible to be graded with NCI-CTCAE v.4.

Table 11.5.3. 6 Shift of Metabolic Abnormalities. Baseline Grade vs. Worst Grade on Treatment.

| | | | | | Worst | Grade | on Trea | atment | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose le | evel/Parameter | Baseline Grade | Gr. 1 Gr. 2 Gr. 3 | | | | | r.3 | Gr. 4 | |
| | | | N | % | N | % | N | % | N | % |
| | Hypercalcemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| DLI | | 4 | | | | | | | | |
| DLI | ••••• | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Hypercalcemia | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| ••• | ••• | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | Hypercalcemia | 0 | | | | | | | | |
| Total | | | | | | | | | | |
| Total | | 4 | | | | | | | | |
| | | 0 | | | | | | | | |

| _ |
|----------|
| • • • |
| 4 |
| <u> </u> |

Notes: Percentages based on number of patients by dose level. (\*) All metabolic abnormalities susceptible to be graded with NCI-CTCAE v.4.

Table 11.5.3. 7 Listing of Patients with Metabolic Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline.

| Dose level Patient Event | NCI-CTCAE v.4 at baseline | NCI-CTCAE v.4<br>at Cycle | Cycle |
|---|---|---|---|
|---|---|---|---|

Table 11.5.3. 8 Supportive Listing: Patients with Grade ≥3 Metabolic Abnormalities

| Dose level | Patient | Lab. test | Cycle | Examination date | * |
|------------|---------|-----------|-------|------------------|---|
|------------|---------|-----------|-------|------------------|---|

Note: (\*) It will include the following: Value at BL, Grade at BL, Onset day, Onset grade, Nadir day, Nadir value, Nadir grade, Recovery day, Recovery value, Recovery grade, Days Grade 3-4.

#### 11.5.4. Coagulation Abnormalities.

Table 11.5.4. 1 Coagulation Abnormalities: Worst Grade per Patient by Dose Level.

Table 11.5.4. 2 Coagulation Abnormalities: Worst Grade per Cycle by Dose Level.

Table 11.5.4. 3 Coagulation Abnormalities: Worst Grade per Patient in the first Cycle by Dose Level.

Tables 11.5.4.1-.3 will have the following pattern but Grade column might be grouped if required.

| Abnormality | DLI | DLII | • • • | DL n | Total |
|--------------------|-----|------|-------|------|-------|
| INR | | | | | _ |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |
| PTT | | | | | _ |
| Grade 1 - 4, n (%) | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |

Table 11.5.4. 4 Shift of Coagulation Abnormalities. Baseline Grade vs. Worst Grade on First Cycle.

| Dose level/Parameter* | | | Worst Grade on Treatment | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Baseline Grade | Gr. 1 | | Gr. 2 | | Gr.3 | |
| | | | N | % | N | % | N | % |
| DLI | INR increase | 0 | | | | | | |
| | | ••• | | | | | | |
| | | 3 | | | | | | |
| | | 0 | |
|-------|--------------|-----|---|
| | | ••• | |
| | | 3 | |
| | INR increase | 0 | |
| | | 3 | |
| ••• | | 0 | |
| | | 3 | |
| | INR increase | 0 | |
| | | ••• | |
| m . 1 | | 3 | |
| Total | | 0 | _ |
| | | 3 | |
| | | 5 | |

Notes: Percentages based on number of patients by dose level. (\*) INR and PTT. If data available.

Table 11.5.4. 5 Shift of Coagulation Abnormalities. Baseline Grade vs. Worst Grade on Treatment.

| | | | | Wors | t Grade | on Treat | ment | |
|---|---|---|---|---|---|---|---|---|
| Dose le | vel/Parameter* | Baseline Grade | G | r. 1 | G | r. 2 | G | r. 3 |
| | | | | % | N | % | N | % |
| | INR increase | 0 | | | | | | |
| DLI | | 3 | | | | | | |
| DLI | | 0 | | | | | | |
| | | ••• | | | | | | |
| | | 3 | | | | | | |
| | INR increase | 0 | | | | | | |
| | | ••• | | | | | | |
| | | 3 | | | | | | |
| ••• | ••• | 0 | | | | | | |
| | | 3 | | | | | | |
| | INR increase | 0 | | | | | | |
| | | ••• | | | | | | |
| Т-4-1 | | 3 | | | | | | |
| Total | ••• | 0 | | | | | | |
| | | ••• | | | | | | |
| | | 3 | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) INR and PTT. If data available.

Table 11.5.4. 6 Listing of Patients with Coagulation Abnormalities >G2 and Experience Grade Increase from Baseline.

| Dose level | Patient | Event | NCI-CTCAE v4 at baseline | NCI-CTCAE v4<br>at Cycle | Cycle |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| Table 11.5.4. 7 | Patients with | missing | Metabolic Evaluations. |
|-----------------|---------------|---------|------------------------|
|-----------------|---------------|---------|------------------------|

| | Ü | | |
|------------|---------|-------|-----------|
| Dose level | Patient | Cycle | Lab. test |

| Dose level | Patient | Cycle | Lab. test |
|------------|---------|-------|-----------|

# 11.6. Vital Signs, Physical Findings, ECG, LVEF and Pregnancy tests.

All statistical outputs in this section, whenever applicable, will be displayed according to assignment to prophylactic CSF use or not as well as per Dose level/Dose group or by cancer type or primary site if adequate number of patients is represented. Total numbers will be displayed independently, if applicable.

# 11.6.1. Vital Signs and Physical Findings.

Table 11.6.1.1 Physical examination during the Study by Cycle and Dose Level.

| | | Baseline | Cycle 1 | Cycle 2 | ••• | Cycle N |
|---|---|---|---|---|---|---|
| Dose<br>level | Patient<br>No | Normal/Abnormal | Normal/Abnormal | Normal/Abnormal | Normal/Abnormal | Normal/Abnormal |
| I | | | | | | |
| ••• | | | | | | |
| N | | | | | | |

Table 11.6.1.2 Performance Status during the Study by Cycle and Dose Level.

| | | Baseline | Cycle 1 | Cycle 2 | ••• | Cycle N |
|---------------|---------------|----------|---------|---------|-----|---------|
| Dose<br>level | Patient<br>No | PS | PS | PS | PS | PS |

I

• • •

N

Table 11.6.1.3 Weight Change during the Study by Dose Level.

| Dogo | Dotiont | Waight at bagalina | Cycle 1 | Cycle 2 | ••• | Cycle N |
|---|---|---|---|---|---|---|
| Dose | Patient | Weight at baseline — | % | % | % | % |
| level | No | (kg) | change | change | change | change |

I

| Dose<br>level | Patient<br>No | Weight at baseline —<br>(kg) | Cycle 1<br>%<br>change | Cycle 2<br>%<br>change | %<br>change | Cycle N<br>%<br>change |
|---|---|---|---|---|---|---|
| N | | | | | | |

# 11.6.2. Electrocardiogram.

Table 11.6.2 1 ECG during the Study by Dose Level.

| | | Baseline | Cycle 1 | Cycle 2 | ••• | Cycle N |
|---|---|---|---|---|---|---|
| Dose<br>level | Patient<br>No | Normal/Abnormal | Normal/Abnormal | Normal/Abnormal | Normal/Abnormal | Normal/Abnormal |
| I | | | | | | |
| ••• | | | | | | |
| N | | | | | | |

Table 11.6.2 2 ECG during the Study by Dose Level.

| | No cycles with delays | DLI | DLII | <br>DL n | Total |
|-------------|-----------------------|-----|------|----------|-------|
| | N | | | | |
| | Mean<br>Median | | | | |
| PR interval | Min | | | | |
| | Max | | | | |
| | STD | | | | |
| | N | | | | |
| | Mean | | | | |
| QT interval | Median | | | | |
| Q1 Interval | Min | | | | |
| | Max | | | | |
| | STD | | | | |
| | N | | | | |
| | Mean | | | | |
| * | Median | | | | |
| •••• | Min | | | | |
| | Max | | | | |
| | STD | | | | |

Note: (\*) Also RR interval, QRS interval, QTcF.

Table 11.6.2 3 QTcF Values during the Study by Dose Level.

| Dogo | Patient | Baseline – | Cycle 1 | Cycle 2 | • • • | Cycle N |
|---|---|---|---|---|---|---|
| Dose<br>level | No | QTcF (msec) | % | % | % | % |
| level | NO | QTCF (IIISEC) | change | change | change | change |
| I | | | | | | |
| ••• | | | | | | |
| N | | | | | | |
| 11 | | | | | | |

Table 11.6.2 4 QTcF (msec) Change per Patient during the Study by Dose Level.

| | | Baseline | Cycle 1 | Cycle 2 | ••• | Cycle N |
|---|---|---|---|---|---|---|
| Dose<br>level | Patient<br>No | QTcF(msec) | QTcF (msec) | QTcF(msec) | QTcF(msec) | QTcF (msec) |
| I | | | | | | |
| N | | | | | | |

Table 11.6.2 5 Shift of QTc. Baseline Grade vs. Worst Grade on Treatment.

| | | | | | Worst | Grade o | n Treati | ment. | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose leve | l/Parameter | Baseline Grade | G | ìr. 1 | G | r. 2 | G | r. 3 | G | r.4 |
| | | | N | % | N | % | N | % | N | % |
| | | 0 | | | | | | | | |
| DLI | QTc corrected | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | | 0 | | | | | | | | |
| ••• | QTc corrected | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | | 0 | | | | | | | | |
| Total | QTc corrected | | | | | | | | | |
| | - | 4 | | | | | | | | |

Table 11.6.2 6 QTcF Values during the Study by Doxorubicin Cumulative Dose.

| 1 4010 11.0.2 0 | Q T CT V d l d CS d d l l | ng the Study by | Donoru | orem ea | imulative Dose. | | |
|---|---|---|---|---|---|---|---|
| | QTcF(msec) | 0-xx (mg/m <sup>2</sup> ) | XX-XX | XX-XX | XX-XX | $xx-450 (mg/m^2)$ | Total |
| | N | | | | | | |
| | Mean | | | | | | |
| Previous to | Median | | | | | | |
| treatment or at Bl | L Min | | | | | | |
| | Max | | | | | | |
| | STD | | | | | | |

| | QTcF(msec) | 0-xx | $(mg/m^2)$ | XX-XX | XX-XX | XX-XX | xx-450 (mg/n | n <sup>2</sup> ) Total |
|---|---|---|---|---|---|---|---|---|
| 1 | V | | | | | | | |
| 1 | Mean | | | | | | | |
| | Median | | | | | | | |
| during treatment 1 | √lin | | | | | | | |
| | Max | | | | | | | |
| S | STD | | | | | | | |
| | | | ~ | | | | | |
| Table 11.6.2 7 L | sting of Patier | nts with ( | $\exists$ rade $\geq 2$ | | | | 0/ -£: 7 | Fotal cumulative do |
| Dose level | Patient | Cycle | QTc value | imeeci | irade NCI-<br>CTC v.4 | QTc at<br>Baseline | | of anthracyclines |
| | | | | | C1C v.4 | Dascillic | HOIIIBL | Of allulacyclines |
| 1.6.3. LVEF | • | | | | | | | |
| able 11.6.3 1 L | VEF (%) Char | ige per P | atient du | ring the S | Study by I | Oose Leve | 1. | |
| | Base | line | Cyc | le 1 | Cyc | de 2 | • • • | Cycle N |
| | ient Normal/A | hnormal | Normal/A | \hnormal | Normal/A | hnormal | Normal/Abnormal | Normal/Abnorm |
| level N | lo Nomal/A | OHOHIKH | 1 VOITIKII/1 | Monomia | 1 WITH AND T | Monomia | 1 VOITIKAI/2 VOITOITIKAI | 1 VOITI RAI/2 VOITOITI |
| I | | | | | | | | |
| • • • | | | | | | | | |
| N | | | | | | | | |
| 14 | | | | | | | | |
| | | | | | • | | | • |
| able 11.6.3 2 M | ledian LVEF V | Values (% | 6) during | the Stud | ly by Doxe | orubicin ( | Cumulative Dose. | |
| | QTcF(msec) | | $(mg/m^2)$ | XX-XX | XX-XX | XX-XX | xx-450 (mg/m | n <sup>2</sup> ) Total |
| 1 | N , | | ( ) | | | | ( 2 | / |
| | Mean | | | | | | | |
| | Median | | | | | | | |
| reatment or at BL 1 | | | | | | | | |
| | Max | | | | | | | |
| 1 | VIGA | | | | | | | |
| | STD | | | | | | | |
| S | STD | | | | | | | |
| <u> </u> | STD<br>N | | | | | | | |
| Accumulated Accumulated | STD<br>N<br>Mean | | | | | | | |
| Accumulated during | STD<br>N<br>Mean<br>Median | | | | | | | |
| Accumulated during | STD<br>N<br>Mean<br>Median<br>Min | | | | | | | |
| Accumulated during treatment | STD<br>N<br>Mean<br>Median<br>Min<br>Max | | | | | | | |
| Accumulated during treatment | STD<br>N<br>Mean<br>Median<br>Min | | | | | | | |
| Accumulated during treatment | STD<br>N<br>Mean<br>Median<br>Min<br>Max | | | | | | | |
| Accumulated during treatment | STD<br>N<br>Mean<br>Median<br>Min<br>Max<br>STD | Baseline | vs Wors | t Grade 4 | on Treatm | ent | | |
| Accumulated during treatment streament streame | STD N Mean Median Min Max STD | | | t Grade ( | on Treatm | | rade on Treatment | |
| Accumulated during treatment | STD N Mean Median Min Max STD | Baseline<br>aseline Gr | | | on Treatm | | rade on Treatment. | Gr. 3 |

| | | N | % | N | % | N | % |
|-------|-----|---|---|---|---|---|---|
| | 0 | | | | | | |
| DLI | ••• | | | | | | |
| | 0 | | | | | | |
| ••• | | | | | | | |
| ••• | ••• | | | | | | |
| | 0 | | | | | | |
| Total | | | | | | | |

Table 11.6.3 4 Listing of Patients with Grade  $\geq$  2 LVEF Decrease.

| Dose level | Patient | Cycle | LVEF<br>value (%) | Grade NCI-<br>CTCAE v.4 | LVEF at<br>Baseline | % of decrease from BL |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

# 11.7. Concomitant and Prophylactic Medication.

# 11.7.1. Concomitant and Prophylactic Medication During Study.

Table 11.7.1.1 Concomitant Medication during Study (ATC Level 1 and 4) by Dose Level.

| Medication Term | Medication Ten | mMedication Term | D | LI | DI | | | • | DL | ı n | To | ıtal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (ATC level 1) | (ATC level 2) | (ATC level 4) | N | % | N | % | N | % | N | % | N | % |

Note: Percentages based on number of patients by dose level.

Table 11.7.1.2 EPO/RBC and PlateletsTransfusions/CSF.

| Medication Term | Medication | Medication | D | LI | DI | | | • | DI | ر n | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (ATC level 1) | Term<br>(ATC level 2) | Term<br>(ATC level 4) | N | % | N | % | N | % | N | % | N | % |

EPO

RBC transfusion

Platelet transfusion

CSF\*

. . .

Notes: Percentages based on number of patients by dose level. (\*) Non-prophylactic CSF use.

Table 11.7.1.3 Patients with EPO/RBC and Platelets Transfusions/CSF.

Note: (\*) Non-prophylactic CSF use.

| Table 11.7.1. | 4 Proph | ylactic M | <b>1</b> edication | during Study | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Medication Ter | m | ] | DLI | DLII | | • • • | | D | Ln | To | otal |
| (ATC level 1)* | | N | % | N | % | N | % | N | % | N | % |
| | | | | | Cycle 1 | | | | | | |
| Steroids | | | | | - 3 | | | | | | |
| 5-HT antagonis | st. | | | | | | | | | | |
| Prokinetics | - | | | | | | | | | | |
| Aprepitant | | | | | | | | | | | |
| Other | | | | | | | | | | | |
| Total | | | | | | | | | | | |
| 1000 | | | | ( | Cycle>1 | | | | | | |
| Steroids | | | | | | | | | | | |
| 5-HT antagonis | st . | | | | | | | | | | |
| Prokinetics | | | | | | | | | | | |
| Aprepitant | | | | | | | | | | | |
| Other | | | | | | | | | | | |
| Total | | | | | | | | | | | |
| | | | | | All | | | | | | |
| Steroids | | | | | | | | | | | |
| 5-HT antagonis | st | | | | | | | | | | |
| Prokinetics | | | | | | | | | | | |
| Aprepitant | | | | | | | | | | | |
| Other | | | | | | | | | | | |
| Total | | | | | | | | | | | |
| Notes: Percentages antiemetic medicat Table 11.7.1. | ion will be a | dded, if clinic | ally indicated. | | | | | | | | , |
| Dose Level | Tumor<br>type | Patno | Cycle | AE prefered<br>Term | NCI-C | TCAE v. | /1 | metics*<br>//N) | Medicatio | n Term | ** |
| Notes:(*) Antieme | _ | | | | | | | Oose Lev | | | |
| Opioids* | | | DLI | DLII | | • • | | | Ln | | otal |
| Орюкь | | N | % | N | % | N | % | N | % | N | % |
| •••• | | | | | | | | | | | |
| ••• | | | | | | | | | | | |
| (*) The ATC classi | | | | | - | | | | | | |
| Table 11.7.1. | / Media | n Numbe | | | | | | | | | |
| Opioids* | | | DLI | DI | LII | | • • • | | DL n | Т | otal |
| N | | | | | | | | | | | |
| Mean | | | | | | | | | | | |
| Median | | | | | | | | | | | |
| Min | | | | | | | | | | | |
| Max | | | | | | | | | | | |
| STD | | 1 | 1, *** | 1 1 . 1 1 | ., ., . | | | | | | |
| (*) The ATC class | meanon meh | uaing aniaids | sand terms wall | ne selected and nm | wided hwel | mical reque | ST | | | | |

| tamida* | Γ | DLI | DLII | | | • | DI | _n | To | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| steroids* | N | % | N | % | N | % | N | % | N | % |
| •• | | | | | | | | | | |
| The ATC classification | n including steroids | and terms will be | selected and | provided by | clinical requ | est. | | | | |
| able 11.7.1.9 Kr | own CYP 3A | 4 Inducers/ | Inhibitor | s/Substra | ates Conc | comitant | Therapie | s at BL. | | |
| TVD 2 A 4* | Γ | DLI | DL: | Π | | • | DI | _n | To | tal |
| CYP3A4* | N | % | N | % | N | % | N | % | N | % |
| nhibitor | | | | | | | | | | |
| ••• | | | | | | | | | | |
| ote: (*) Also the possibi | lity of displaying or | ne table for each ( | category of Ir | ducers/Inhil | oitors or subs | trates. Some | medication v | vill be exclud | ed by clinica | reques |
| examethasone). | , , , , | | | | | | | | • | • |
| | | | ~ | | | oncomit | ant Thora | nies Dur | ing Treat | |
| able 11 7 1 10 L | isting of CYF | 3A4 Induc | ers/Inhih | 1fors/S111 | ostrates ( | | | | | ment |
| Table 11.7.1.10 L | | | | | | | | * | _ | |
| Dose Pat No | isting of CYF<br>Type* | 2 3A4 Induc<br>Literal Term | | ATC2 | | Sta | rt End | Reason for | _ | |
| | | | | | | | rt End | * | _ | |
| Dose Pat No | | | | | | Sta | rt End | * | _ | |

# 12. Appendix III. Efficacy Evaluation.

All statistical outputs will be displayed according to Dose level (grouped)/Cohort/Cancer type or primary site/CSF use or not/other clinical relevant variable (e.g. 2<sup>nd</sup> line SCLC by CTFI), whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

# 12.1. Efficacy Analysis.

### 12.1.1. Response.

Table 12.1.1.1 Overall response by Dose Level: Treated Patients.

| Or your Handra cards | D | LI | D | LII | • • | | | DL n | | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| Overall response | N | % | N | % | N | % | N | % | N | % |
| RECIST v.1.1 | | | | | | | | | | |
| CR | | | | | | | | | | |
| PR | | | | | | | | | | |
| SD < 4 months | | | | | | | | | | |
| SD≥4 months | | | | | | | | | | |
| PD | | | | | | | | | | |
| NE | | | | | | | | | | |
| Total | | | | | | | | | | |
| Other evaluation criteria (if | | | | | | | | | | |
| needed) | | | | | | | | | | |
| CR | | | | | | | | | | |
| PR | | | | | | | | | | |
| SD < 4 months | | | | | | | | | | |
| SD≥4 months | | | | | | | | | | |
| PD | | | | | | | | | | |
| NE | | | | | | | | | | |
| Total | | | | | | | | | | |

Note: Percentages based on number of patients by dose level.

Table 12.1.1.2 Overall response by Tumor type and Dose Level: Treated Patients.

| Townset | Or roundly more aware | D | DLI | | DLII | | • • • | | DL n | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Tumortype | Overall response | N | % | N | % | N | % | N | % | N | % |
| Breast | CR | | | | | | | | | | |
| | PR | | | | | | | | | | |
| | SD<4 months | | | | | | | | | | |
| | SD≥4 months | | | | | | | | | | |
| | PD | | | | | | | | | | |
| * | | | | | | | | | | | |
| | Total | | | | | | | | | | |
| Notes: Demontrops based on r | number of nations by doce level (*) Code | dimorta | <b>3</b> 000 | | | | | | | | |

Notes: Percentages based on number of patients by dose level. (\*) Coded tumor types.

| Oramil manage | DLI | DL | II | | DL n | Total |
|---|---|---|---|---|---|---|
| Overall response | N | % N | % N | % | N % | N % |
| R | | | | | | |
| 3 | | | | | | |
| O<4 months | | | | | | |
| D≥4 months | | | | | | |
| D | | | | | | |
| otal | | | | | | |
| ote: Percentages based on numb | per of evaluable patients by do | ose level. | | | | |
| able 12.1.1.4 Overall | Response by Tumo | | | le Patien | | m . 1 |
| Tumortype | Overall respon | nse DL<br>N | I DLII<br>% N % | <br>N | DL % N | Ln Total % N % |
| reast | CR | 11 | /0 14 /0 | 11 | /0 IN | /0 11 / |
| .casi | PR | | | | | |
| | SD<4 months | | | | | |
| | SD≥4 months | | | | | |
| * | PD | | | | | |
| * | | | | | | |
| ••• | Total | | | | | |
| tes: Percentages based on num | ber of evaluable patients by o | dose level. (*) Coded t | umortypes. | | | |
| able 12.1.1.5 SD $\geq$ 4 1 | months by Dose Lev | vel: Evaluable | Patients. | | | |
| | | | Patients. | | DLn | Total |
| able 12.1.1.5 SD $\geq$ 4 months | DLI | DLII | | | DL n | Total<br>N % |
| SD≥4 months | | | | 6 N | | Total<br>N % |
| SD≥4 months | DLI | DLII | | ó N | | |
| SD≥4 months<br>to<br>es | DLI | DLII | | ó N | | |
| SD≥4 months to es otal | DLI<br>N % | DLII<br>N % | | 6 N | | |
| SD≥4 months to es otal | DLI<br>N % | DLII<br>N % | | <u></u> 6 Л | | |
| SD≥4 months o es otal ote: Percentages based on numb | DLI<br>N %<br>per of evaluable patients by do | DLII<br>N %<br>ose level. | | 6 N | | |
| SD≥4 months o es otal ote: Percentages based on numb | DLI<br>N %<br>per of evaluable patients by do | DLII N % ose level. During Study. | <br>o N % | 6 N | N % | N % |
| SD≥4 months To es otal ote: Percentages based on numb | DLI<br>N %<br>per of evaluable patients by do | DLII<br>N %<br>ose level. | <br>N % | | % | N % |
| SD≥4 months for the second of the second o | DLI N % Der of evaluable patients by definition Description Descr | DLII N % ose level. During Study. Baseline | N % Cycle 1 Tumor marker | Tur | N % mor marker | N % Cycle N Tumor marke |
| SD≥4 months ores otal ote: Percentages based on numb able 12.1.1.6 Tumor I | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months o es otal ote: Percentages based on numb able 12.1.1.6 Tumor I | DLI N % Der of evaluable patients by definition Description Descr | DLII N % ose level. During Study. Baseline | N % Cycle 1 Tumor marker | Tur<br>e value | N % mor marker | N % Cycle N Tumor marke |
| SD≥4 months ores otal ote: Percentages based on numb able 12.1.1.6 Tumor I | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months o es otal ote: Percentages based on numb able 12.1.1.6 Tumor I | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months or tes total ote: Percentages based on numbrable 12.1.1.6 Tumor I Dose Patient level No | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months for the second of the second o | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months or tes total ote: Percentages based on numbrable 12.1.1.6 Tumor I Dose Patient level No | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months for one of the state of the st | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| for fees fortal forter. Percentages based on number able 12.1.1.6 Turnor I for feel for feel feel feel feel feel feel feel fee | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months for fessotal ote: Percentages based on numbrable 12.1.1.6 Tumor I Dose Patient level No I | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months lo lo lo lo lo lote: Percentages based on numb able 12.1.1.6 Tumor I Dose Patient level No I | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months for fessortal ote: Percentages based on numbrable 12.1.1.6 Tumor I Dose Patient level No I N | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months [o fes otal ote: Percentages based on numb able 12.1.1.6 Tumor I Dose Patient level No I | DLI N % Der of evaluable patients by definition D Turnor type/ | DLII N % ose level. During Study. Baseline Tumor marker | N % Cycle 1 Tumor marker value / (%) chang | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months for essortal ote: Percentages based on numbrable 12.1.1.6 Tumor I Dose Patient level No I N | DLI N % Der of evaluable patients by der Marker Evolution D Tumor type/ Tumor marker* | DLII N % oselevel. During Study. Baseline Tumor marker value | Cycle 1 Tumor marker value / (%) chang from BL | Tur<br>e value | mor marker /(%) change | N % Cycle N Tumor market value / (%) char |
| SD≥4 months o es otal ote: Percentages based on numb able 12.1.1.6 Tumor I Dose Patient level No I N offavailable data able 12.1.1.7 Charact | DLI N % Der of evaluable patients by definition D Turnor type/ Turnor marker* | DLII N % oselevel. During Study. Baseline Tumor marker value | Cycle 1 Tumor marker value / (%) chang from BL | Tur<br>e value<br>f | mor marker /(%) change from BL | Cycle N Tumor marke value / (%) char from BL |
| SD≥4 months o es otal ote: Percentages based on numb able 12.1.1.6 Tumor I Dose Patient level No I N | DLI N % Der of evaluable patients by defended by the series of Patients value of Pa | DLII N % Osselevel. During Study. Baseline Tumor marker value with Clinical Be Best TTI | Cycle 1 Tumor marker value / (%) chang from BL | Tur<br>e value<br>f | mor marker /(%) change from BL | Cycle N Tumor market value / (%) chart from BL |

| PS | lines of treatmen | t) Previous | CT | PM01183 | Reason |
|----|-------------------|-------------|----|---------|--------|
| | previous | CT | | | |
| | treatment | | | | |

Note: (\*) "Evidence of Clinical Benefit" when response is CR, PR or SD≥4 months and/or no evidence of PD with increase tumor markers, if non-evaluable as per RECIST v.1.1.

Table 12.1.1.8 Characteristics of Patients with Clinical Benefit based on any Specific Tumor Marker Criteria.

| Dose<br>level | Patient<br>No | Sex/<br>Age/<br>PS | Tumor<br>type | Number of lines of previous treatment | Agents (previous treatment) | Best<br>Response<br>Previous CT | TTP<br>Previous<br>CT | Cycles<br>Received<br>PM01183 | Overall<br>Response<br>for tumor<br>marker | * |
|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|

Notes: (\*Also overall response by RECIST v1.1, TTP, OS, Treatment discontinuation reason, e.g. CA-125 value at BL, Nadir value CA-125. In patients for whom response to treatment are evaluated by both RECIST v1.1 and any specific turnor marker criteria, the date of response and progression will be the earliest date of the two methods.

#### Table 12.1.1.9 Progression-Free Survival: Evaluable Patients.

Summary\*

N=XX

Events X(XX.X%)

Censored X (XXXX%)

Median X.X 95% CI (X.X-X.X)

PFS at 3 months XX.X% 95% CI XX.X%-XX.X%)

PFS at 6 months XX.X% 95% CI XX.X%-XX.X%)

Note: (\*) If any particular tumor type or any other clinically relevant variable is adequately represented and PFS at 12, and 24 months also if available data.

#### Table 12.1.1.10 Duration of Response.

Summary\*

N=XX

Events X(XXX%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

Duration of Response at 3 months XX.X% 95% CIXX.X%-XX.X%)

Duration of Response at 6 months XX.X% 95% CIXX.X%-XX.X%)

(\*) If any particular tumor type or any other clinically relevant variable is adequately represented and DR at 12 and 24 months also if available data.

#### Table 12.1.1.11 Overall survival.

Summary\*

N=XX

Events X(XX.X%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

OS at 6 months XX.X% 95% CIXX.X%-XX.X%)

OS at 12 months XX.X% 95% CIXX.X%-XX.X%)

OS at 18 months XX.X% 95% CIXX.X%-XX.X%)

(\*) Only for Cohort B but if requested also for cohort A.

# 13. Figures.

All statistical outputs will be displayed according to Dose level (grouped)/Cohort/Cancer type or primary site/CSF use or not/other clinical relevant variable (e.g. 2nd line SCLC by CTFI), whenever applicable and if an adequate number of patients is represented. The figures' layout may change to adequately accommodate cohort/group size as appropriate



Figure 13.1 1 Pattern of Hematological/non Hematological DLTs in Individual Patients.

Also if applicable pattern for Neutropenia for patients with prophylactic CSF vs. No CSF.



Figure 13.1 2 Transaminase Series in Individual Patients.





Figure 13.1 4 Barcharts of Adverse Events or Laboratory Abnormalities by Dose Level/Cohort/Tumor type/ or Other Clinical Relevant Variable.



Figure 13.1 5 Hematology/Transaminase Worst Severity by Cycle.



Figure 13.1 6 LVEF/QTcF Boxplot by Dose Level.



Figure 13.1 7 Boxplot QTcF Worst Value by Cycle.



Figure 13.1 8 Duration of Response.



Kaplan-Meier curve of duration of response (If any response is observed).

Figure 13.1 9 Progression-free Survival by Dose level/Cohort/Tumor type/ or Other Clinical Relevant Variable.



Figure 13.1 10 Overall Survival.



Figure 13.1 11 Waterfall Graphs.



Waterfall graphs will be displayed in measurable lesions by RECIST v.1.1Also graphs for each tumor type/cohort and for responders.

Figure 13.1 12 Spider plot: Evolution of RECIST v.1.1 Assessments.



Spider plot will be displayed individually for each tumor type/cohort / or Other clinical relevant variable, if required.

Figure 13.1 13 Best RECIST v.1.1 Efficacy Assessment in Evaluable pts per Tumour Type.



Figure 13.1 14 Treatment Exposure and Reasons for Discontinuation per Tumour Type.



Figure 13.1 15 Best RECIST v.1.1 Response According to Line of Treatment.







Figure 13.1 17 Number of Cycles, Reason for Treatment Discontinuation for Patients with Response or Clinical Benefit.







Figure 13.1 19 Number of Cycles, Reason for Treatment Discontinuation and Response in Patients who Received PM001183 Alone.



# 14. Database Listings.

- Listing 14.1 Patient Registration.
- Listing 14.2 Demography.
- Listing 14.3 Patient Disposition.
- Listing 14.4 Protocol Deviations.
- Listing 14.5 Patient Populations.
- Listing 14.6 Selection Criteria.
- Listing 14.7 Medical History.
- Listing 14.8 Cancer History.
- Listing 14.9 Current Disease.
- Listing 14.10 Prior Surgery.
- Listing 14.11 Prior Radiotherapy.
- Listing 14.12 Prior Anticancer Therapy.
- Listing 14.13 Signs and Symptoms.
- Listing 14.14 Tumor Assessment (Target Lesions).
- Listing 14.15 Tumor Assessment (Non Target Lesions).
- Listing 14.16 Tumor Assessment (New Lesions).
- Listing 14.17 Radiological Response (RECIST v.1.1).
- Listing 14.18 Clinical Evaluation Response.
- Listing 14.19 Tumor Marker Evaluation Response.
- Listing 14.20 Overall Cycle Response.
- Listing 14.21 Treatment Exposure.
- Listing 14.22 Hematology Laboratory Results.
- Listing 14.23 Clinical Chemistry and Coagulation Laboratory Results.
- Listing 14.24 Physical Examination and Performance Status (PS).
- Listing 14.25 Vital Signs.
- Listing 14.26 ECG Results.
- Listing 14.27 Left Ventricular Ejection Fraction (LVEF) Results.
- Listing 14.28 Other Tests and Procedures Results.
- Listing 14.29 Adverse Events.
- Listing 14.30 Concomitant Therapy.

Listing 14.31 End of Treatment.

Listing 14.32 Follow-up.

Listing 14.33 Follow-up: Antitumor therapy.

Listing 14.34 Death Report.

Listing 14.35 Best Study Overall Response.

Listing 14.36 Off Study.

Listing 14.37 Signature Report.

# 15. SAP Version History.

# 15.1.SAP Version History v1.

After the first version of the SAP was approved by the responsible physician, the medical writer and the biostatistics manager, a new protocol "substantial amendment No. 1" was included; therefore the SAP has been updated (highlighted in *italic bold*) in accordance with the new version (version 2) of the protocol as follows:

- Changes in Study design/dose escalation and G-CSF/CSF primary prophylaxis and MTD definition has been rephrased in order to maintain consistency between DLT and MTD definitions.
- Changes in Inclusion/exclusion criteria have been done: a maximum age limit of 75 years old has been set and the inclusion of patients with mesothelioma has been allowed.
- Some minor changes and corrections have been done in the text and the mock shells to allow a clear and unambiguous communication of the science and statistics of the trial.

## **Summary of proposed changes from section 2.1 to 8:**

### **Section 2.1 Primary Objective:**

#### **Original text:**

• To determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 in combination with doxorubicin in patients with selected advanced solid tumors.

## Change to:

• To determine the MTD and the RD of PM01183 in combination with doxorubicin with primary prophylaxis with G-CSF in patients with selected advanced solid tumors (if DLTs of the combination without G-CSF prophylaxis are exclusively related to neutropenia).

### Section 3. Study design:

## **Original text:**

..... All evaluable patients within a dose level will be followed for at least one cycle (i.e., three weeks) before dose escalation may proceed. Dose escalation will be terminated once the MTD or the last dose level (DL4) is reached, whichever occurs first.

#### Change to:

... All evaluable patients within a dose level will be followed for at least one cycle (i.e., three weeks) before dose escalation may proceed. **Dose escalation will be terminated once the** MTD or the last dose level (DL4) is reached, whichever occurs first, except if all DLTs

occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than 7 days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis.

## Section 5.2.1.1 Determination of MTD and RD

## **Original text**:

......If >1 evaluable patient during dose escalation at a given DL experience a DLT during Cycle 1, that DL will be considered the MTD and dose escalation will be terminated. The DL immediately below the MTD, or DL4 if the MTD is not yet defined during dose escalation before the last DL (i.e., DL4) is reached, will be expanded up to a minimum of nine evaluable patients. If less than three among the first nine evaluable patients treated within the expansion cohort experience a DLT during Cycle 1, this DL will be the RD.

## Change to:

......If >1 evaluable patient during dose escalation at a given DL experience a DLT during the first cycle, that level will be considered the MTD and dose escalation will be terminated except if all DLTs occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than 7 days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis.

#### **Section 8.1 Stratification and Covariate Analysis:**

### **Original text:**

No stratification by prognostic factors or tumor types is planned. If a disease is adequately represented, response rates might be analyzed descriptively, and time-related parameters might be analyzed according to the Kaplan-Meier method. Efficacy parameters could also be subjected to further analysis (if appropriate), considering correlation with factors of probable prognostic value such as subject PS at entry, disease burden, prior therapies, other disease-specific known prognostic factor, or population characteristics, etc. using the appropriate test (Fisher's exact test, Spearman test, etc.).

# Change to:

No stratification by prognostic factors or tumor types is planned. If a disease is adequately represented, response rates might be analyzed descriptively, and time-related parameters might be analyzed according to the Kaplan-Meier method. Efficacy parameters could also be subjected to further analysis (*if appropriate*), considering correlation with factors of *known* prognostic value such as subject PS at entry, disease burden, prior therapies, other disease-specific known prognostic factor, *or population characteristics*, etc. using the appropriate test (Fisher's exact test, Spearman test, etc.).

### **Section 8.3 Subgroups Analysis:**

## **Original text:**

If any cancer groups of patients are sufficiently represented, a separate analysis by tumor type and evaluation criteria (RECIST, GCIC) will be performed.

If there is a representative number of patients who receive a maximal total cumulative dose of 450 mg/m<sup>2</sup> of doxorubicine and continue treatment with PM01183 alone at the recommended dose as a single agent, a separate analysis will be performed and tables, listings and graphic representations for this population will be provided when applicable.

Exploratory safety and efficacy analyses considering the three groups (below RD, RD and over RD) will be performed if appropriate.

#### Change to:

If any cancer subtype or any other baseline characteristics of patients are adequately represented, a separate analysis by tumor type and efficacy as per RECIST v1.1, will be performed.

If there is a representative number of patients who receive a maximal total cumulative dose of 450 mg/m<sup>2</sup> of doxorubicin and continue treatment with PM01183 alone, a separate analysis will be performed and tables, listings and graphic representations for this population will be provided when applicable.

## Summary of changes in Section 9. Tables, Listings and Graphs:

The following new paragraphs have been added,

#### **Original text:**

Statistical outputs, whenever is applicable, will be displayed according to assignment to prophylactic G-CSF factors use or not as well as per Dose level. Totals numbers will be displayed independently, if applicable. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort size as appropriate.

Patients included and treated over 75 yrs old will be excluded from all tables, listings and graphs in this SAP. Detailed narratives of these patients will be shown in the CSR.

If the number of categories or items would not yield appropriate tabular or graphic representations, detailed listings will be shown instead.

#### Change to:

Statistical outputs, whenever is applicable, will be displayed according to assignment to prophylactic CSF factors use or not as well as per Dose level/Dose group or by cancer type or primary site if adequate number of patients is represented. Totals numbers will be displayed independently, if applicable. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort size as appropriate.

If the number of categories or items would not yield appropriate tabular or graphic representations, detailed listings will be shown instead.

Patients included and treated over 75 **years** old will be excluded from all tables, listings and graphs in this SAP. Detailed narratives of these patients will be shown in the clinical study report CSR.

## **Summary of changes in Section 10. Appendix I. Patients disposition:**

New tables and variables have been included after clinical request and some minor changes and corrections have been done in the text and the mock shells to allow a clear and unambiguous communication of the science and statistics of the trial.

## **Section 10.1.1 Patients Treated, Elegible, and Evaluable:**

In Table 10.1.1.4 Number of Patients Evaluable for the Analysis, a footnote has been added and categories have been reordered. Note:(\*) Efficacy by RECIST v.1.1. A listing of patient non evaluable by RECIST v.1.1 will be provided.

#### Section 10.1.2 Treatment discontinuation:

Table 10.1.2.1 Treatment Discontinuation by Dose Level adds two more tables and the possibility of include other reasons for treatment discontinuation not included in the CRF categories and added, after clinical review. Notes:(\*) Reasons for treatment discontinuation for patients who discontinued while the combination or PM alone will be provided, if required. (\*\*) If applicable, a supporting listing 10.1.2.1.a will be provided and reasons for treatment discontinuation may suffer re-categorization after clinical review. A new table have been added Table 10.1.2.4 Listing of patients with Discontinuation after cycle 9. All tables have been renumbered.

Table 10.1.2.1 Treatment Discontinuation by Dose Level adds the following Note:(\*) If applicable, a supporting listing 10.1.2.1.a will be provided and reasons for treatment discontinuation may suffer re-categorization after clinical review.

Table 10.1.2.4 Listing of patients with Discontinuation with PM01183 alone has been included.

#### **Section 10.2.1 Patients Characteristics at Baseline:**

Table 10.2.1.1 Age at Entry by Dose Level: categories of age are between 18 and 75 years (both inclusive).

Tables from Previous Section 10.2.9 Physical Examination, Vital Sings, Electrocardiogram and Other Tests have been moved to Section 10.2.1 Patient Characteristics at Baseline.

Table 10.2.1.8 has been renamed to Demographic Parameters by Dose level and added the footnote Note: (\*) Height (cm) and BSA (DuBois formula).

#### **Section 10.2.2 Cancer History:**

New tables have been added. Table 10.2.2.3 TTP Last Prior Therapy.

Table 10.2.2.4 Stage at Diagnosis by Dose Level and Table 10.2.2.5 Tumor Type by Dose level have been deleted by clinical indication and 10.2.2.4 Tumor type by dose level include the following footnote: Note: (\*) CRF categories will be shown and a supportive table 10.2.2.6.a will be provided for subcategories (e.g. sarcomas).

New variables have been added to Table 10.2.2.7. See footnote as last TTP prior therapy and best response to prior therapy.

#### Section 10.2.3 Sites involved:

All tables included in this section will be shown by dose level and/or tumor type, if required.

Two new tables have been included: Table 10.2.3.5 Bulky Disease and Dose Level. Table 10.2.3.6 Median Sum of Diameter of Target Lesions (mm).

### **Section 10.2.4 Previous Treatment Summary.**

Table 10.2.4.2 Previous systemic therapy type by dose level/tumor type has been added.

## **Section 10.2.7 Previous Anticancer Medical History.**

All tables of this section have now the possibility of being displayed by Tumor type, if required. In addition, tables from Tables 10.2.7.1 Agents of Previous Anticancer Therapy (ATC level 1&4) by Dose Level/Tumor Type to Table 10.2.7.3 Summary Statistics. No of Lines of Prior Anticancer Therapy by Dose Level/Tumor Type will show only therapies with chemotherapy containing and excluding hormonal therapy.

A new table has been added: Table 10.2.7.5 No of Agents of Last Prior Anticancer Therapy before PM01183 treatment by Dose Level/Tumor type.

**Section 10.2.8 to 10.2.11:** All statistical outputs, whenever applicable, will be displayed according to assignment to prophylactic G-CSF factors use or not as well as per Dose level. Totals numbers will be displayed independently, if applicable.

## Section 10.2.12 Signs and Symptoms at Baseline:

Table 10.2.12.2 has been renamed to Listing of Adverse events Grade > 1.

#### Section 10.2.13 Concomitant and Prophylactic Medication Starting Pre-Study:

New tables have been added: Table 10.2.13.4 No of Patients with Opioids Treatment at Baseline by Dose Level, Table 10.2.13.5 Median Number of No of Opioids at Baseline per patient by Dose Level. Table 10.2.13.6 No of patients with Steroids Treatment at Baseline by Dose Level. Table 10.2.13.7 Known CYP 3A4 Inducers/Inhibitors/Substrates Concomitant Therapies at BL and Listing 10.2.13.8 Known CYP 3A4 Inducers/ Inhibitors/Substrates) Concomitant Therapies at BL.

In addition, tables 10.2.13.4 and 10.3.5 have been renumbered to 10.2.13.7 and 10.2.13.8 and the following footnote has been added: Note: (\*) Also the possibility of display one table for each category Inducers/Inhibitors or substrates. Some medication will be excluded by clinical request (e.g. Dexamethasone)

### **Summary of changes in Section 11. Appendix II Safety Evaluation:**

All statistical outputs in this section, whenever applicable, will be displayed according to the discontinuation of the combination treatment. Treatment exposure, delays, omissions and reductions will be shown before and after discontinuation. Dose level may suffer categorization (e.g. RD\le or RD), if required.

Each specific table and listing will have a comprehensive header identifying the group/cohort of treatment and/or the specific study drug, whenever necessary.

New tables and variables have been included after clinical request and some minor changes and corrections have been done in the text and the mock shells to allow a clear and unambiguous communication of the science and statistics of the trial.

## Section 11.1.1 Cumulative Dose, Dose Intensity and Relative Dose Intensity:

Table 11.1.2.12 Reasons for Doxorubicin Dose reduction by Dose Level has been deleted because any dose reductions of doxorubicin will be a deviation and will be described in the Protocol Deviation section.

Tables 11.1.2.14 and 11.1.3.6 Listing of Cycles Delays/Reductions due to Nausea/Vomiting have been renamed to Listing of Cycles Delays due to Non-Hematological Adverse Events.

### **Section 11.2.1 Dose-Limiting Toxicities:**

A new table has been added: Table 11.2.1.1 Summary of patients with DLT by Dose Level.

#### **Section 11.3.1 Display of Adverse Events:**

All statistical outputs, whenever applicable, will be displayed according to assignment to prophylactic CSF use or not as well as per Dose level. Total numbers will be displayed independently, if applicable.

#### **Section 11.4.2 Serious Adverse Events:**

The following text has been added. All serious adverse events will be listed only for the purpose of reconciliation with the database of pharmacovigilance. The listings provided by the Product Safety department will be used for the clinical study report.

#### **Section 11.5.1 Hematological abnormalities:**

New tables have been added: Table 11.5.1.6 Shift of Hematological Abnormalities. Baseline Grade vs. Worst Grade on First Cycle. and Table 11.5.1.8 Listing of patients with Biochemical Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline and 11.5.1.9 Summary of Characteristics of Wpp Hematological Abnormalities G3-4.

## **Section 11.5.2 Biochemical Abnormalities:**

New tables have been included: Table 11.5.2.7 Listing of patients with Biochemical Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline and 11.5.2.8 Summary of Characteristics of Wpp Biochemical Abnormalities G3-4.

#### **Section 11.5.3 MetabolicAbnormalities:**

New tables have been added in this section: Table 11.5.3.5 Shift of Metabolic Abnormalities. Baseline Grade vs Worst Grade on First Cycle. Table 11.5.3.6 Shift of Metabolic Abnormalities. Baseline Grade vs Worst Grade on Treatment. Table 11.5.3.7 Listing of Patients with Metabolic Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline. Table 11.5.3.8 Supportive Listing: Patients with Grade  $\geq$  3 Metabolic Abnormalities.

## **Section 11.5.4 Coagulation Abnormalities:**

New tables have been added in this section: Table 11.5.4.4 Shift of Coagulation Abnormalities. Baseline Grade vs Worst Grade on First Cycle. Table 11.5.4.5 Shift of Coagulation Abnormalities. Baseline Grade vs Worst Grade on Treatment. Table 11.5.4.6 Listing of Patients with Metabolic Abnormalities >G2 and Experience Grade Increase (wpp) from Baseline.

#### Section 11.6.2 Electrocardiogram.

Tables of this section have been renumbered and new tables added. Table 11.6.2.5 Shift of QTc. Baseline Grade vs. Worst Grade on Treatment. Table 11.6.2.7 Listing of Patients with Grade  $\geq$  2 QTc Interval Prolonged.

#### Section 11.6.3 LVEF.

Tables of this section have been renumbered and new tables added. Table 11.6.3.3 Shift of LVEF. Baseline Grade vs. Worst Grade on Treatment. Table 11.6.3.4 Listing of Patients with Grade ≥ 2 LVEF Decrease.

### Section 11.6.4 Pregnancy Test and Adequate Contraception.

Table 11.6.4.1 Patients with Positive Pregnancy Test and Not Adequate Contraception Method has been deleted. If any patients are positive for the pregnancy test or are not using an adequate contraception method, they will be reported in the Protocol Deviation section.

#### **Section 11.7 Concomitant and Prophylactic Medication:**

The titles of Tables 11.7.1.2 and 11.7.1.3 have been modified to EPO/RBC and Platelets transfusions/CSF. Also, the following footonote has been added: Note: (\*) Non-prophylactic CSF use.

New tables have been added: Table 11.7.1.5 Known CYP 3A4 Inducers/Inhibitors/Substrates Concomitant Therapies During Study and Table 11.7.1.6. are renamed and depending on the number of observations will be shown separately and include the footnote Note: (\*) Also the possibility of display one table for each category Inducers/Inhibitors or substrates. Some medication will be excluded by clinical request (e.g. Dexamethasone)

New tables have been included in this section, and therefore all tables have been renumbered. Table 11.1.7.5 No of Patients with Opioids Treatment During Treatment by Dose Level, Table 11.1.7.6 Median Number of No of Opioids During Treatment per Patient by Dose Level. Table 11.1.7.7 No of Patients with Steroids Treatment During Treatment by Dose Level.

### Section 11.7.1 Concomitant and Prophylactic Medication During Study.

This subsection includes new Table 11.7.1.5 Known CYP 3A4 Inducers/Inhibitors/Substrates Concomitant Therapies During Study and Table 11.7.1.6 Listing of CYP 3A4 Inducers or Inhibitors (or Substrates) Concomitant Therapies During Study.

## **Summary of changes in Section 12. Appendix III Efficacy Evaluation:**

The Clinical Benefit criterion has been changed from when response is CR, PR or SD≥3 months to when response is CR, PR or SD≥4 months. In addition, the possibility of calculating time-to-event parameters PFS and DR at 12 and/or 24 months has been added.

Some other minor changes and corrections have been done in the text and the mock shells to allow a clear and unambiguous communication of the science and statistics of the trial.

## **Summary of changes in Section Figures 13.**

A new Figure 13.6 Boxplot QTcF worst value by cycle has been included.

**Section 15 SAP Version History** has been included in order to be consistent with the Protocol amendment No. 1 of this study and due to the inclusion of new TLGs for the cancer subgroups that could be adequately represented in accordance with PharmaMar's SOPs.

## 15.2.SAP Version History v2.

Some other changes were implemented in a new version of the SAP (v.3) for adequate representation of cancer subgroups (highlighted in *italic bold*) and a summary of changes are shown at the end of this section.

### Summary of changes implemented in SAP (v.3).

- All TLGs detailed in Section 9 will be represented per Dose level or Dose group (RD<, etc..) and/or also per cancer type or primary site if an adequate number of patients is represented.</li>
- The granulocyte colony-stimulating factor may be abbreviated indistinctively as CSF or as G-CSF in the tables and text detailed in Section 9.

- Some minor changes and corrections have been done in the text and the mock shells in order to provide a clear and unambiguous communication of the science and statistics of the trial.
- In addition to these changes, minor typographic corrections have been done throughout the document.

## Summary of proposed changes by section:

Section 10.2.2 Cancer History

Table 10.2.2.5 has been renamed to 10.2.2.5 Summary of Cancer History per Patient *and Tumor Type.* A footnote has been added to this listing to include the possibility of displaying any specific characteristics of previous Patient History for each Tumor type. If required, tabulations for specific categories will be shown as Supportive tables.

Section 10.2.7 Previous Systemic Therapies

New tables have been included: Table 10.2.7.7 Agents of Prior Anticancer Therapy by Tumor Type/Dose Level and Table 10.2.7.9 Platinum-Free Survival by Tumor Type/Dose level

Section 11.5 Clinical Laboratory Evaluation

New tables have been included: Table 11.5.1.10 Anemia wpp/wpc and Use of EPO per Dose Level, 11.5.1.11 Patients with Anemia Grade 3/4 in Cycle >1 and Use of EPO., Table 11.5.1.14 Thrombocytopenia wpp/wpc and Use of Transfusions per Dose Level in Cycle>1., Table 11.5.1.15 Patients with Thrombocytopenia Grade 3/4 in Cycle >1 and Use of Transfusions; Table 11.5.18 Neuthropenia wpp/wpc and Use of Prophylactic CSF per Dose Level in Cycle>1, 11.5.13.19 Patients with Neutrophenia Grade 3/4 in Cycle>1 and Use of Prophylactic CSF.

Section 11.7 Concomitant and Prophylactic Medication

A new table has been included: Table 11.7.1.5 Patients with Nausea and /or Vomiting G3/4 and Use of Antiemetics in Cycle >1.

In Figure 13.1, the possibility of drawing pattern for Neutropenia for patients with prophylactic CSF vs. No CSF has been added.

New Figures 13.10 and 13.15 have been included for graphic representation of the subgroup populations and specific characteristics.

## 15.3.SAP Version History v3.

Two substantial protocol amendments "No. 2 and No. 3" and one "non-substancial protocol amendment "No.1" have been implemented after the approval of SAP v3; therefore, the SAP has been updated (highlighted in *italic bold*) in accordance with the current version of the protocol (version 4.0) as follows:

• Dose escalation began at PM01183 3.0 mg FD and DOX 50.0 mg/m2 q3wk. Patients received DOX capped at 2.0 m² of BSA up to a maximum cumulative dose (MCD) of 450 mg/m². After DOX withdrawal, PM01183 administration could continue alone at its full single-agent RD (7.0 mg FD or 4.0 mg/m² on D1 q3wk). A first amendment to the protocol set a maximum age of 75 years for patients enrolled in the study and allowed primary G-CSF prophylaxis during dose escalation to explore the potential of this approach to reach a higher RD. However, DLTs occurred at the same dose level regardless of primary G-CSF prophylaxis, and they included grade 3/4 FN, grade 4 thrombocytopenia and grade 4 septic shock. Based on these results, the MTD was defined at PM01183 5.0 mg FD and DOX 50.0 mg/m² regardless of G-CSF support. The immediately lower DL (PM01183 4.0 mg and DOX 50.0 mg/m²) was then expanded, and DLTs were found in none of three patients with G-CSF and in one of ten (10%) patients without G-CSF (FN). Thus, PM01183 4.0 mg FD and DOX 50.0 mg/m² was defined as the RD for this combination, and was not further expanded with primary G-CSF prophylaxis.

Objective antitumor activity was found in more than one third of patients across most tumor types at all DLs explored. It was particularly promising in small cell lung cancer (SCLC) patients treated as second-line after chemotherapy failure and in endometrial cancer patients. Hence, the RD was further expanded to confirm the preliminary antitumor activity observed in these settings. All DLTs found after RD expansion were myelosuppression-related. Three of 14 patients with endometrial cancer had DLTs. Less than one third of second-line SCLC patients had DLTs, but more than 20% of them had FN, thus suggesting further dose adjustment was also required in this subsetting.

Following these findings, the initial RD underwent a 20% reduction in the DOX dose to 40 mg/m². In addition, the PM01183 dose was adapted to a BSA-based dose of 2.0 mg/m², after a logistic regression analysis of pooled data from phase II clinical trials with single-agent PM01183 in several solid tumors had suggested that patients with the lowest BSA values could have a greater risk of developing grade 3/4 thrombocytopenia.

- In the new cohort B, exploratory assessment for progression-free survival (PFS) and overall survival (OS) will be performed and patients will be followed for survival for up to 18 months after the first study dose.
- All TLGs described by DL will be also done by most adequate dose grouping/cohort/tumor type or other clinical relevant variable where appropriate. The tables' layout and headings may change to adequately accommodate cohort/group as appropriate.
- Some minor changes (e.g. clarify dose level grouping to dose level/cohort/Tumor type or other clinical relevant variable) and corrections in the text and in the mock shells have been done in order to achieve a clear, unambiguous communication of the science and statistics of the trial.

## Summary of changes implemented in SAP (v.4).

#### **Section 2.1 Primary Objective:**

### **Original text:**

• To determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 in combination with doxorubicin with primary prophylaxis with granulocyte colony-stimulating factor (G-CSF) in patients with selected advanced solid tumors [if dose-limiting toxicities (DLTs) of the combination without G-CSF prophylaxis are exclusively related to neutropenia].

### **Changes to:**

• To determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 in combination with doxorubicin in patients with selected advanced solid tumors.

## **Section 2.1 Secondary Objectives:**

#### **Original text:**

- To characterize the safety profile and feasibility of this combination in patients with selected advanced solid tumors.
- To characterize the pharmacokinetics (PK) of this combination and to detect major drug-drug PK interactions.
- To obtain preliminary information on the clinical antitumor activity of this combination in non-heavily pretreated selected solid tumor patients.
- To evaluate the pharmacogenomics (PGx) in tumor samples of patients exposed to PM01183 and doxorubicin at the RD in order to assess potential markers of response and/or resistance.

#### **Changes to:**

- To determine the MTD and the RD of PM01183 in combination with doxorubicin with primary prophylaxis with granulocyte-colony stimulating factor (G-CSF) in patients with selected advanced solid tumors [if dose-limiting toxicities (DLTs) of the combination without G-CSF prophylaxis are exclusively related to neutropenial.
- To characterize the safety profile and feasibility of this combination in patients with selected advanced solid tumors.
- To characterize the pharmacokinetics (PK) of this combination and to detect major drug-drug PK interactions.
- To obtain preliminary information on the clinical antitumor activity of this combination in non-heavily pretreated selected solid tumor patients.
- Based on promising findings, to explore the feasibility, safety and efficacy of a potential improvable dose of this combination in selected tumor types [i.e. small cell lung cancer (SCLC) and endometrial cancer).

• To evaluate the pharmacogenomics (PGx) in tumor samples of patients exposed to PM01183 and doxorubicin at the RD in order to assess potential markers of response and/or resistance.

#### Section 3 Study design:

## **Original text:**

. . . . .

Cohorts of three to six patients will be included at each dose level (DL). If no DLT occurs in more than one patient within each cohort, escalation will proceed to the following dose level. If one of the first three evaluable patients experiences a DLT, the dose level should be expanded up to six patients. The MTD will be the lowest dose level explored during the dose escalation at which more than one evaluable patient experience a DLT in Cycle 1. All evaluable patients within a dose level will be followed for at least one cycle (i.e., three weeks) before dose escalation may proceed. Dose escalation will be terminated once the MTD or the last dose level (DL4) is reached, whichever occurs first, except if all DLTs occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than 7 days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis.

In the event of DLTs occurring in the first patient at the first level, the second and third patients will be included at least two weeks apart. Otherwise and/or at subsequent dose levels, all patients within a dose level may be treated simultaneously.

Patients treated at the expansion cohort must be evaluable by the RECIST version 1.1 and/or by serum markers (carbohydrate antigen-125, CA-125) in the case of ovarian cancer, as appropriate [according to the Gynecologic Cancer Intergroup (GCIG) specific criteria] (see study protocol, section 9.7), and must have documented disease progression according to any of these criteria. The tumor type(s) that will be eligible to be included in the expansion cohort at the RD will be chosen according to the preliminary efficacy observed among those previously treated during the escalation phase, and will be discussed and agreed between the investigators and the Sponsor.

Intermediate dose levels could be tested on agreement between the Investigator and the Sponsor, if deemed appropriate.

Patients will receive PM01183 and doxorubicin until progression, unacceptable toxicity, consent withdrawal or while it is considered to be in their best interest. More specifically, doxorubicin will be administered in the absence of disease progression or unacceptable toxicity until a maximal total cumulative dose of 450 mg/m² is reached; once this dose has been reached, the patients may continue treatment with PM01183 alone at the established single-agent RD, 7.0 mg FD q3wk.

Tumor assessments will be done every six weeks while on treatment. After treatment discontinuation, patients will be followed every four weeks until resolution or stabilization of all toxicities, if any. Patients discontinuing treatment without progression will be followed every two months until disease progression, other antitumor therapy, death or the date of study termination, whichever occurs first (see study protocol, section 5.9).

Antitumor response will be assessed using the RECIST version 1.1 and/or serum tumor markers as appropriate (e.g., ovarian cancer markers).

Patients will be evaluated at scheduled visits on three study periods: Pre-treatment, Treatment and Follow-up (see study protocol, section 5.2).

## Changes to:

. . . . .

Cohorts of three to six patients will be included at each dose level (DL). If no DLT occurs in more than one patient within each cohort, escalation will proceed to the following dose level.

The MTD will be the lowest dose level explored during the dose escalation at which more than one evaluable patient experience a DLT in Cycle 1. All evaluable patients within a dose level will be followed for at least one cycle (i.e., three weeks) before dose escalation may proceed. Dose escalation will be terminated once the MTD or the last dose level (DL4) is reached, whichever occurs first, except if all DLTs occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than seven days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis. An expansion cohort to complete a minimum of nine evaluable patients will be recruited at the immediate lower dose level, or at the last dose level (DL4) if the MTD is not defined yet. This level will be confirmed as the RD if less than one third of the first nine evaluable patients experience DLT during Cycle 1.

Further to the finding of encouraging antitumor activity in the first 43 evaluable patients (13 responses, including four complete responses, with five partial responses in eight patients with small cell lung cancer, and one complete and one partial response in three patients with endometrial cancer), expansion of the cohort treated at the RD has been increased to include approximately 30 additional patients, for a total of around 39 patients.

In addition, a new cohort B of 20 evaluable patients with small cell lung cancer (SCLC) who failed treatment after first-line standard cytotoxic-containing therapy and at least nine evaluable patients with endometrial cancer will be included to further define the efficacy, safety and feasibility of a doxorubicin dose adaptation (doxorubicin 40 mg/m² and PM01183 2.0 mg/m²). Patients in this cohort who have received ten cycles of the doxorubicin/PM01183 combination or have to discontinue doxorubicin due to a cardiac AE may continue receiving treatment with single-agent PM01183 at 4.0 mg/m² q3wk if patient benefit is perceived according to the Investigator. These patients will be followed every three months until death or the date of study termination, whichever occurs first.

Patients will be divided into two cohorts. Cohort A will consist of all patients included before the implementation of protocol amendment #3, and Cohort B will consist of all patients included after the implementation of protocol amendment #3.

. . . . . .

Patients will receive PM01183 and doxorubicin until progression, unacceptable toxicity, consent withdrawal or while it is considered to be in their best interest. More specifically,

doxorubicin will be administered in the absence of disease progression or unacceptable toxicity before a maximal total cumulative dose of 450 mg/m<sup>2</sup> is reached. Thus, a maximum of ten cycles of the combination will be administered to patients with SCLC and endometrial cancer included in the new cohort B. Once this dose has been reached, the patients may continue treatment with PM01183 alone at the established single-agent RD, 7.0 mg FD q3wk and for patients included in the new cohort B they may continue treatment with PM01183 alone at 4.0 mg/m<sup>2</sup> q3wk.

Tumor assessments will be done every six weeks while on treatment. After treatment discontinuation, patients will be followed every four weeks until resolution or stabilization of all toxicities, if any. Patients discontinuing treatment without progression will be followed every two months until disease progression, other antitumor therapy, death or the date of study termination, whichever occurs first (see study protocol, section 5.9).

In the new cohort B, patients with SCLC and endometrial cancer will be followed every three months until death or the date of study termination, whichever occurs first. Antitumor response will be assessed using the RECIST v.1.1 and/or serum tumor markers as appropriate (e.g., ovarian cancer markers).

No serum markers will be evaluated in patients with SCLC and endometrial cancer included in the new cohort B. Patients will be evaluated at scheduled visits on three study periods: Pre-treatment, Treatment and Follow-up (see study protocol, section 5.2).

In addition, a new cohort B of 20 evaluable patients with small cell lung cancer (SCLC) who failed treatment after first-line standard cytotoxic-containing therapy and at least nine evaluable patients with endometrial cancer will be included to further define the efficacy, safety and feasibility of a doxorubicin dose adaptation. These patients will be treated with doxorubicin at 40 mg/m² administered as an i.v. bolus/short infusion followed by PM01183 at 2.0 mg/m² as a 1-hour i.v. infusion on Day 1 q3wk. The administered doses of both PM01183 and doxorubicin will be capped at 2.0 m² of body surface area (BSA) for any patients exceeding this BSA value. Patients in this cohort who have received ten cycles of the doxorubicin/PM01183 combination or have to discontinue doxorubicin due to a cardiac AE may continue receiving treatment with single-agent PM01183 at 4.0 mg/m² q3wk if patient benefit is perceived according to the Investigator. These patients will be followed every three months until death or the date of study termination, whichever occurs first.

#### **Section 4.1 Sample size:**

#### **Original text:**

The number of patients may vary depending both on the tolerability to PM01183 combined with doxorubicin and the number of dose levels required to identify the MTD. Approximately between four and 27 evaluable patients will participate in this study.

## Changes to:

The number of patients may vary depending both on the tolerability to PM01183 combined with doxorubicin and the number of dose levels required to identify the MTD. *Approximately*, 100 evaluable patients will participate in this study.

#### **Section 4.2 Dose escalation:**
# **Original text:**

The dose escalation schedule is summarized in the following table:

Dose escalation schedule

| DL | No. of patients | | Dose of doxorubicin<br>(mg/m²) / PM01183 (mg FD)<br>on Day 1 q3wk |
|---|---|---|---|
| DL-1 | 0-6 | 100 / 42.85 | 50 / 3.0 |
| DL1 | 3-6 | 100 / 50 | 50 / 3.5 |
| DL2 | 3-6 | 100 / 71.4 | 50 / 5.0 |
| DL3 | 3-6 | 100 / 85.7 | 50 / 6.0 |
| DL4 | 3-6 | 100 / 100 | 50 / 7.0 |

The DL-1 level is to be explored only if DL1 is defined as the MTD.

DI, dose intensity; DL, dose level; FD, flat dose.

. . . .

Intra-patient dose escalation will not be allowed under any circumstances.

# **Changes to:**

The dose escalation schedule is summarized in the following table:

Dose escalation schedule (cohort A).

| DL | No. of patients | | Dose of doxorubicin<br>(mg/m²) / PM01183 (mg FD)<br>on Day 1 q3wk |
|---|---|---|---|
| DL-1 | 0-6 | 100 / 42.85 | 50 / 3.0 |
| DL1 | 3-6 | 100 / 50 | 50 / 3.5 |
| DL2 | 3-6 | 100 / 71.4 | 50 / 5.0 |
| DL3 | 3-6 | 100 / 85.7 | 50 / 6.0 |
| DL4 | 3-6 | 100 / 100 | 50 / 7.0 |

The DL-1 level is to be explored only if DL1 is defined as the MTD.

DI, dose intensity; DL, dose level; FD, flat dose.

. . . .

Intra-patient dose escalation will not be allowed under any circumstances.

# New cohort after implementation of protocol amendment #3 (Cohort B):

Patients with SCLC and endometrial cancer will consecutively receive the following on Day 1 q3wk (three weeks = one treatment cycle):

- Doxorubicin: i.v. bolus/short infusion at a dose of 40 mg/m<sup>2</sup>, administered as described above, immediately followed by:
- PM01183: i.v. infusion over one hour at a dose of 2.0 mg/m<sup>2</sup>, administered as described above.

Both doxorubicin and PM01183 doses will be capped at 2.0  $m^2$  of BSA for individuals exceeding this BSA value. Doses will have to be recalculated for patients showing  $a \ge 10\%$  change in total body weight value compared to previous cycle.

PM01183 doses will be rounded to the first decimal, if necessary. Doxorubicin doses will be rounded according to institutional guidelines/standard practices.

#### Section 5.1 Patient evaluability criteria:

### **Original text:**

. . .

The "All Evaluable for Efficacy Patients" analysis set is defined as all evaluable patients measured according to the RECIST v.1.1 at least six weeks after treatment initiation in all patients with measurable disease, and/or by CA-125 levels if applicable, i.e. ovarian cancer with at least 2 x upper limit of normal (ULN) at baseline [according to the Gynecologic Cancer Intergroup (GCIG/Rustin) specific criteria].

If early progression occurs (i.e., before six weeks since treatment) or if treatment should be discontinued due to any treatment-related toxicity before appropriate tumor assessments have been performed, the patient's objective response will be considered as a treatment failure or progressive disease (PD); therefore, their data will be included in the analysis of objective response as per RECIST v.1.1.

All analyses will be performed as per protocol rather than on an intention-to-treat-basis. Any departure from the planned treatment according to the study schedule will be listed and documented in the clinical study report.

# Changes to:

. . . .

The "All Evaluable for Efficacy Patients" analysis set is defined as all evaluable patients measured according to the RECIST v.1.1 at least six weeks after treatment initiation in all patients with measurable disease, and/or by CA-125 levels if applicable, i.e. ovarian cancer with at least 2 x upper limit of normal (ULN) at baseline [according to the Gynecologic Cancer Intergroup (GCIG/Rustin) specific criteria]. No serum markers will be evaluated in patients with SCLC and endometrial cancer included in the new cohort B.

If early progression occurs (i.e., before six weeks since treatment) or if treatment should be discontinued due to any treatment-related toxicity before appropriate tumor assessments have been performed, the patient's objective response will be considered as a treatment failure or progressive disease (PD); therefore, their data will be included in the analysis of objective response as per RECIST v.1.1.

In the new cohort B of patients with SCLC and endometrial cancer, a patient evaluable for efficacy should have received at least one complete cycle (including observation period) and be evaluable as per RECIST, except if non-evaluability is due to treatment failure such as drug-related toxicity, death or early unequivocal PD outside the central nervous system.

All analyses will be performed as per protocol rather than on an intention-to-treat-basis. Any departure from the planned treatment according to the study schedule will be listed and documented in the clinical study report.

#### Section 5.2.1.1 Determination of MTD and RD:

# **Original text:**

A minimum of three patients will be included at each dose level. If no patients experience a DLT during the first cycle, the dose will be escalated. If one of three patients experiences a DLT, three additional patients will be included at that level. If >1 evaluable patient during dose escalation at a given dose level experience a DLT during the first cycle, that level will be considered the MTD and dose escalation will be terminated except if all DLTs occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than 7 days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis

Determination of the maximum tolerated dose.

| No. of patients<br>evaluable*<br>for DLT | No. of patients with DLTs in Cycle 1 | Action |
|---|---|---|
| | 0 | Escalate DL until DL4 is reached |
| 3 | 1 | Add 3 patients |
| | >1 | MTD |
| 6 | 1 | Escalate DL until DL4 is reached |
| O | >1 | MTD |
| DL, dose level; DLT, dose-limiting toxicities; MTD, maximum tolerated dose. | | |
| * Patients not evalua | ble for DLT during do | ose optimization must be replaced. |

Decisions on delayed-onset DLTs (i.e., those DLTs occurring after Cycle 1) will be individually discussed between the Investigators and Sponsor, and might end affecting the definition of the proposed RD for phase II clinical trials.

# Changes to:

A minimum of three patients will be included at each dose level. If no patients experience a DLT during the first cycle, the dose will be escalated. If one of three patients experiences a DLT, three additional patients will be included at that level. If >1 evaluable patient during dose escalation at a given dose level experience a DLT during the first cycle, that level will be considered the MTD and dose escalation will be terminated except if all DLTs occurring at a given dose level are related to neutropenia (e.g., febrile neutropenia, grade 4 neutropenia lasting more than 7 days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the lowest dose level where exclusively neutropenia-related DLTs have occurred, and will follow the same original schedule but with compulsory primary G-CSF prophylaxis *The DL immediately below the MTD*, or DL4 if the MTD is not reached during dose escalation and the last dose level (DL4) is reached, was to be initially expanded up to a minimum of nine evaluable patients. If less than three among the first nine evaluable patients treated within the expansion cohort experience a DLT during Cycle 1 this DL will be the RD.

Further to the finding of encouraging antitumor activity in the first 43 evaluable patients (13 responses, including four complete responses, with five partial responses in eight patients with SCLC, and one complete and one partial response in three patients with

endometrial cancer), expansion of the cohort treated at the RD has been increased to include approximately 30 additional patients, for a total of around 39 patients.

Determination of the maximum tolerated dose.

| No. of patients<br>evaluable*<br>for DLT | No. of patients with DLTs in Cycle 1 | Action |
|---|---|---|
| | 0 | Escalate DL until DL4 is reached |
| 3 | 1 | Add 3 patients |
| | >1 | MTD |
| 6 | 1 | Escalate DL until DL4 is reached |
| U | >1 | MTD |

DL, dose level; DLT, dose-limiting toxicities; MTD, maximum tolerated dose.

Decisions on delayed-onset DLTs (i.e., those DLTs occurring after Cycle 1) will be individually discussed between the Investigators and Sponsor, and might end affecting the definition of the proposed RD for phase II clinical trials.

In the new cohort B of patients with SCLC and endometrial cancer, a patient evaluable for efficacy should have received at least one complete cycle (including observation period) and be evaluable as per RECIST, except if non-evaluability is due to treatment failure such as drug-related toxicity, death or early unequivocal PD outside the central nervous system.

#### **Section 5.2.2.2 Efficacy:**

#### **Original text:**

Although it is not the main objective of this study, antitumor activity will be measured according to the RECIST v.1.1 at least six weeks after treatment initiation in all patients with measurable disease, or by evaluation of tumor markers if applicable (e.g., ovarian cancer). Patients included at the RD in the expansion cohort must be evaluable per RECIST v.1.1 or by evaluation of tumor markers (see Section 7.4 for efficacy evaluation).

If any particular tumor type is adequately represented, time-related parameters [i.e., progression-free survival (PFS), overall survival (OS)] will be analyzed according to the Kaplan-Meier method, if appropriate.

. . . .

# **Changes to:**

Although it is not the main objective of this study, antitumor activity will be measured according to the RECIST v.1.1 at least six weeks after treatment initiation in all patients with measurable disease, or by evaluation of tumor markers if applicable (e.g., ovarian cancer). Patients included at the RD in the expansion cohort must be evaluable per RECIST v.1.1 or by evaluation of tumor markers (see Section 7.4 for efficacy evaluation).

No serum markers will be evaluated in patients with SCLC and endometrial cancer included in the new cohort B.

<sup>\*</sup> Patients not evaluable for DLT during dose optimization must be replaced.

<sup>\*\*</sup> For replacement of patients and replacement of patients after implementation of Amendment #3 (see Protocol section 5.3).

If any particular tumor type is adequately represented, time-related parameters [i.e., progression-free survival (PFS), overall survival (OS)] will be analyzed according to the Kaplan-Meier method, if appropriate.

In the new cohort B, exploratory assessment for progression-free survival (PFS) and overall survival (OS) will be performed.

In addition, patients with SCLC and endometrial cancer included in the new cohort B will be followed for survival for up to 18 months after the first study dose.

....

# Section 7.3.1 Treatment Administration and Exposure

#### **Original text:**

Exposure to each treatment will be described by dose level (or most adequate dose grouping) for all patients who have received at least one of the study treatments.

. . . . .

The number of cases, median, standard deviations, 95% confidence interval (CI), minimum and maximum values for the parameters defined above will be tabulated by dose level (or most adequate dose grouping) and drug (PM01183 and doxorubicin).

### Changes to:

. . . .

Exposure to each treatment will be described by dose level (or most adequate dose grouping/cohort/tumor type or other clinical relevant variable) for all patients who have received at least one of the study treatments.

<u>...</u>

The number of cases, median, standard deviations, 95% confidence interval (CI), minimum and maximum values for the parameters defined above will be tabulated by dose level (or most adequate dose grouping/cohort/tumor type or other clinical relevant variable) and drug (PM01183 and doxorubicin).

# Section 7.4.1. Exploratory Analysis of Antitumor Activity:

#### **Original text:**

. . . .

Response rates will be characterized using descriptive statistics (95% confidence interval). If applicable, overall response rate (percentage of patients with PR or CR), percentages for PR or CR separately and percentage of patients with  $SD \ge 3$  and/or 4 months will be analyzed.

. . .

The characteristics of the patients achieving an objective response or  $SD \ge 3$  and/or 4 months by RECIST v.1.1, or a clinically significant improvement measured by tumor markers, will be displayed.

# **Changes to:**

. . . .

Response rates will be characterized using descriptive statistics (95% confidence interval). If applicable, overall response rate (percentage of patients with PR or CR), percentages for PR or CR separately and percentage of patients with  $SD \ge 4$  months will be analyzed.

. . . .

The characteristics of the patients achieving an objective response or  $SD \ge 4$  months by RECIST v.1.1, or a clinically significant improvement measured by tumor markers, will be displayed.

In addition, patients with SCLC and endometrial cancer included in the new cohort B will be followed for survival for up to 18 months after the first study dose.

#### Section 9. Tables, Listings and Figures:

# **Original text:**

Statistical outputs, whenever is applicable, will be displayed according to assignment to prophylactic CSF use or not as well as per Dose level/Dose group or by cancer type or primary site if adequate number of patients is represented. Totals numbers will be displayed independently, if applicable. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort size as appropriate.

If the number of categories or items would not yield appropriate tabular or graphic representations, detailed listings will be shown instead.

Patients included and treated over 75 years old will be excluded from all tables, listings and graphs in this SAP. Detailed narratives of these patients will be shown in the clinical study report CSR.

. . . .

#### Changes to:

After the implementation of Amendment #3, a new cohort B of patients with SCLC and endometrial cancer has been included. All statistical outputs will be displayed according to dose level (grouped)/cohort/tumor type or primary site/CSF use or not/other relevant clinical variable, whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

If the number of categories or items would not yield appropriate tabular or graphic representations, detailed listings will be shown instead.

Patients included and treated over 75 years old will be excluded from all tables, listings and graphs in this SAP. Detailed narratives of these patients will be shown in the clinical study report (CSR).

The abbreviation DL shown in the mock tables might refer to dose level (grouped <RD, RD, etc...)/cohort (i.e. Cohort A and B)/tumor type or primary site (i.e. Ovarian, SCLC (2nd line), etc...)/CSF use or not/other clinical relevant variable .....

Sections 10.2.8 Hematological Evaluation at Baseline to 10.2.11 Other Metabolic Evaluations at Baseline; 11.3.1 Display of Adverse Events; 11.5 Clinical Laboratory Evaluations; 11.6 Vital Signs, Physical findings and Pregnancy tests, ECG,LVEF; **Appendix III 12.1 Efficacy Analysis** 

The following paragraph has been removed from the aforementioned sections:

"All statistical outputs in this section, whenever applicable, will be displayed according to assignment to prophylactic CSF use or not as well as per Dose level/Dose group or by cancer type or primary site if adequate number of patients is represented. Total numbers will be displayed independently, if applicable."

And the following text replaces the removed paragraph in the following sections: 10. Appendix I. Patients Characteristics; 11. Appendix II. Safety Evaluation; 12. Appendix III. Efficacy Evaluation.

"All statistical outputs will be displayed according to dose level (grouped)/cohort/tumor type or primary site/ CSF use or not/other relevant clinical variable, whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate."

#### Section 10.2.1 Patients Characteristics at Baseline

A footnote has been added.

Table 10.2.1.1. Age at Entry by Dose Level.

| Age at entry | DLI | | DLII · | | | | | DL n | | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % | N | % |
| 18-45 years | | | | | | | | | | |
| 18-45 years<br>46-55 years | | | | | | | | | | |
| ••• | | | | | | | | | | |
| < 76* years | | | | | | | | | | |
| Total | | | | | | | | | | |

Note: Percentages based on number of patients by dose level. (\*) Example categories.

# **Section 10.2.7 Previous Anticancer Medical Therapy**

New tables have been included:

Table 10.2.7.9 CTFI by Dose Level/Cohort/Tumor type

| CTFI/TFI* | DLI | | DLII | | • • • | | DL n | | Total | |
|-----------|-----|---|------|---|-------|---|------|---|-------|---|
| CILILIL. | N | % | N | % | N | % | N | % | N | % |
| Resistant | | | | | | | | | | |

Sensitive

Note: (\*) CTFI (chemotheraphy free interval)/for SCLC patients and TFI (Systemic chemotherapy free interval) for Endometrial patients. Calculated from the last therapy previous therapy with ATC coded "L01XA" and calculated as the difference from the end of therapy to the PD, e.g. for SCLC patients Categories R (resistant) and S (sensitive).

Table 10.2.7.10 Summary Statistics: CTFI by Dose Level/Cohort/Tumor type.

| Tumor range | type*/Median | and <sub>DLI</sub> | DLII | ••• | DL n | Total |
|---|---|---|---|---|---|---|
| N | | | | | | |
| Mean | | | | | | |
| Median | | | | | | |
| Min | | | | | | |
| Max | | | | | | |
| STD | | | | | | |

Note: (\*) Tumor type, if apply

# Section 11. Safety Evaluation.

### **Original:**

All statistical outputs in this section, whenever applicable, will be displayed according to the discontinuation of the combination treatment. Treatment exposure, delays, omissions and reductions will be shown before and after discontinuation.

# **Changes to:**

All statistical outputs in this section, whenever applicable, will be displayed according to the discontinuation of the combination treatment. Treatment exposure, delays, omissions and reductions will be shown considering the whole study treatment and/or before and after discontinuation, if appropriate.

Table 11.1.1.4. Dose Intensity by Dose Level:

# Original table:

| Drug | Dose intensity | DLI | DLII | • • • | DL n | Total |
|---|---|---|---|---|---|---|
| PM01183<br>(mg/week) | N<br>Mean<br>Median<br>Min<br>Max | | | | | |
| Doxorubicin<br>(mg/m²/week) | N<br>Mean<br>Median<br>Min<br>Max | | | | | |

# **Changes to:**

| Drug | Dose intensity | DLI | DLII | ••• | DL n | Total |
|--------------|----------------|-----|------|-----|------|-------|
| | N | | | | | |
| | Mean | | | | | |
| PM01183* | Median | | | | | |
| (mg/week) | Min | | | | | |
| | Max | | | | | |
| | STD | | | | | |
| | N | | | | | |
| DM011024 | Mean | | | | | |
| PM01183* | Median | | | | | |
| (mg/m²/week) | Min | | | | | |
| | Max | | | | | |

| Drug | Dose intensity | DLI | DLII | • • • | DL n | Total |
|--------------|----------------|-----|------|-------|------|-------|
| | STD | | | | | |
| | N | | | | | |
| | Mean | | | | | |
| Doxorubicin | Median | | | | | |
| (mg/m²/week) | Min | | | | | |
| | Max | | | | | |
| | STD | | | | | |

<sup>(\*)</sup> Results of dose intensity maybe grouped and presented in mg/m²/week for patients treated in the Cohort A, if appropriate,

# **Section 11.3.1 Display of Adverse Events.**

The following paragraph is added:

All adverse events tables will be listed by cohort and dose level (or most adequate dose grouping/tumor type/other clinical relevant variable or according to the discontinuation of the combination treatment, if required).

### **Section 12. Efficacy Evaluation.**

# **Original:**

All statistical outputs will be displayed according to Dose level (grouped)/Cohort/Cancer type or primary site/CSF use or not/other clinical relevant variable, whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

# **Changes to:**

All statistical outputs will be displayed according to Dose level (grouped)/Cohort/Cancer type or primary site/CSF use or not/other clinical relevant variable (e.g. 2<sup>nd</sup> line SCLC by CTFI), whenever applicable and if an adequate number of patients is represented. Summary tables will have source data footnotes that will refer to the relevant listings. The tables' layout may change to adequately accommodate cohort/group size as appropriate.

# Section 12.1.1 Response.

Table 12.1.1.9 add the following footnote:

Note: (\*) If any particular turnor type or any other clinically relevant variable is adequately represented and PFS at 12, and 24 months also if available data.

The following category has been added to Table 12.1.1.10.

Table 12.1.1.10 Duration of Response.

Summary\*

N=XX

Events X(XX.X%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

Duration of Response at 3 months XX.X% 95% CIXX.X%-XX.X%)

Duration of Response at 6 months XXX% 95% CIXXX%-XXX%)

(\*) If any particular tumor type or any other clinically relevant variable is adequately represented and DR at 12 and 24 months also if available data.

The following new Table 12.1.1.11 has been added.

#### Table 12.1.1.11 Overall survival.

Summary\*

N=XX

Events X(XX.X%)

Censored X (XX.X%)

Median X.X 95% CI (X.X-X.X)

OS at 6 months XX.X% 95% CI XX.X%-XX.X%)

OS at 12 months XX.X% 95% CIXX.X%-XX.X%)

OS at 18 months XX.X% 95% CIXX.X%-XX.X%)

(\*) Only for Cohort B but if requested also for cohort A.

# Section 13. Figures.

The following paragraph is added:

All statistical outputs will be displayed according to Dose level (grouped)/Cohort/Cancer type or primary site/CSF use or not/other clinical relevant variable (e.g. 2nd line SCLC by CTFI), whenever applicable and if an adequate number of patients is represented. The figures' layout may change to adequately accommodate cohort/group size as appropriate.

Figures from this section have changed table numbering due to the inclusion of new graphs and the modification of others.

# Original graph:

Figure 13.1.3 Barcharts of Hematological/Biochemical Abnormalities by Dose level



# Changes to:

Figure 13.1.3 Barcharts of Adverse Events or Laboratory Abnormalities



Figure 13.1.3 Barcharts of Adverse Events or Laboratory Abnormalities by Dose Level/Cohort/Tumor type/or Other Clinical Relevant Variable.



The following graphics representations have been included:

Figure 13.1.9 Waterfall Graphs change to 13.1.11 and change layout to allow grouping graphical representations.



Figure 13.1.10 Overall Survival



Figure 13.1.12 Spider plot: Evolution of RECIST v1.1 Assessments.



Figure 13.1.18 Efficacy and individual TTP in Selected Patients by BSA/CTFI and Treatment Discontinuation.



Figure 13.1.19 Number of Cycles, Reason for Treatment Discontinuation and Response in Patients who Received PM001183 alone.

